Document status: Final SAP Version 2.0 Amendment 1.0



## STATISTICAL ANALYSIS PLAN

A Phase 1b/2a, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Recombinant Human Plasma gelsolin (rhu-pGSN) Added to Standard of Care in Subjects Hospitalized for Acute Community-acquired Pneumonia (CAP)

Protocol No.: BT-201

**Product Code:** rhu-pGSN

**PREPARED FOR:** BioAegis Therapeutics, Inc. (BTI)

675 US-1, North Brunswick Township,

NJ 08902,

**USA** 

Phone: +1 203-952-6373

PREPARED BY: Novotech (Australia) Pty Ltd

Level 3, 235 Pyrmont Street

Pyrmont, NSW, 2009

Australia

**DATE OF ISSUE:** 27 August 2018 (Draft Version 0.1)

19 September 2018 (Draft Version 0.5)

03 October 2018 (Final Draft 0.9) 02 November 2018 (Final 1.0)

03 December 2018 (Final 2.0 Amendment 1.0)

**VERSION/STATUS:** Final 2.0 Amendment 1.0

**VERSION DATE:** 03 December 2018

**AUTHOR:** Jan Steyn


## **SUMMARY OF CHANGES FROM SAP VERSION 1.0**

# Section 11.2.2 page 25, the following text has been added:

Additionally, counts (%) of number subjects with values out of normal range at each scheduled time point will also be presented along with shift tables that will represent the changes in normal range categories across post-baseline time points.

# Section 17, the following tables have been added:

| No. | Title | Analysis<br>Population |
|---|---|---|
| 14.3.4.1.2.1 | SD: Summary of CBC Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.1.2.2 | MAD: Summary of CBC Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.2.2.1 | SD: Summary of Coagulation Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.2.2.2 | MAD: Summary of Coagulation Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.3.2.1 | SD: Summary of Comprehesive Metabolic Profile Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.3.2.2 | MAD: Summary of Comprehesive Metabolic Profile Shifts from Baseline (Low, Normal, High) | Safety |

# Section 18, the following listings have been added:

| No. | Title | Analysis Population |
|---|---|---|
| 16.2.8.1.2.1 | SD: Abnormal CBC | Intent-to-Treat |
| 16.2.8.1.2.2 | MAD: Abnormal CBC | Intent-to-Treat |
| 16.2.8.2.2.1 | SD: Abnormal Coagulation | Intent-to-Treat |
| 16.2.8.2.2.2 | MAD: Abnormal Coagulation | Intent-to-Treat |
| 16.2.8.3.2.1 | SD: Abnormal Comprehensive Metabolic Profile | Intent-to-Treat |
| 16.2.8.3.2.2 | MAD: Abnormal Comprehensive Metabolic Profile | Intent-to-Treat |


# **SAP APPROVAL**

By my signature, I confirm that this SAP has been reviewed by BioAegis Therapeutics, Inc., and has been approved for use on the BT-201 study:

| Name | Title / Company | Signature | Date |
|---|---|---|---|
| Mark DiNubile | CMO. BioAegis | Mad D. Narle | Dec. 3, 2018 |
| Jan Steyn | Principal<br>Biostatistician/<br>Novotech | Blue | 3DEC2018 |

# Table of contents

| 1. | IN | TRODUCTION | 8 |
|-----|------|------------------------------------|----|
| 2. | PR | OJECT OVERVIEW | 9 |
| 2 | 2.1 | Study Design | 9 |
| 2 | 2.2 | Objectives | 9 |
| 2 | 2.3 | Sample Size | 10 |
| 2 | 2.4 | Randomization | 10 |
| 3. | STA | ATISTICAL CONSIDERATIONS | 11 |
| 4. | ΑN | IALYSIS POPULATIONS | 13 |
| 4 | 1.1 | Population Descriptions | 13 |
| 5. | PR | OTOCOL DEVIATIONS | 14 |
| 6. | SU | BJECT DISPOSITION | 15 |
| 7. | DE | MOGRAPHIC AND BASELINE INFORMATION | 16 |
| - | 7.1 | Demographics | 16 |
| - | 7.2 | Medical history | 16 |
| 7 | 7.3 | Pregnancy Test (Serum and Urine) | 16 |
| 7 | 7.4 | Serology | 16 |
| - | 7.5 | Other baseline characteristics | 16 |
| 8. | ST | UDY DRUG ADMINISTRATION | 17 |
| 9. | PH | ARMACOKINETICS (PK) | 18 |
| g | 9.1 | Definition of variables | 18 |
| g | 9.2 | Biostatistical methods | 19 |
| 10 | . 1 | PHARMACODYNAMICS (Efficacy) | 22 |
| - | 10.1 | Definition of variables | 22 |
| 2 | 10.2 | Biostatistical methods | 22 |
| 11. | | SAFETY | 23 |
| - | 11.1 | Adverse Events | 23 |
| 2 | l1.2 | Safety Laboratory Assessments | 24 |
| 2 | 11.3 | Vital Signs Measurements | 26 |
| 2 | L1.4 | 12 - Lead Electrocardiogram (EKG) | 27 |
| 2 | 11.5 | Physical Examinations | 27 |
| 2 | 11.6 | Outcome Prediction Models | 27 |
| - | L1.7 | Concomitant Medications | 28 |
| - | 11.8 | Other safety evaluations | 28 |
| 12 | . 1 | IMMUNOGENICITY ENDPOINTS | 30 |

| 13. | EXPLORATORY ENDPOINTS | . 31 |
|------------|---------------------------------|------|
| 14. | HANDLING OF MISSING DATA | . 32 |
| 15. | CHANGES TO THE PLANNED ANALYSIS | . 33 |
| 15.3 | I Final Analysis (End of Study) | 34 |
| 16. | SOFTWARE | . 35 |
| <i>17.</i> | TABLES | 36 |
| 18. | LISTINGS | 39 |
| 19. | FIGURES | 42 |
| 20. | APPENDICES | . 43 |
| 21. | REFERENCES | . 44 |


# **List of Abbreviations**

| Abbreviation | Description |
|---|---|
| AUC <sub>0-t</sub> | The area under the plasma concentration-time curve, from time 0 (time of dosing) to the last time point with measurable analyte concentration, calculated by the log down, linear up trapezoidal method. |
| AE | Adverse Event |
| ATC | Anatomical Therapeutic Class |
| AUC <sub>0-inf</sub> | The area under the plasma concentration-time curve from time 0 extrapolated to infinity. $AUC_{0-inf}$ is calculated as the sum of $AUC_{0-t}$ plus the ratio of the last measurable plasma concentration to the elimination rate constant ( $k_{el}$ ). |
| AUC <sub>0-8</sub> | The area under the plasma concentration-time curve, from time 0 (time of dosing) to the 8 hours concentration, calculated by the log down, linear up trapezoidal method. |
| BLQ | Below the quantitation limit |
| CAP | Community-Acquired Pneumonia |
| CBC | Complete Blood Count |
| C <sub>max</sub> | Maximum observed concentration |
| C <sub>min</sub> | Minimum observed concentration over the dosing interval. |
| CL/F | Apparent clearance calculated as Dose/AUC <sub>0-inf</sub> . |
| CS | Clinically Significant |
| CSR | Clinical Study Report |
| CV | Coefficient of variation |
| DLT | Dose Limiting Toxicity |
| DN_AUC <sub>0-inf</sub> | Dose-normalized AUC <sub>0-inf</sub> , calculated as AUC <sub>0-inf</sub> divided by dose. |
| DN_AUC <sub>0-t</sub> | Dose-normalized AUC <sub>0-t</sub> , calculated as AUC <sub>0-t</sub> divided by dose. |
| DN_AUC <sub>0-8</sub> | Dose-normalized AUC <sub>0-8</sub> , calculated as AUC <sub>0-8</sub> divided by dose. |
| DN_C <sub>max</sub> | Dose-normalized $C_{\text{max}}$ , calculated as $C_{\text{max}}$ divided by dose. |
| EKG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EOS | End of Study |
| GCP | Good Clinical Practice |
| geo CV | Geometric Coefficient of Variation |
| HIV | Human Immunodeficiency Virus |
| ITT | Intention-to-treat |
| IV | Intravenous |
| IWRS | Interactive web response system |
| k <sub>el</sub> | Apparent terminal elimination rate constant, calculated by linear regression of the terminal linear portion of the log concentration vs. time curve. |
| LLQ | Lower Limit of Quantification |
| MAD | Multiple-Ascending Dose |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMSE | Mini-Mental State Exam |
| N/A | Not Applicable |
| NCS | Not Clinically Significant |

Protocol Number: BT-201 Document status: Final SAP Version 2.0 Amendment 1.0

| Abbreviation | Description |
|---|---|
| NK | Not Known |
| PE | Physical Examination |
| PI | Principal Investigator |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PSI | Pneumonia Severity Index |
| PT | Preferred Term |
| rhu-pGSN | Recombinant human plasma Gelsolin |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Single Dose |
| SD* | Standard Deviation |
| S.I. | International System of Units |
| SOC* | Standard of Care |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| t <sub>1/2</sub> | Apparent elimination half-life, calculated as ln(2)/k <sub>e</sub> l. |
| TEAE | Treatment Emergent Adverse Event |
| T <sub>max</sub> | Time to maximum observed drug concentration. If the maximum value occurs at more than one time point, $T_{\text{max}}$ is defined as the first time point with this value. |
| V <sub>z</sub> /F | Apparent volume of distribution at the terminal phase, calculated as Dose/ $(k_{el} \times AUC_{0-inf})$ . |
| WHO-DD | World Health Organization Drug Dictionary |


#### 1. INTRODUCTION

The following Statistical Analysis Plan (SAP) provides the outline for the statistical analysis of the data from the BT-201 study.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post hoc, or unplanned, exploratory analyses performed will be clearly identified as such in the final CSR.


#### 2. PROJECT OVERVIEW

## 2.1 Study Design

Study BTI-201 is a Phase 1b/2a, double-blind, placebo-controlled, dose-escalation study to evaluate the safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) of recombinant human plasma gelsolin (rhu-pGSN) added to standard of care (SOC\*) in subjects hospitalized for acute community-acquired pneumonia (CAP). Each dosing cohort will include 8 subjects randomized 3:1 rhu-pGSN:placebo (6 rhu-pGSN subjects:2 placebo subjects).

There will be 1 single dose cohort (Cohort 1) and 3 multiple dose cohorts (Cohorts 2, 3 and 4).

Dose will be based on actual body weight. Dose escalation will involve 3 dose levels of rhupGSN (6, 12, and 24 mg/kg) in patients admitted for CAP. Dose escalation will only occur after post-therapy safety information on all subjects in the prior cohort has been reviewed at Day 7 for the single-dose (SD) and multiple-ascending dose (MAD\*) arms.

The MAD portion of the study will commence once single doses of 6 mg/kg of rhu-pGSN are shown to be acceptably safe. The first 2 doses must be administered in the hospital, but the third dose can be given in a monitored outpatient setting where appropriate.

Discharged subjects will return for follow-up 7 days after the initiation of therapy (Day 7) and on Day 28 for the End-of-Study (EOS) Visit.

To assess safety and tolerability, subjects will undergo physical examinations (PE; including vital sign measurements), AE assessments, concomitant medication assessments, safety laboratory testing and Electrocardiogram (EKGs - completed locally), and other testing as per local custom.

#### 2.2 Objectives

## 2.2.1 Primary objective

The primary objective of the study will be to evaluate the safety and tolerability of single and multiple ascending doses of rhu-pGSN administered by once-daily intravenous (IV) push to hospitalized subjects with a primary admitting diagnosis of CAP.

## 2.2.2 Secondary objectives

The secondary objective of the study will be to characterize the PK profile of rhu-pGSN after single or multiple IV doses

#### 2.2.3 Exploratory objective.

The exploratory objectives of the study will be to investigate the following:

- To assess the quantitative relationship of pGSN levels at baseline with clinical outcomes, changes in prognostic indices and inflammatory biomarkers, and etiologic pathogen type.
- To assess the relationship between rhu-pGSN dose and clinical response and changes in surrogate biomarkers of efficacy.

# 2.2.4 Immunogenicity objective.

The immunogenicity objective of the study will be to investigate the post-treatment development of antibodies against rhu-pGSN by Day 28.


#### 2.3 Sample Size

The sample size of N=6 rhu-pGSN recipients per dose level and combined placebo in the SD and MAD portions of the trial were chosen based on limiting exposure to pGSN in this initial study in the current development program. The sample sizes in this trial have the following properties in relation to interpretation of Adverse Events (AEs) incidence rates (Table 1).

Table 1 presents the Minimum Sample Size such that there is 90% probability of observing at least 1 AE of a certain type if the TRUE underlying AE rate.

Table 1: Minimum Sample Size Calculations

| Sample Size | TRUE underlying AE rate |
|--------------------------|-------------------------|
| 6 (each pGSN dose level) | 32% |
| 8 (pooled placebo) | 21% |
| 24 (pooled pGSN) | 10% |

With each sample size presented in the table above, if zero AEs of a certain type are observed, one could be "90% confident" the TRUE underlying rate for that AE is at most the rate indicated above.

#### 2.4 Randomization

Following screening, subjects qualified for study entry will be randomized to receive rhupGSN or placebo during the treatment period. Randomization will be done centrally using the Interactive web response system (IWRS). All eligible subjects will be assigned a randomization number.

There will be 1 single dose cohort (Cohort 1) and 3 multiple dose cohorts (Cohorts 2, 3 and 4). Eight subjects will be sequentially randomized to each cohort for a total number randomized of 32 subjects.

Subjects will be randomized in a 3:1 ratio to rhu-pGSN or placebo (6 rhu-pGSN subjects:2 placebo subjects).

The investigational site team and the subject will be kept blinded to the treatment allocation of each participant. Only the designated pharmacist(s) will be unblinded to the treatment allocation. The unblinded pharmacist will utilize the IWRS system to randomly assign a treatment allocation. The treatment allocation will be available to the unblinded pharmacist(s).

03 December 2018

Protocol Number: BT-201


#### 3. STATISTICAL CONSIDERATIONS

Data will be handled and processed per the sponsor's representative (Novotech) Standard Operating Procedures (SOPs), which are written based on the principles of good clinical practice (GCP).

All data collected on the eCRFs will be presented in the data listings and will be listed and sorted by SD/MAD, treatment, subject number and visit, where applicable. All summaries will present the data by SD/MAD (apart from PK summaries), treatment group and overall (total subjects), as applicable. In addition, all placebo subjects will be combined into a single placebo group for purposes of summarizing the data.

• <u>Continuous variables</u>: Descriptive statistics will include the number of non-missing values (N), mean, standard deviation (SD\*), median, minimum, maximum.

The minimum and maximum values will be displayed to the same decimal precision as the source data, the arithmetic mean, SD\* and median values will be displayed to one more decimal than the source data for the specific variable.

The appropriate precision for derived variables will be determined based on the precision of the data on which the derivations are based, and statistics will be presented in accordance with the abovementioned rules.

- <u>PK data</u>: For PK data the arithmetic mean, standard deviation, median, minimum, maximum, coefficient of variation (CV%), geometric mean and geometric coefficient of variation (geo CV%) values will be presented. For the ratio of concentration data to the (within 30 minutes) pre-dose concentration on Day 1, the ln(SD\*) will also be presented.
- <u>Categorical variables</u>: Descriptive statistics will include frequency counts and percentages per category. Percentages will be rounded to one decimal place, with the denominator being the number of subjects in the relevant population with non-missing data, unless otherwise specified.
- <u>Time to Event Analysis</u>: Through the Kaplan-Meier method, nonparametric estimates of the survivor function will be represented by quartile estimates (Q1, Median and Q3) along with 95 Cls. Product limit estimates will be presented as part of appendices to the study outputs (SAS output).
- Imputation: No missing data will be imputed.
- <u>Baseline</u>: Baseline values will be defined as the last valid, non-missing observation for each subject prior to the first dose of study medication. For the PK analysis, baseline will be defined as the pre-dose value for each study day.
- <u>Repeat assessments (Safety)</u>: No repeat assessments will be included in summary presentations (Tables, Figures). Only the original values will be used in summary presentations. All repeat assessments captured in the Electronic Data Capture (EDC) system will be presented in the data listings.
- Assessment windows: All assessments will be included in the data listings and no visit windows will be applied to exclude assessments that were performed outside of the protocol specified procedure windows.
- <u>Date and time display conventions:</u> The following display conventions will be applied in all outputs where dates and/or times are displayed:

o Date only: DDMMMYYYY

o Date and time: DDMMMYYYY /HH:MM


If only partial information is available, unknown components of the date or time will be presented as 'NK' (not known), i.e., '2016-NK-NK'. Times will be reported in military time.

In the summary tables and figures, treatment groups will be summarized separately for SD/MAD, each cohort, combined placebo and overall (all subjects). Study outcomes will be summarized as follows:

- For each active dose level (overall):
  - o SD Phase:
    - rhu-pGSN 6 mg/kg
    - Placebo
    - Overall
  - o MAD Phase
    - rhu-pGSN 6 mg/kg
    - rhu-pGSN 12 mg/kg
    - rhu-pGSN 24 mg/kg
    - Combined Active
    - Combined Placebo
    - Overall


#### 4. ANALYSIS POPULATIONS

In this study, four analysis populations are defined: Intention-to-treat (ITT), Safety, Pharmacokinetic and the Per Protocol populations (PP).

Furthermore, any additional exploratory analysis not identified in the SAP will be identified in the final CSR as exploratory post hoc analyses. This may include the addition of additional study populations or subgroups of interest.

The number and percentage of subjects in each analysis population will be summarized.

#### 4.1 Population Descriptions

#### 4.1.1 Intention-to-treat (ITT) population

The ITT population will be defined as all randomized subjects. Subjects will be analyzed per the randomized treatment they received if different from the actual treatment received.

All disposition, demographic and pharmacodynamic (PD) analyses will be based on the ITT population. All listings will be presented by the ITT population.

## 4.1.2 Safety population

The safety population will be defined as all enrolled subjects who received at least one dose of the study drug and will be based on actual treatment received.

If the safety population differs from the ITT population in that subjects received a different treatment to that they were randomized, or did not receive treatment whatsoever after randomization, the demographic and pharmacodynamic analyses will be repeated for the safety population.

All safety analyses will be based on the safety population.

## 4.1.3 Pharmacokinetic (PK) population

The PK population will comprise all subjects in the safety population who provide adequate PK samples to calculate the PK parameters. Subjects with important protocol deviations will be assessed on a subject-by-subject basis for inclusion in the PK Population. The PK analysis will be conducted using the Pharmacokinetic population.

## 4.1.4 Per Protocol (PP) population

The PP population will comprise all subjects in the safety population excluding subjects who missed doses and/or randomly discontinued the study before the primary Day 7 Visit. Furthermore, subject that had any relevant important protocol deviations will be excluded from the PP population.

03 December 2018

Protocol Number: BT-201


#### 5. PROTOCOL DEVIATIONS

In case protocol deviations/violations are reported, all protocol deviations/violations will be listed for each subject in the by-subject data listings. Prior to database lock and during the blinded review of database, all protocol deviations/violations will be reviewed and assigned a status of important or not.

Important protocol deviations/violations may include the following, depending on the timing and nature of the deviation:

- INFORMED CONSENT DEVIATION: Subject not consented prior to study procedures being performed or subject not re-consented to study at next scheduled study visit following local approval of an updated PIS-CF.
- ENTRY DEVIATION: Subject enrolled in violation of eligibility criteria.
- WITHDRAWAL DEVIATION: Subject developed withdrawal criteria during the study, but were not withdrawn.
- DOSING DEVIATION: Subject received the wrong treatment or incorrect dose of investigational product or comparator; Subject received treatment at incorrect timepoint in study; Subject received treatment that had not been stored per protocol.
- OPERATIONAL DEVIATION: Informed consent deviations (other than consent not being obtained prior to study entry, which would be considered an Entry Deviation), IRB/IEC expired approval, significant visit window deviations, or other issues that may significantly impact subject safety or data integrity.


#### 6. SUBJECT DISPOSITION

Outcomes will be summarized by the treatment groups as specified in section 3.

## 6.1.1 Subject disposition

Subject disposition will be summarized using counts and percentages and will be based on the ITT Population. The number of screened subjects, number and percentage of randomized subjects, subjects discontinued from the study as well as the primary reason for discontinuation will also be summarized.

All disposition information collected will be listed together with the date that the subject provided informed consent and the date and time of the first study drug administration.

If the there is a difference between the ITT, Safety populations or the PP population, the disposition summary tables will be repeated for that population.

## 6.1.2 Analysis Populations

The number of subjects included in of each of the defined analysis populations will be summarized using counts and percentages and will be based on the ITT Population.

In addition, the inclusion/exclusion of each subject into/from each of the defined analysis populations will be listed.


#### 7. DEMOGRAPHIC AND BASELINE INFORMATION

Demographic and baseline body measurements will be summarized using the ITT Population and may be repeated for the safety population and per protocol populations if different from the ITT population.

All information will be presented by the treatment groups as specified in section 3.

## 7.1 Demographics

#### 7.1.1 Definition of variables

- Age (years);
- Sex;
- Child Bearing Potential;
- Method of Birth Control;
- Race;
- Height (cm);
- Weight (kg);

#### 7.1.2 Biostatistical methods

Quantitative and categorical summaries will be presented for demographic variables at the screening visit.

A by-subject data listing for demographic and baseline characteristics will be generated.

#### 7.2 Medical history

Past medical history will be coded using the Medical Dictionary for Regulatory Activities, (MedDRA - latest version), and will be presented in the by-subject data listings including the MedDRA codes.

## 7.3 Pregnancy Test (Serum and Urine)

Pregnancy test results will be included in the by-subject data listings. This includes the pregnancy test results at Screening and Day 28/End of Study.

## 7.4 Serology

The following viral detection results (serologies) at Screening will be listed for each subject when available: Hepatitis B, Hepatitis C and HIV status.

## 7.5 Other baseline characteristics

Confirmation of CAP (both clinical and radiographic) will be presented in the by-subject data listings.


## 8. STUDY DRUG ADMINISTRATION

Study drug administration results will be presented using the ITT Population.

A by-subject data listing will be generated for study medication administration. These listings will include randomized dose assignment, Date/Time of Injection, Study Drug Administered (mL), duration of administrations, reason whole study drug dose was not administered, injection interruptions, re-start and reason for any interruptions. Subjects who receive the wrong IP (rhu-pGSN vs. placebo) will be flagged.


#### 9. PHARMACOKINETICS (PK)

All PK summary tables and figures will be based on the PK Population. All listings will be based on the Safety Population (Actual Treatment). All analyses will be done by treatment group.

For the 1 dose in the SD arm and the first 2 doses in the MAD arms, blood will be drawn within 30 minutes pre-dose, and 5-10 minutes after the end of administration, as well as 2, 8, 12 and/or 16, and 24 hours after the end of administration (± 30 minutes) for analysis. Identical PK sampling is encouraged on Day 3 where feasible (but not required) in the multiple-dose arms.

In this section (section 9):

- The rhu-pGSN treatment group will be referred to the Active treatment group.
- Exogenous pGSN concentrations will be referred to as rhu-pGSN concentrations.
- Endogenous pGSN + Exogenous pGSN (total) will be referred to as pGSN

#### 9.1 Definition of variables

The following PK parameters for pGSN will be estimated For Day 1(SD/MAD), Day 2 (MAD) and Day 3 (MAD). PK Parameters will only be calculated for the Active (rhu-pGSN) treatment group. No PK parameters will be calculated for the Placebo treatment group:

Day 1: SD/MAD & Day 2/3: MAD

| AUC <sub>0-t</sub> | The area under the plasma concentration-time curve, from time 0 (time of dosing) to the last time point (24 hours) with measurable analyte concentration, calculated by the log down, linear up trapezoidal method. $AUC_{0t} \text{ will additionally be calculated for the estimated rhu-pGSN profile for both the change from pre-dose on each study day and the double-delta method.}$ |
|---|---|
| AUC <sub>0-8</sub> | The area under the plasma concentration-time curve, from time 0 (time of dosing) to the 8 hours concentration, calculated by the log down, linear up trapezoidal method. |
| | AUC <sub>0-8</sub> will additionally be calculated for the estimated rhu-pGSN profile for both the change from pre-dose on each study day and the double-delta method. |
| AUC <sub>0-inf</sub> | The area under the plasma concentration-time curve from time 0 extrapolated to infinity. AUC $_{0\text{-inf}}$ is calculated as the sum of AUC $_{0\text{-t}}$ plus the ratio of the last measurable plasma concentration to the elimination rate constant ( $k_{el}$ ). |
| C <sub>max</sub> | Maximum observed concentration. |
| | C <sub>max</sub> will additionally be calculated for the estimated rhu-pGSN profile for both the change from pre-dose on each study day and the double-delta method. |
| T <sub>max</sub> | Time to maximum observed drug concentration. If the maximum value occurs at more than one time point, $T_{\text{max}}$ is defined as the first time point with this value. |


| <b>k</b> el | Apparent terminal elimination rate constant calculated by linear regression of the terminal linear portion of the log concentration vs. time curve. |
|---|---|
| t <sub>1/2</sub> | Apparent elimination half-life, calculated as In(2)/kel |
| %AUC <sub>ext</sub> | Percentage of the extrapolated area under the plasma concentration-time curve, calculated as 100% * [AUC0-inf - AUC0-t]/ AUC0-inf |
| C <sub>L</sub> /F | Apparent clearance calculated as Dose/AUC <sub>0-inf</sub> . |
| V <sub>z</sub> /F | Apparent volume of distribution at the terminal phase, calculated as Dose/ $(k_{\text{el}} \times AUC_{0\text{-inf}})$ . |
| DN_C <sub>max</sub> | Dose-normalized $C_{\text{max}}$ , calculated as $C_{\text{max}}$ divided by dose DN_ $C_{\text{max}}$ will additionally be calculated for the estimated rhu-pGSN profile for both the change from pre-dose day 1 and the double-delta method |
| DN_AUC <sub>0-inf</sub> | Dose-normalized AUC <sub>0-inf</sub> , calculated as AUC <sub>0-inf</sub> divided by dose |
| DN_AUC <sub>0-t</sub> | Dose-normalized AUC <sub>0-t</sub> , calculated as AUC <sub>0-t</sub> divided by dose DN_AUC <sub>0-t</sub> will additionally be calculated for the estimated rhu-pGSN profile for both the change from pre-dose on each study day and the double-delta method. |
| DN_AUC <sub>0-8</sub> | Dose-normalized AUC $_{0-24}$ , calculated as AUC $_{0-24}$ divided by dose DN_AUC $_{0-8}$ will additionally be calculated for the estimated rhu-pGSN profile for both the change from pre-dose on each study day and the double-delta method. |

## 9.2 Biostatistical methods

#### Plasma pGSN

Individual plasma pGSN concentrations will be summarized by nominal sampling time.

Plasma pGSN concentrations that are below the quantitation limit (BQL) will be set to 0 if before the first quantifiable concentration, and to ½ the lower level of quantification elsewhere for calculation of summary statistics for concentration data at each time point.

The actual blood sampling dates and times relative to dosing time will be listed by subject and nominal sampling time, with time deviations calculated for all subjects with available plasma concentration data, including subjects excluded from the PK Population.

Individual (for each subject) and mean plasma pGSN concentration over time will be displayed graphically in linear and semi-logarithmic plot of pGSN concentration versus time. The actual collection time will be used for individual plasma pGSN concentration curve and the nominal time will be used for plot of mean plasma pGSN concentration curve.

Plasma concentrations vs. time data will be analyzed using validated PK software (Phoenix WinNonlin version 6.3 or higher), by standard non-compartmental model. Actual collection time will be used in the calculation of plasma PK parameters. For the calculation of the PK parameters, all plasma concentrations that are BLQ prior to the first measurable


concentration will be set to  $\frac{1}{2}$  the lower level of quantification. The BLQ values that are between measurable concentrations will be set to  $\frac{1}{2}$  LLOQ. The BLQ values that occur at the end of the profile (after the last quantifiable concentration) will also be set to  $\frac{1}{2}$  the lower level of quantification.

#### Ratio of Plasma pGSN

For subjects that do not have quantifiable pre-dose concentration values on each day, the pre-dose value will be set to ½ lower limit of quantification (LLQ).

Individual plasma pGSN: Day 1, 2 and Day 3 pGSN concentration ratios from each day's predose will be summarized by nominal sampling time.

Plasma pGSN concentrations that are below the quantitation limit (BQL) will be set to ½ the lower level of quantification post dose for calculation of summary statistics for concentration ratio data at each time point.

## Ratio of Pre-dose and Placebo Adjusted Plasma pGSN

For the active treatment groups, plasma concentration of pGSN will further be evaluated (adjusted) in terms of the mean Placebo pGSN at each time point as well as the pre-dose (baseline value) for each study day:

- Pre-dose values on each study day will be presented as recorded;
- Pre-dose values on each study day that are BLQ will be set to ½ LLQ;
- Subsequent BLQ values (post the first quantifiable concentration on each day) will be set to ½ LLQ.
- Pre-dose and Placebo Adjusted Concentration
  - = (Active Treatment Group natural log Concentration on Day z at Time Point y Day z Pre-dose natural log Concentration) (Placebo Treatment Group natural log Concentration on Day z at Time Point y Placebo Day z Pre-dose natural log Concentration) [results will be back-transformed to the ratio of ratios scale.]

Baseline and Placebo corrected Individual plasma pGSN concentrations will be summarized by nominal sampling time.

#### Analysis of Estimated rhu-pGSN

This analysis will exclude the placebo treatment group:

- Pre-dose values on each study day will be presented as recorded;
- Pre-dose values on each study day that are BLQ will be set to ½ LLQ;
- Subsequent BLQ values (post the first quantifiable concentration on each day) will be set to ½ LLQ.
- Estimated rhu-pGSN concentration
  - = concentration on Day z at Time Point y Day z Pre-dose concentration

Individual estimated rhu-pGSN concentrations will be summarized by nominal sampling time. Geometric summary statistics will not be calculated for estimated rhu-pGSN concentrations, as these values could be lower than or equal to 0.

Estimated Individual (for each subject) and mean estimated plasma rhu-pGSN concentration over time will be displayed graphically in linear plots of estimated rhu-pGSN concentration versus time. The actual collection time will be used for individual estimated plasma rhu-pGSN concentration curve and the nominal time will be used for plot of mean estimated plasma rhu-pGSN concentration curve.


Estimated plasma concentrations vs. time data will be analyzed using SAS software. Actual collection time will be used in the calculation of plasma PK parameters. The following parameters (including dose normalized parameters) will be calculated for each study day:

- AUC<sub>0-t</sub>
- AUC<sub>0-8h</sub>
- C<sub>max</sub>

#### Double Delta Analysis of Estimated rhu-pGSN

- Pre-dose values on each study day will be presented as recorded;
- Pre-dose values on each study day that are BLQ will be set to ½ LLQ;
- Subsequent BLQ values (post the first quantifiable concentration on each day) will be set to ½ LLQ.
- Estimated rhu-pGSN will be calculated as follows:
  - = (Active Treatment Group Concentration on Day z at Time Point y Day z Pre-dose Concentration) (Mean Placebo Treatment Group Concentration on Day z at Time Point y Mean Placebo Day z Pre-dose Concentration)

Estimated rhu-pGSN concentrations will be summarized by nominal sampling time. Geometric summary statistics will not be calculated for estimated rhu-pGSN concentrations, as these values could be lower than or equal to 0.

Estimated Individual (for each subject) and mean estimated plasma rhu-pGSN concentration over time will be displayed graphically in linear plots of estimated rhu-pGSN concentration versus time. The nominal time will be used for individual estimated plasma rhu-pGSN concentration curve and the nominal time will be used for plot of mean estimated plasma rhu-pGSN concentration curve.

Estimated rhu-pGSN plasma concentrations vs. time data will be analyzed using SAS software. Nominal time will be used in the calculation of plasma PK parameters. The following parameters (including dose normalized parameters) will be calculated for each study day:

- AUC<sub>0-t</sub>
- AUC<sub>0-8h</sub>
- C<sub>max</sub>


## 10. PHARMACODYNAMICS (EFFICACY)

All PD summary tables, figures and listings will be based on the ITT Population. All analysis will be done by study part (SD/MAD) by each treatment group.

As a sensitivity analysis, the analysis will be repeated based on the PP population.

#### 10.1 Definition of variables

The following biomarkers will be analyzed:

- Procalcitonin;
- pGSN;
- TNFα;
- TGFβ;
- IL1β;
- IL1ra;
- IL2;
- IL4;
- IL6;
- IL10;
- IL17a.`

#### 10.2 Biostatistical methods

Biomarker will be summarized via counts and percentages of subjects for categorical variables, and by summary statistics for baseline, each observed time point, and ratio from baseline at each observed time point for continuous variables (as for the PK analysis with the exception of CV% and Geometric CV%) by treatment group and overall.


#### 11. SAFETY

Safety endpoints will be analyzed using the Safety Population. All information will be presented by study part, for each treatment group and overall.

#### 11.1 Adverse Events

#### 11.1.1 Definition of variables

- Adverse event (AE)
- Serious adverse event (SAE)
- Treatment emergent adverse event (TEAE)

AEs and SAEs are defined in the study protocol. TEAEs are defined as adverse events that occurred or worsened following the first administration of study medication. Adverse events that have missing onset dates will be considered treatment-emergent, unless the stop date is known to be prior to the first administration of the study medication.

#### 11.1.2 Biostatistical methods

All AEs will be coded using MedDRA.

All AE summaries will be restricted to TEAEs only. Summary tables will include the number of subjects (%) experiencing an event and the number of events. Subjects will be counted only once at each system organ class (SOC) and preferred term (PT) level of summary.

The TEAE summaries will include:

- TEAE summary by SOC and PT
- TEAE summary of serious events by SOC and PT
- TEAE summary of deaths by SOC and PT
- TEAE summary by severity (NCI-CTCAE) by SOC and PT
- TEAE summary by causality to Study Drug by SOC and PT
- TEAE summary by causality to Study Procedure by SOC and PT
- TEAE summary of events leading to treatment discontinuation (Drug withdrawn) by SOC and PT

All AEs will be listed and will include verbatim term, PT, SOC, treatment, severity, causality, seriousness, and action taken with regards to the study drug. Separate listings will be created for SAEs, deaths and events leading to treatment discontinuation (Drug withdrawn).

Overall survival (time to death in days) will be analyzed through Kaplan-Meier methods and censored at the time of the study exit visit. Date of death will be taken as the SAE end date for which the outcome is stated to be fatal. Overall survival (days) = Date of event outcome of death/ Date of study exit - Date of first study drug administration + 1.

03 December 2018

Protocol Number: BT-201


## 11.2 Safety Laboratory Assessments

Blood samples will be collected at the time points specified in the Schedule of Events (refer to the Protocol) to conduct Complete blood count (CBC), Coagulation and Comprehensive Metabolic Profile analyses.

#### 11.2.1 Definition of variables

The following tests will be performed within each of the specified test panels:

Complete blood count (CBC):

- Hematocrit (HCT);
- Hemoglobin (HGB);
- Red Blood Cells (RBC)
- White Blood Cells (WBC) with differential (including Eosinophils (EOS), Neutrophils (NEUT), Basophils (BASO), Lymphocytes (LYM) and Monocytes (MONO);
- Platelets (PLAT);
- Reticulocyte count

## Coagulation:

- Prothrombin Time (PT) / International Normalized Ratio (INR);
- Partial Thromboplastin Time (PTT).

Comprehensive Metabolic Profile:

- Albumin (ALB)
- Blood Urea Nitrogen (BUN)
- Creatinine (CREAT)
- C-Reactive Protein (CRP)
- Lactate Dehydrogenase (LDH)
- Creatine phosphokinase (CPK)
- Alanine Aminotransferase (ALT)
- Aspartate Aminotransferase (AST)
- Total Bilirubin (BILI)
- Alkaline Phosphatase (ALP)
- Amylase
- Lipase

#### 11.2.2 Biostatistical Methods

All laboratory data collected at scheduled and unscheduled visits will be included in the listings, but only results collected as scheduled visits will be included in the summary tables.

Results for individual parameters may be reported in different units depending on the analyzing laboratory. If required, the results (and the corresponding normal range cut-off values) for individual parameters may be converted to International System of Units (S.I.) units to summarize the data.


For the all parameters where a unit value has been reported, the parameter names that will be used in the outputs will comprise of the test name and the unit of measure, for example, 'Albumin (g/L)'. Parameters will be sorted alphabetically within tables and listings.

For all parameters where a normal range limit value is reported, the normal range will be derived based on the available lower and upper limit values and any reported mathematical symbols. If both a lower and upper limit value is available, the normal range will be presented as '(Lower, Upper)'.

The reported results for each parameter with a defined normal range will be classified ('Low', 'Normal', 'High') in relation to the defined normal range limits. If a result is equal to the normal range cut-off value, the result will be considered 'Normal'.

The change from baseline values at each post-baseline visit will be calculated for all parameters with continuous results (except for specific gravity and pH).

The decimal precision for each parameter will be based on the maximum number of decimals to which the reported result or the normal range limits are presented to in the raw data. The results and normal ranges will be displayed to the same decimal precision in the listings.

If a result for a parameter that is normally considered continuous is reported as a range (i.e., the result for basophils is reported as '<0.01' for a single time point), the result may be converted to a numeric value that is smaller than the reported result to contribute to the derivations and the summary statistics. Any conversion rules that are applied will be highlighted in the footnotes of the affected tables and listings. The original reported result value will however be included in the listing.

The laboratory result tables will present summary statistics for each laboratory parameter within the specific test panel. For each parameter, summaries will be presented for the baseline and each scheduled post-baseline visit. In addition, summaries will be presented for the change from baseline values at each scheduled post-baseline visit.

Additionally, counts (%) of number subjects with values out of normal range at each scheduled time point will also be presented along with shift tables that will represent the changes in normal range categories across post-baseline time points.

The listings of laboratory parameters will include all the information (fields) collected. In addition, the observations that are used as the baseline record (value) for each parameter will be flagged, and the change from baseline values at each post-baseline visit will be presented.

For all parameters, standardized values will be reported.


## 11.3 Vital Signs Measurements

#### 11.3.1 Definition of variables

The following vital signs measurements will be taken at the time points specified in the Schedule of Events (refer to the Protocol):

- Heart Rate (beats/min);
- Systolic blood pressure (SBP) (mmHg)
- Diastolic blood pressure (DBP) (mmHg)
- Respiratory rate (breaths/min)
- Temperature (°C)
- Pulse Oximetry (%)
- Overall Investigator Interpretation

#### 11.3.2 Biostatistical Methods

All vital signs data collected at scheduled and unscheduled visits will be included in the listings, but only results collected as scheduled visits will be included in the summary tables.

The parameter names that will be used in the outputs will comprise of the test name and the unit of measure, for example, 'Systolic Blood Pressure (mmHg)'. Parameters will be sorted in the order that the measurements were collected in on the Vital Signs eCRF page within the tables and listings.

The change from baseline to the pre-dose assessment at each post-baseline visit will be calculated for all parameters.

The decimal precision for each parameter will be based on the maximum number of decimals to which the results were reported on the eCRF.

Vital signs measurements will present summary statistics for the results at the baseline and each scheduled post-baseline visit for each of the parameters. In addition, summaries will be presented for the change from baseline values at each scheduled post-baseline visit.

The summary of overall interpretation results table will present counts and percentages for the reported results at baseline and each post-baseline visit/time point. Result categories will be ordered as 'Normal', 'Abnormal not clinical significant (NCS)' and 'Abnormal clinical significant (CS)'.

The listings of vital signs measurements will include all the information collected. In addition, the observations that are used as the baseline record (value) for each parameter will be flagged, and the change from baseline values at each post-baseline visit will be presented.


#### 11.4 12 - Lead Electrocardiogram (EKG)

#### 11.4.1 Definition of variables

The following EKG measurements will be taken at the time points specified in the Schedule of Events (refer to the Protocol):

- Heart Rate (beats/min);
- PR Interval (ms)
- QRS Interval (ms)
- QT Interval (sec)
- QTcF Interval (ms) = QT interval /cube root of the RR interval
- Overall Investigator Interpretation

#### 11.4.2 Biostatistical Methods

All EKG data collected at scheduled and unscheduled visits will be included in the listings, but only results collected as scheduled visits will be included in the summary tables.

The parameter names that will be used in the outputs will comprise of the test name and the unit of measure, for example, 'Heart Rate (beats/min)'. Parameters will be sorted in the order that the measurements were collected in on the EKG eCRF page within the tables and listings.

For study visits where, multiple EKG measurement are taken, the mean of the measurements will be summarized and the worst-case overall investigator interpretation for the multiple measurements will be presented.

The change from baseline to the pre-dose assessment at each post-baseline visit will be calculated for all parameters.

The decimal precision for each parameter will be based on the maximum number of decimals to which the results were reported on the eCRF.

EKG measurements will present summary statistics for the results at the baseline and each scheduled post-baseline visit for each of the parameters. In addition, summaries will be presented for the change from baseline values at each scheduled post-baseline visit.

The summary of overall interpretation results table will present counts and percentages for the reported results at baseline and each post-baseline visit/time point. Result categories will be ordered as 'Normal', 'Abnormal NCS' and 'Abnormal CS'.

The listings of EKG measurements will include all the information collected and calculated (mean results). In addition, the observations that are used as the baseline record (value) for each parameter will be flagged, and the change from baseline values at each post-baseline visit will be presented.

#### 11.5 Physical Examinations

Physical Examination assessments will be listed for all time points.

#### 11.6 Outcome Prediction Models

#### 11.6.1 Definition of variables

The following outcome prediction models will be taken at the time points specified in the Schedule of Events (refer to the Protocol):

CURB-65 Score;


- Pneumonia Severity Index (PSI) Score
- Pneumonia Severity Index (PSI) Risk Class
- SOFA Score
- Mini-Mental State Exam (MMSE) Score

## 11.6.2 Biostatistical Methods

All outcome prediction model data collected at scheduled and unscheduled visits will be included in the listings, but only results collected as scheduled visits will be included in the summary tables.

The change from baseline to the pre-dose assessment at each post-baseline visit will be calculated for all parameters.

The decimal precision for each parameter will be based on the maximum number of decimals to which the results were reported on the eCRF.

Outcome prediction model scores will present summary statistics for the results at the baseline and each scheduled post-baseline visit for each of the parameters. In addition, summaries will be presented for the change from baseline values at each scheduled post-baseline visit.

The summary of PSI Risk Class will present counts and percentages for the reported results at baseline and each post-baseline visit/time point. Result categories will be ordered by risk class.

The listings of outcome prediction model data will include all the information collected. In addition, the observations that are used as the baseline record (value) for each parameter will be flagged, and the change from baseline values at each post-baseline visit will be presented.

#### 11.7 Concomitant Medications

Concomitant and prior medications will be coded using World Health Organization Drug Dictionary (WHO-DD, September 2015).

Prior medications are defined as any medication where the use was stopped prior to the first administration of the study medication. Prior medications will be listed only.

Concomitant medications are defined as any medication (other than the study drug) that was used at least once after the first administration of the study medication. Medications that were stopped on the same date as the first study drug infusion will be analyzed as concomitant medications. If a clear determination cannot be made (partial medication end dates) the medication will be classified as concomitant.

Concomitant medications will be summarized by WHO-DD Anatomical Therapeutic Chemical (ATC) class Level 3, and preferred term using frequency counts and percentages by study part and treatment group. Subjects who take the same medication more than once will be counted only once for that preferred term. Subjects will also only be counted once for each ATC3 class, regardless of the number of medications they have taken within that class

## 11.8 Other safety evaluations

Hospitalization follow-up will be presented in by-subject listings by study part and treatment group. Length of stay in hospital defined as date and time of discharge or date of study exit if still hospitalized at the time of death or study exit (censored at 23:59) - date and time of Hospitalization admission due to CAP in hours, length of ICU stay and the period of intubation in days will be listed and presented through Kaplan-Meier (K-M) methods.


The length of stay in ICU and period of intubation analysis will be restricted to subjects that stayed in the ICU and were intubated. The event investigated will be the cessation of ICU stay and the cessation of intubation.


# 12. IMMUNOGENICITY ENDPOINTS

All Immunogenicity endpoints will be listed using the safety population by study part and treatment. Specimens from placebo recipients will serve as a negative control.

Antibodies against rhu-pGSN will be blindly assayed from frozen specimens to determine whether the investigational product induces an antibody response in recipients.


# 13. EXPLORATORY ENDPOINTS

Other analyses to be performed include:

- Blood, sputum, and other cultures as clinically indicated (note that a sputum culture is mandatory if a sputum specimen can be obtained and blood cultures are strongly encouraged at entry into the study).
- Sputum neutrophil elastase (where feasible at entry and near the conclusion of study therapy).

Exploratory endpoints will be listed only.


# 14. HANDLING OF MISSING DATA

Missing, unused, or spurious data will be handling in the following manner:

- There will be no imputations or substitution made for missing PD or safety data points;
- For the PK analyses, imputations will be made for missing data points. Please see section 9 for more detail.


# 15. CHANGES TO THE PLANNED ANALYSIS

No planned changes.


# 15.1 Final Analysis (End of Study)

The final analysis will be conducted after all subjects have completed the study, the clinical database has been locked and the analysis populations have been approved.

The final analysis will be based on the final version of the SAP. Any deviations from the planned analysis will be documented in the CSR.


# 16. SOFTWARE

The following software will be used to perform the statistical analyses:

- SAS® Version 9.4 or higher (SAS Institute, Cary, North Carolina, USA).
- The following software will be used to perform the PK analysis: Phoenix WinNonlin® version 6.3 or higher.

# 17. TABLES

| No. | Title | Analysis<br>Population |
|---|---|---|
| 14.1.1.1 | SD: Summary of Subject Enrolment and Disposition | Intent-to-Treat |
| 14.1.1.2 | MAD: Summary of Subject Enrolment and Disposition | Intent-to-Treat |
| 14.1.2.1 | SD: Summary of Demographics and Baseline Characteristics | Intent-to-Treat |
| 14.1.2.2 | MAD: Summary of Demographics and Baseline Characteristics | Intent-to-Treat |
| 14.2.1.1 | Day 1: Summary of Plasma pGSN Concentrations (unit) by Timepoint | PK |
| 14.2.1.2 | Day 2: Summary of Plasma pGSN Concentrations (unit) by Timepoint | PK |
| 14.2.1.3 | Day 3: Summary of Plasma pGSN Concentrations (unit) by Timepoint | PK |
| 14.2.1.4 | Day 1: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint | PK |
| 14.2.1.5 | Day 2: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint | PK |
| 14.2.1.6 | Day 3: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint | PK |
| 14.2.2.1 | Day 1: Summary of Plasma pGSN PK Parameters | PK |
| 14.2.2.2 | Day 2: Summary of Plasma pGSN PK Parameters | PK |
| 14.2.2.3 | Day 3: Summary of Plasma pGSN PK Parameters | PK |
| 14.2.3.1 | Day 1: Summary of Estimated Plasma rhu-pGSN PK Parameters | PK |
| 14.2.3.2 | Day 2: Summary of Estimated Plasma rhu-pGSN PK Parameters | PK |
| 14.2.3.3 | Day 3: Summary of Estimated Plasma rhu-pGSN PK Parameters | PK |
| 14.2.4.1 | SD: Summary of PD Parameters | Intent-to-Treat |
| 14.2.4.2 | MAD: Summary of PD Parameters | Intent-to-Treat |
| 14.2.5.1 | SD: Summary of PD Parameters | Per Protocol |
| 14.2.5.2 | MAD: Summary of PD Parameters | Per Protocol |
| 14.3.1.1 | SD: Summary of Concomitant Medication | Safety |
| 14.3.1.2 | MAD: Summary of Prior and Concomitant Medication | Safety |
| 14.3.3.1.1 | SD: Overall Summary of Treatment-Emergent Adverse Events | Safety |
| 14.3.3.1.2 | MAD: Overall Summary of Treatment-Emergent Adverse Events | Safety |
| 14.3.3.2.1 | SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT) | Safety |
| 14.3.3.2.2 | MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT) | Safety |
| 14.3.3.3.1 | SD: Summary of Treatment-Emergent Deaths (Summary by SOC, PT) | Safety |
| 14.3.3.3.2 | MAD: Summary of Treatment-Emergent Deaths (Summary by SOC, PT) | Safety |
| (1 | - IT-L | A in a last |
|---|---|---|
| .02 | | Analysis<br>Population |
| | | r opulation |
| 14.3.3.4.1 | SD: Summary of Serious Treatment-Emergent Adverse Events (Summary by SOC, PT) | Safety |
| 14.3.3.4.2 | MAD: Summary of Serious Treatment-Emergent Adverse Events (Summary by SOC, PT) | Safety |
| 14.3.3.5.1 | SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and NCI-CTCAE Grade) | Safety |
| 14.3.3.5.2 | MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and NCI-CTCAE Grade) | Safety |
| 14.3.1.6.1 | SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study Drug) | Safety |
| 14.3.3.6.2 | MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study Drug) | Safety |
| 14.3.3.7.1 | SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study Procedure) | Safety |
| 14.3.3.7.2 | MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study Procedure) | Safety |
| 14.3.3.8.1 | SD: Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation (Summary by SOC, PT) | Safety |
| 14.3.3.8.2 | MAD: Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation (Summary by SOC, PT) | Safety |
| 14.3.3.9.1 | | Safety |
| 14.3.3.9.2 | MAD: Summary of Overall Survival | Safety |
| 14.3.4.1.1.1 | SD: Summary of CBC (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.1.1.2 | MAD: Summary of CBC (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.1.2.1 | SD: Summary of CBC Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.1.2.2 | MAD: Summary of CBC Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.2.1.1 | SD: Summary of Coagulation (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.2.1.2 | MAD: Summary of Coagulation (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.2.2.1 | SD: Summary of Coagulation Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.2.2.2 | MAD: Summary of Coagulation Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.3.1.1 | SD: Summary of Comprehesive Metabolic Profile (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.3.1.2 | MAD: Summary of Comprehesive Metabolic Profile (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.3.2.1 | SD: Summary of Comprehesive Metabolic Profile Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.3.2.2 | MAD: Summary of Comprehesive Metabolic Profile Shifts from Baseline (Low, Normal, High) | Safety |
| 14.3.4.4.1 | SD: Summary of Vital Signs (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.4.2 | MAD: Summary of Vital Signs (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.5.1 | SD: Summary of Vital Signs Interpretation by Timepoint | Safety |
| 14.3.4.5.2 | MAD: Summary of Vital Signs Interpretation by Timepoint | Safety |
| 14.3.4.6.1 | SD: Summary of Mean EKG (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.6.2 | MAD: Summary of Mean EKG (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |

| No. | Title | Analysis<br>Population |
|---|---|---|
| 14.3.4.7.1 | SD: Summary of EKG Interpretation (Worst) by Timepoint | Safety |
| 14.3.4.7.2 | MAD: Summary of EKG Interpretation (Worst) by Timepoint | Safety |
| 14.3.4.8.1 | SD: Summary of CURB-65 Score(Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.8.2 | MAD: Summary of CURB-65 Score (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.9.1 | SD: Summary of PSI Score (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.9.2 | MAD: Summary of PSI Score (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.10.1 | SD: Summary of PSI Risk Class by Timepoint | Safety |
| 14.3.4.10.2 | MAD: Summary of PSI Risk Class by Timepoint | Safety |
| 14.3.4.11.1 | SD: Summary of SOFA Score (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.11.2 | MAD: Summary of SOFA Score (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.12.1 | SD: Summary of MMSE Score (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.12.2 | MAD: Summary of MMSE Score (Summary of Actual and Change from Baseline Values) by Timepoint | Safety |
| 14.3.4.13.1 | SD: Summary of Hospitalization | Safety |
| 14.3.4.13.2 | MAD: Summary of Hospitalization | Safety |

Protocol Number: BT-201 Document status: Final SAP Version 2.0 Amendment 1.0

### 18. LISTINGS

| No. | Title | Analysis<br>Population |
|---|---|---|
| 16.2.1.2.1 | SD: Subject Disposition | Intent-to-Treat |
| 16.2.1.2.2 | MAD: Subject Disposition | Intent-to-Treat |
| 16.2.2.1 | SD: Protocol Deviations | Intent-to-Treat |
| 16.2.2.2 | MAD: Protocol Deviations | Intent-to-Treat |
| 16.2.3.1 | SD: Analysis Populations | Intent-to-Treat |
| 16.2.3.2 | MAD: Analysis Populations | Intent-to-Treat |
| 16.2.4.1.1 | SD: Demographics and Baseline Characteristics | Intent-to-Treat |
| 16.2.4.1.2 | MAD: Demographics and Baseline Characteristics | Intent-to-Treat |
| 16.2.4.2.1 | SD: Viral Serology | Intent-to-Treat |
| 16.2.4.2.2 | MAD: Viral Serology | Intent-to-Treat |
| 16.2.4.3.1 | SD: Medical History | Intent-to-Treat |
| 16.2.4.3.2 | MAD: Medical History | Intent-to-Treat |
| 16.2.4.4.1 | SD: Pregnancy Test Results | Intent-to-Treat |
| 16.2.4.4.2 | MAD: Pregnancy Test Results | Intent-to-Treat |
| 16.2.4.5.1 | SD: Confirmation of CAP | Intent-to-Treat |
| 16.2.4.5.2 | MAD: Confirmation of CAP | Intent-to-Treat |
| 16.2.4.6.1 | SD: Eligibility Assessment | Intent-to-Treat |
| 16.2.4.6.2 | MAD: Eligibility Criteria | Intent-to-Treat |
| 16.2.4.7.1 | SD: Prior Medications | Intent-to-Treat |
| 16.2.4.7.2 | MAD: Prior Medications | Intent-to-Treat |
| 16.2.5.1.1 | SD: Randomization | Intent-to-Treat |
| 16.2.5.1.2 | MAD: Randomization | Intent-to-Treat |
| 16.2.5.2.1 | SD: Study Drug Administration | Intent-to-Treat |
| 16.2.5.2.2 | MAD: Study Drug Administration | Intent-to-Treat |
| 16.2.5.3.1 | SD: Study Drug Interruption | Intent-to-Treat |
| 16.2.5.3.2 | MAD: Study Drug Interruption | Intent-to-Treat |
| 16.2.6.1.1 | SD: Individual pGSN Plasma Concentrations (unit) | Intent-to-Treat |

| | | 1 |
|---|---|---|
| No. | Title | Analysis |
| | | Population |
| 16.2.6.1.2 | MAD: Individual pGSN Plasma Concentrations (unit) | Intent-to-Treat |
| 16.2.6.2.1 | SD: Individual Estimated Plasma rhu-pGSN Concentrations (unit) | Intent-to-Treat |
| 16.2.6.2.2 | MAD: Individual Estimated Plasma rhu-pGSN Plasma Concentrations (unit) | Intent-to-Treat |
| 16.2.6.3.1 | SD: Individual pGSN Plasma PK Parameters | Intent-to-Treat |
| 16.2.6.3.2 | MAD: Individual pGSN Plasma PK Parameters by Day | Intent-to-Treat |
| 16.2.6.4.1 | SD: Individual Estimated Plasma rhu-pGSN Plasma PK Parameters | Intent-to-Treat |
| 16.2.6.4.2 | MAD: Individual Estimated Plasma rhu-pGSN Plasma PK Parameters by Day | Intent-to-Treat |
| 16.2.6.5.1 | SD: Anti-rhu-pGSN Antibodies | Intent-to-Treat |
| 16.2.6.5.2 | MAD: Anti-rhu-pGSN Antibodies | Intent-to-Treat |
| 16.2.6.6.1 | SD: Biomarkers | Intent-to-Treat |
| 16.2.6.6.2 | MAD: Biomarkers | Intent-to-Treat |
| 16.2.6.7.1 | SD: Sputum and Blood Culture | Intent-to-Treat |
| 16.2.6.7.2 | MAD: Sputum and Blood Culture | Intent-to-Treat |
| 16.2.7.1.1 | SD: Adverse Events | Intent-to-Treat |
| 16.2.7.1.2 | MAD: Adverse Events | Intent-to-Treat |
| 16.2.7.2.1 | SD: Serious Adverse Events | Intent-to-Treat |
| 16.2.7.2.2 | MAD: Serious Adverse Events | Intent-to-Treat |
| 16.2.7.3.1 | SD: Adverse Events Leading to Study Medication Discontinuation | Intent-to-Treat |
| 16.2.7.3.2 | MAD: Adverse Events Leading to Study Medication Discontinuation | Intent-to-Treat |
| 16.2.7.4.1 | SD: Overall Survival | Intent-to-Treat |
| 16.2.7.4.2 | MAD: Overall Survival | Intent-to-Treat |
| 16.2.8.1.1.1 | SD: CBC | Intent-to-Treat |
| 16.2.8.1.1.2 | MAD: CBC | Intent-to-Treat |
| 16.2.8.1.2.1 | SD: Abnormal CBC | Intent-to-Treat |
| 16.2.8.1.2.2 | MAD: Abnormal CBC | Intent-to-Treat |
| 16.2.8.2.1.1 | SD: Coagulation | Intent-to-Treat |
| 16.2.8.2.1.2 | MAD: Coagulation | Intent-to-Treat |
| 16.2.8.2.2.1 | SD: Abnormal Coagulation | Intent-to-Treat |
| 16.2.8.2.2.2 | $\overline{}$ | Intent-to-Treat |
| 16.2.8.3.1.1 | $\overline{}$ | Intent-to-Treat |
| 16.2.8.3.1.2 | MAD: Comprehensive Metabolic Profile | Intent-to-Treat |

Novotech - Strictly Confidential

| No. | Title | Analysis<br>Population |
|---|---|---|
| 16.2.8.3.2.1 | SD: Abnormal Comprehensive Metabolic Profile | Intent-to-Treat |
| 16.2.8.3.2.2 | MAD: Abnormal Comprehensive Metabolic Profile | Intent-to-Treat |
| 16.2.9.1 | SD: Vital Signs | Intent-to-Treat |
| 16.2.9.2 | MAD: Vital Signs | Intent-to-Treat |
| 16.2.10.1 | SD: EKG | Intent-to-Treat |
| 16.2.10.2 | MAD: EKG | Intent-to-Treat |
| 16.2.11.1 | SD: Physical Examination | Intent-to-Treat |
| 16.2.11.2 | MAD: Physical Examination | Intent-to-Treat |
| 16.2.12.1.1 | SD: Outcome Prediction Models CURB-65 | Intent-to-Treat |
| 16.2.12.1.2 | MAD: Outcome Prediction Models CURB-65 | Intent-to-Treat |
| 16.2.12.2.1 | SD: Outcome Prediction Models PSI (Port Score) | Intent-to-Treat |
| 16.2.12.2.2 | MAD: Outcome Prediction Models PSI (Port Score) | Intent-to-Treat |
| 16.2.12.3.1 | SD: Outcome Prediction Models SOFA Score | Intent-to-Treat |
| 16.2.12.3.2 | MAD: Outcome Prediction Models SOFA Score | Intent-to-Treat |
| 16.2.12.4.1 | SD: Outcome Prediction Models MMSE Score | Intent-to-Treat |
| 16.2.12.4.2 | MAD: Outcome Prediction Models MMSE Score | Intent-to-Treat |
| 16.2.13.1 | SD: Concomitant Medications | Intent-to-Treat |
| 16.2.13.2 | MAD: Concomitant Medication | Intent-to-Treat |
| 16.2.14.1 | SD: Hospitalization Follow-Up | Intent-to-Treat |
| 16.2.14.2 | MAD: Hospitalization Follow-Up | Intent-to-Treat |

## 19. FIGURES

| No. | Title | Analysis<br>Population |
|---|---|---|
| 14.2.1.1 | Individual pGSN Plasma Concentrations (ng/mL) (Linear scale) by Day | PK |
| 14.2.1.2 | Individual pGSN Plasma Concentrations (ng/mL) (Semi-logarithmic) by Day | PK |
| 14.2.2.1 | ual Estimated Plasma rhu-pGSN F | PK |
| | by Day | |
| 14.2.2.2 | Individual Estimated Plasma rhu-pGSN Plasma Concentrations (ng/mL) based on the Double Delta Analysis (Linear scale) | PK |
| | by Day | |
| 14.2.3.1 | Mean (+/-SD) pGSN Plasma Concentrations (ng/mL) (Linear scale) by Day | PK |
| 14.2.3.2 | Mean (+/-SD) pGSN Plasma Concentrations (ng/mL) based on Changes from Pre-Injection (Linear scale) by Day (Semi- | PK |
| | logarithmic) by Day | |
| 14.2.4.1 | Mean (+/-SD) Estimated Plasma rhu-pGSN Plasma Concentrations (ng/mL) based on Changes from Pre-Injection (Linear | PK |
| | scale) by Day | |
| 14.2.4.2 | Mean (+/-SD) Estimated Plasma rhu-pGSN Plasma Concentrations (ng/mL) based on the Double Delta Analysis (Linear | PK |
| | scale) by Day | |
| 14.3.1.1 | SD: Kaplan-Meier Plot of Overall Survival Time | Safety |
| 14.3.1.2 | MAD: Kaplan-Meier Plot of Overall Survival Time | Safety |
| 14.3.2.1 | SD: Kaplan-Meier Plot of Length of Stay in Hospital (hours) | Safety |
| 14.3.2.2 | MAD: Kaplan-Meier Plot of Length of Stay in Hospital (hours) | Safety |
| 14.3.3.1 | SD: Kaplan-Meier Plot of Duration of ICU Stay | Safety |
| 14.3.3.2 | MAD: Kaplan-Meier Plot of Duration of ICU Stay | Safety |
| 14.3.4.1 | SD: Kaplan-Meier Plot of Duration of Intubation | Safety |
| 14.3.4.2 | MAD: Kaplan-Meier Plot of Duration of Intubation | Safety |

## 20. APPENDICES

| No. | Title | Analysis<br>Population |
|---|---|---|
| 14.3.3.9.1 | 14.3.3.9.1 SD: Summary of Overall Survival | Safety |
| 14.3.3.9.2 | 14.3.3.9.2 MAD: Summary of Overall Survival | Safety |
| 14.3.4.13.1 | 14.3.4.13.1 SD: Summary of Hospitalization | Safety |
| 14.3.4.13.2 | 14.3.4.13.2 MAD: Summary of Hospitalization | Safety |

Protocol Number: BT-201 03 December 2018


#### 21. REFERENCES

1) Clinical Study Protocol Amendment 1.0, 30 April 2018.

# **BTI-201: Mock Tables: Table of Contents**

### Tables

| Table 14.1.1.1 SD: Summary of Subject Enrolment and Disposition | 9 |
|---|---|
| y of | / |
| Table 14.1.2.1 SD: Summary of Demographics and Baseline Characteristics | $\infty$ |
| : Summary of Demographics | 0 |
| Table 14.2.1.1 Day 1: Summary of Plasma pGSN Concentrations (unit) by Timepoint | $\vdash$ |
| 2: Summary of Plasma pGSN Concentrations (unit) | 3 |
| 3: Summary of Plasma | 5 |
| Table 14.2.1.4 Day 1: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint | 9 |
| Table 14.2.1.5 Day 2: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint | ∞ |
| Table 14.2.1.6 Day 3: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint | 0 |
| Day 1: Summary of Plasma | 7. |
| e 14.2.2.2 Day 2: Summary of Plasma | 7 |
| Day 3: Summary of Plasma | 33 |
| Table 14.2.3.1 Day 1: Summary of Estimated Plasma rhu-pGSN PK Parameters | 4 |
| Table 14.2.3.2 Day 2: Summary of Estimated Plasma rhu-pGSN PK Parameters | Ď. |
| Table 14.2.3.3 Day 3: Summary of Estimated Plasma rhu-pGSN PK Parameters | 9 |
| Table 14.2.4.1 SD: Summary of PD Parameters | 7 |
| Table 14.2.4.2 MAD: Summary of PD Parameters | ∞. |
| SD: | 6 |
| .5.2 MAD: Summary of PD Parameters | 30 |
| of Concomitant Medication | 31 |
| e 14.3.1.2 MAD: Summary of Prior and Concomitant Medication | 32 |
| .1.1 SD: Overall Summary of Treatment-Emergent Adverse Events | 33 |
| Overall Summary of Treatment-Emergent Adverse Events | 34 |
| e 14.3.3.2.1 SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT) | 35 |
| y of Treatment-Emergent Adverse Events (Summary by SOC, PT) | 36 |
| of Treatment-Emergent Deaths (Summary by SOC, PT) | 37 |
| of Treatment-Emergent Deaths (Summary by SOC, PT) | 38 |
| Table 14.3.3.4.1 SD: Summary of Serious Treatment-Emergent Adverse Events (Summary by SOC, PT) | 6 |
| f Serious Treatment-Emergent Adverse Events (Summary by SOC, PT) | 40 |
| Table 14.3.3.5.1 SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and NCI-CTCAE Grade) | 41 |
| Table 14.3.3.5.2 MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and NCI-CTCAE Grade) | 12 |
| Table 14.3.1.6.1 SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study Drug) | 13 |
| able 14.3.3.6.2 MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study | 4 |
| Table 14.3.3.7.1 SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study Procedure) | _ ı |
| | 45 |

| Table 14.3.3.7.2 MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study | - |
|---|---|
| TIOCEGUIE).<br>Table 14.3.3.8.1 SD: Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation (Summary by SOC,<br>PT) | : 4 |
| Table 14.3.3.8.2 MAD: Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation (Summary by SOC<br>PT) | : 4 |
| Table 14.3.3.9.1 SD: Summary of Overall Survival | . 4 |
| e 14.3.3.9.2 MAD: Summary of Overall | . 5 |
| e 14.3.4.1.1.1 SD: | .5 |
| e 14.3.4.1.1.2 MAD: Summary of CBC | .5 |
| e 14.3.4.1.2.1 SD: Summary of CBC Shifts from Baseline (Low, Normal, E | 5 |
| Table 14.3.4.1.2.2 MAD: Summary of CBC Shifts from Baseline (Low, Normal, High) | . 5 |
| e 14.3.4.2.1.1 SD. Summary of Coaquiation (Summary of Actual and Change from Baseline Values) by 1<br>e 14.3.4.2.1.2 MAD: Summary of Coaquiation (Summary of Actual and Change from Baseline Values) by | : : |
| e 14.3.4.2.2.1 SD: Summary of Coagulation Shifts from Baseline (Low, Normal, High) | .5 |
| : Summary of Coaqulation Shifts from Baseline (Low, Normal, | . 55 |
| e 14.3.4.3.1.1 SD: Summary of Comprehensive Metabolic Profile (Summary of Actu | ì |
| Timepoint | رن<br>کیر |
| C 11.0.1.0.1.1 INTO COMMUNITY OF COMPTONIES OF COCCUS OF TAXABLE CONTROL OF COCCUS OF | . کر<br>: کر |
| Table 14.3.4.3.2.1 SD: Summary of Comprehensive Metabolic Profile Shifts from Baseline (Low, Normal, High) | . 6 |
| Table 14.3.4.3.2.2 MAD: Summary of Comprehensive Metabolic Profile Shifts from Baseline (Low, Normal, High) | 6 |
| Table 14.3.4.4.1 SD: Summary of Vital Signs (Summary of Actual and Change from Baseline Values) by Timepoint | 6 |
| Table 14.3.4.4.2 MAD: Summary of Vital Signs (Summary of Actual and Change from Baseline Values) by Timepoint | ·9 |
| e 14.3.4.5.1 SD: Summary of Vital Signs Interpretation by T | 6 |
| e 14.3.4.5.2 MAD: Summary of Vital Signs Interpretation by Timepoint | 6( |
| e 14.3.4.6.1 SD: Summary of Mean EKG (Summary of Actual and C | . 6 |
| e 14.3.4.6.2 MAD: Summary of Mean EKG (Summary of Actual a | 9: |
| e 14.3.4.7.1 SD: Summary of EKG Interpretation (Worst) by T | 6 |
| e 14.3.4.7.2 MAD: Summary of EKG Interpretation (Worst) by Timepoint | ا<br>: |
| e 14.3.4.8.1 SD: Summary of CURB-65 Score(Summary of Actual and Change from Baseline Values) by Ti | - |
| e 14.3.4.8.2 MAD: Summary of CURB-65 Score (Summary of Actual and Change from Baseline Val | : |
| e 14.3.4.9.1 SD: Summary of PSI Score (Summary of Actual and C | . 7 |
| e 14.3.4.9.2 MAD: Summary of PSI Score (Summary of | · ' |
| Table 14.3.4.10.1 SD: Summary of PSI Risk Class by Timepoint | : ' |
| e 14.3.4.11.1 SD: Summary of SOFA Score (Summary | |
| e 14.3.4.11.2 MAD: Summary of SOFA Score (Summary of Actual and | |
| Table 14.3.4.12.1 SD: Summary of MMSE Score (Summary of Actual and Change from Baseline Values) by Timepoint | |
| Table 14.3.4.12.2 MAD: Summary of MMSE Score (Summary of Actual and Change from Baseline Values) by Timepoint | ∞: |

| 12-03 | | 81 | 82 |
|---|---|---|---|
| 2018-12-03 | | | |
| 0 | | lization81 | talization82 |
| ocument status: Mock EOS Tables, Final V2.0 Amendment V1.0 | | | |
| nendm | | | |
| V2.0 AI | | | |
| s, Final | | | |
| S Table | | | |
| lock EC | | | |
| atus: N | | n | on |
| ment st | | ization | izati |
| Docu | | itali | pital |
| | | Hosp | of Hos |
| | | ary of | nary |
| | | Summs | : Sum |
| | | 1 SD: | 2 MAD |
| I-201 | | 4.13. | 4.13. |
| No: BT | | 14.3. | 14.3. |
| Protocol No: BTI-201 | | Table 14.3.4.13.1 SD: Summary of Hospita. | Table 14.3.4.13.2 MAD: Summary of Hospit |
| | , | | |

# **GENERAL COMMENTS**

- Where a count is 0, the percentage will not be shown (e.g. 0 (0.0%) will be displayed as 0)
- Unless otherwise states, parameters will be listed in alphabetical order
- Percentages and their 95% CI, where appropriate, will be presented to one decimal place
- The minimum and maximum values will be presented to the same number of decimal places as recorded in the electronic Case Report Form (eCRF)
- Mean, median, and SD will be presented to one more decimal place than the raw data
- Percentages will be rounded to one decimal place, with the denominator being the number of subjects in the relevant population with non-missing data, unless otherwise specified
- Change from Baseline:

Change from Baseline will be calculated as:

Change from baseline = new value - baseline value

- Unscheduled visits will be excluded from summary tables
- Names and order of Treatment Groups
- rhu-pGSN 6 mg/kg;
  - Placebo;
- Overall.

### MAD:

- rhu-pGSN 6 mg/kg;
- rhu-pGSN 12 mg/kg;
- rhu-pGSN 24 mg/kg;
  - Combined Placebo;
    - - Overall.

Names of visits SD:

Screening
Day 1
Day 3/4
Day 7/4
Day 14
Day 14
Day 18 / Early Termination (Combined visit for safety and PD)

MAD:

Screening

Day 1
Day 2
Day 3
Day 4
Day 7
Day 7

Day 28 / Early Termination (Combined visit for safety and PD)

Column widths and text-wrapping may be altered in final output in order to best present the data

Footnotes may be added/amended if required

Table 14.1.1.1 SD: Summary of Subject Enrolment and Disposition Protocol: BTI-201 Intent-to-Treat Population

Protocol No: BTI-201

| | rhu-pGSN<br>6 mg/kg<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|
| Number of Subjects Screened | ×× | ×× | ×× |
| Number of Screening Failures <sup>1</sup> | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| Number of Subjects Randomized | ×× | XX | ×× |
| Number of Subjects who Completed the Study | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects Discontinued | (XX.X%) | xx (xx.x%) | (xx.x%) |
| Primary Reason for Discontinuation of Study | | | |
| Due to Adverse Event | (xx.x%) | (xx.x%) | (%x.x%) xx |
| Subject withdrew consent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Investigator Decision | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Non-Compliance with the study procedures/protocol | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Any clinically significant change in subject's medical condition | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Sponsor ended study | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) |
| Lost to follow-up | (×x.x%) | XX (XX.X%) | XX (XX.X%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects included in the ITT Population | (XX.X%) | (xx.x%) xx | (xx.x%) |
| Number of Subjects included in the Safety Population | ( XX.X%) X | XX (XX.X%) | XX (XX.X%) |
| Number of Subjects included in the PK Population | ( XX.X%) X | XX (XX.X%) | XX (XX.X%) |
| Number of Subjects included in the PP Population | (×x.x%) x | xx (xx.x%) xx | xx (xx.x%) |

<sup>&</sup>lt;sup>1</sup>Percentages are based on number of subjects screened.

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Table 14.1.1.2 MAD: Summary of Subject Enrolment and Disposition Protocol:  ${\tt BTI-201}$  Intent-to-Treat Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Repeat Table 14.1.1.1 Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Programming Note:

Combined Active;

Combined Placebo;

Overall


Table 14.1.2.1 SD: Summary of Demographics and Baseline Characteristics Protocol: BTI-201 Intent-to-Treat Population


| | | rhu-pGSN<br>6 mg/kg<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Age (Years) at Screening | а | ×× | ×× | ×× |
| | Mean | ×.× | x.xx | x.xx |
| | Median | × . × × | x.xx | x.xx |
| | SD | ×.<br>× | ×.× | XX.XX |
| | Minimum | ×× | ×× | ×× |
| | Maximum | ×× | ×× | ×× |
| Sex n(%) | Female | (×.xx) xx | xx (xx.x%) | xx (xx.x%) |
| | Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Race n(%) | Asian | (%x.x%) xx | (xx.x%) | (xx.x%) |
| | Pacific Islander | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) |
| | Black or African | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| | Pacific Islander | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| | Aborigine/Torres Strait Islander | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | White | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Childbearing Potential n(%)* | Yes | (xx.x%) | XX (XX.X%) | XX (XX.X%) |
| | No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>\*</sup>Percentages are based on the number of female participants. SD: Standard Deviation

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Table 14.1.2.1 SD: Summary of Demographics and Baseline Characteristics Protocol: BTI-201 Intent-to-Treat Population


| | | rhu-pgsN<br>6 mg/kg<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Height (cm) | и | ×× | ×× | ×× |
| | Mean | XXX.X | XX.XX | xx.x |
| | Median | XX.X | XX.XX | xx.x |
| | SD | ×.× | ×.× | x.xx |
| | Minimum | XX | XX | XX |
| | Maximum | XX | XX | XX |
| Weight (kg) | n | ×× | ×× | XX |
| | Mean | x.xx | XX.X | x.xx |
| | Median | x.xx | XX.X | x.xx |
| | SD | ×.× | ×.× | x.xx |
| | Minimum | ×× | XX | ×× |
| | Maximum | XX | ×× | ×× |

<sup>\*</sup>Percentages are based on the number of female participants. SD: Standard Deviation

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Table 14.1.2.2 MAD: Summary of Demographics and Baseline Characteristics Protocol:  ${\tt BTI-201}$  Intent-to-Treat Population

Programming Note: Repeat Table 14.1.2.1

Include: rhu-pGSN 6 mg/kg;

rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active;

Combined Placebo;

Overall


Table 14.2.1.1 Day 1: Summary of Plasma pGSN Concentrations (unit) by Timepoint Protocol: BTI-201
PK Population

| | | | SD/MAD | | | MAD | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | rhu-pgsN | | | rhu-pgsN | | | |
| | | | 6 mg/kg | | | 12 mg/kg | | Pl | Placebo |
| Time Point | | | (N=XX) | | | (N=xx) | | () | (N=xx) |
| | | | | Ratio from | | | Ratio from | | |
| | | | | Pre- | | | Pre- | | |
| | | | | Injection/<br>Placebo | | | Injection/<br>Placebo | | |
| | | | Ratio | Ratio from | | Ratio | Ratio from | | Ratio |
| | | Actual | from Pre- | Pre- | Actual | from Pre- | Pre- | Actual | from Pre- |
| | | Value | Injection | Injection | Value | Injection | Injection | Value | Injection |
| Pre-Injection | п | × | | | × | | | × | |
| | Mean | ×. × | | | ×× | | | ×.× | |
| | Median | × : | | | ×. | | | ×. | |
| | SD | ×. × | | | ×.× | | | ×.× | |
| | Minimum | × | | | × | | | × | |
| | Maximum | × | | | × | | | × | |
| | CV% | ×. × | | | ×× | | | ×. × | |
| | GeoMean | ×.× | | | ×. × | | | ×. × | |
| | GeoCV% | ×: × | | | ×: | | | ×.× | |
| | BLQ | ( XX. X%) | | | ( XX · X%) | | | ( XX · X%) | |
| 5 to 10 mins post | а | × | × | × | × | × | × | × | × |
| 4 | Mean | ×.× | ×.× | ×. × | ×. | ×. × | ×.× | ×.× | ×.× |
| | SD | ×. | ×. | ×.× | ×. | ×.× | ×. × | ×. | ×.× |
| | Minimum | ×. × | ×. × | ×: × | ×.× | ×.× | ×.× | ×.× | ×.× |
| | Median | × | × | × | × | × | × | × | × |
| | Maximum | × | × | × | × | × | × | × | × |
| | CV% | ×. × | ×:× | ×: × | ×: | ×. × | ×: × | ×.× | ×.× |
| | ln SD | | ×:× | ×: × | | ×. × | ×: × | | ×.× |
| | GeoMean | ×. × | ×.× | ×× | ×× | ×.× | ×: × | ×. × | ×.× |
| | GeoCV% | ×.<br>× | ×. × | ×: × | × . | ××× | ×. × | × | ×.× |

<sup>....</sup> Sp: Standard Deviation; GeoMean: Geometric Mean; GeoCV%: Geometric CV%; BLQ: Below Limit of Quantification

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat for all timepoints.

( ×x · x %) ×

( %x.x%) × × ×

x (xx.x%) x (%x.x%)

x (xx.x%) x

x (xx.x%) ×

x (xx.x%) x (%x.x%)

x (xx.x%) x

( XX.X%) ×

GeoMean GeoCV% BLQ

Table 14.2.1.1 Day 1: Summary of Plasma pGSN Concentrations (unit) by Timepoint (continued) Protocol: BTI-201 PK Population

| Time Point | | MAD<br>rhu-pgSN<br>24 mg/kg<br>(N=xx) | Ratio from Pre- | <u>а</u> | Placebo<br>(N=xx) |
|---|---|---|---|---|---|
| | Actual Value | Ratio from<br>Pre-Injection | Injection/<br>Placebo Ratio<br>from Pre-<br>Injection | Actual Value | Ratio<br>from Pre-Injection |

| | | | | | | | | | | × | ×: × | ×: × | × : | × | × | × · × | ** | ×: × | × : | (%x.x%) x |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| × | ×.× | ×:× | ×:× | × | × | ×:× | ×:× | ×:× | x (xx.x%) | × | ×.× | ×.× | ×:× | × | × | ×:× | | ×.× | ×:× | (XX.X%) |
| | | | | | | | | | | × | ×.× | ×.× | ×:× | × | × | ×:× | ×.× | ×.× | ×:× | x (xx.x%) |
| | | | | | | | | | | × | ×.× | ×.× | ×.× | × | × | ×.× | ×.× | ×.× | ×.× | (XX.X%) |
| × | ×.× | ×:× | × : | × | × | × : | ×: × | × : | (XX.X%) | × | ×: × | ×: × | ×: × | × | × | ×:× | | ×: × | ××× | (×.xx) x |
| п | Mean | Median | SD | Minimum | Maximum | CV% | GeoMean | GeoCV% | BLQ | ч | Mean | SD | Minimum | Median | Maximum | CV% | ln SD | GeoMean | GeoCV% | BLQ |
| Pre-Injection | | | | | | | | | | 5 to 10 mins post | | | | | | | | | | |

SD: Standard Deviation; GeoMean: Geometric Mean; GeoCV%: Geometric CV%; BLQ: Below Limit of Quantification

Clinical cut-off date: DDMMMYYYY Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat for all timepoints.

Table 14.2.1.2 Day 2: Summary of Plasma pGSN Concentrations (unit) by Timepoint Protocol: BTI-201PK Population

| | | | MAD | | | MAD | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | rhu-pgsN | | | rhu-pgsN | | | |
| | | | 6 mg/kg | | | 12 mg/kg | | Pl | Placebo |
| Time Point | | | (N=XX) | | | (N=XX) | | ( ) | (N=XX) |
| | | | | Ratio from | | | Ratio from | | |
| | | | | Pre- | | | Pre- | | |
| | | | | Injection/ | | | Injection/ | | |
| | | | | Placebo | | | Placebo | | |
| | | | Ratio | Ratio from | | Ratio | Ratio from | | Ratio |
| | | Actual | from Pre- | Pre- | Actual | from Pre- | Pre- | Actual | from Pre- |
| | | Value | Injection | Injection | Value | Injection | Injection | Value | Injection |
| Pre-Injection | ជ | × | | | × | | | × | |
| | Mean | ×. | | | ×.× | | | ×.× | |
| | Median | ×. × | | | ×. × | | | ×. × | |
| | SD | ×. | | | ×.× | | | ×.× | |
| | Minimum | × | | | × | | | × | |
| | Maximum | × | | | × | | | × | |
| | CV% | ×. × | | | ×. × | | | ×. × | |
| | GeoMean | ×. × | | | × : | | | × . | |
| | GeoCV% | ×. × | | | ×. × | | | × : | |
| | BLQ | x (xx.x%) | | | ( XX.X%) | | | x (xx.x%) | |
| 5 to 10 mins post | ч | × | × | × | × | × | × | × | × |
| | Mean | ×. × | ×.× | ×. × | ×. × | ×. × | ××× | ×.× | ×.× |
| | SD | ×. × | ×.× | ×.× | ×. × | ×.× | ×.× | ×. × | ×.× |
| | Minimum | ×: × | ×.× | ×.× | ×. × | ×. × | ×.× | ×.× | ×.× |
| | Median | × | × | × | × | × | × | × | × |
| | Maximum | × | × | × | × | × | × | × | × |
| | CV% | ×: × | ×.× | ×.× | ×. × | ×. × | ×.× | ×.× | ×.× |
| | ln SD | | ×. × | ×. × | | ×.× | ×.× | | ×.× |
| | GeoMean | × | × | × | ×<br>× | × : | × : | × | ×: |

<sup>...</sup> SD: Standard Deviation; GeoMean: Geometric Mean; GeoCV%: Geometric CV%; BLQ: Below Limit of Quantification

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:NM

Programming Note: Repeat for all timepoints.

(%x.xx) x

(%x.xx) x × ×

x (xx.x%)

(%x.x%) x

x (xx.x%)

x (xx.x%)

x (xx.x%)

( ×x.x%) ×

× ×

× × × ×

× × × ×

× × × ×

GeoCV%

×


Table 14.2.1.2 Day 2: Summary of Plasma pGSN Concentrations (unit) by Timepoint (continued) Protocol: BTI-201 PK Population

| | | Placebo | (N=xx) | Ratio<br>Actual Value from Pre-Injection | × | х.х | X.X | ×.× | × | × | х.х | х.х | х.х | x (xx.x%) | × | X.X X.X | X.X X.X | x.x | × | × | х.х | х.х | x.x | x.x | x (xx.x%) x (xx.x%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Ratio from Pre-<br>Injection/<br>Placebo Ratio<br>from Pre-<br>Injection | | | | | | | | | | | × | ×.× | ×.× | ×.× | × | × | ×.× | ×.× | ×:× | ×:× | (XX.X%) |
| MAD | TIU-DOSN | 24 mg/kg | (N=XX) | Ratio from<br>Pre-Injection | | | | | | | | | | | × | ×:× | ×:× | ×.× | × | × | ×:× | ×:× | ×:× | ×:× | x (xx.x%) |
| | | | | Actual Value | × | ×: × | ×: × | ×: × | × | × | ××× | ××× | ××× | x (xx.x%) | × | ×: × | ×: × | ×: × | × | × | ×:× | | ×: × | ×: × | x (xx.x⋄) |
| | | | | | п | Mean | Median | SD | Minimum | Maximum | CV% | GeoMean | GeoCV% | BLQ | น | Mean | SD | Minimum | Median | Maximum | CV% | ln SD | GeoMean | GeoCV% | BLQ |
| | | | Time Point | | Pre-Injection | | | | | | | | | | 5 to 10 mins post | | | | | | | | | | |

SD: Standard Deviation; GeoMean: Geometric Mean; GeoCV%: Geometric CV%; BLQ: Below Limit of Quantification

Clinical cut-off date: DDMMMYYYY Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat for all timepoints.

Table 14.2.1.3 Day 3: Summary of Plasma pGSN Concentrations (unit) by Timepoint Protocol: BTI-201
PK Population


Programming Note: Repeat Table 14.2.1.2 for Day 3.


Table 14.2.1.4 Day 1: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint Protocol: BTI-201 PK Population

| | | | SD/MAD<br>rhu-pgsN | | | MAD<br>rhu-pGSN | | | |
|---|---|---|---|---|---|---|---|---|---|
| E | | | 6 mg/kg | | | 12 mg/kg<br>(N=××) | | . P. | Placebo (N=v*) |
| | | | 1 | (Change from Pre-<br>Injection) - | | | (Change from Pre-<br>Injection) - | | |
| | | Actual | Change<br>from Pre-<br>Thiection | Change from Pre- | Actual | Change<br>from Pre-<br>Injection | Change from Pre- | Actual | Change<br>from Pre- |
| | | | | (1) | | | | | |
| Pre-Injection | п | × | | | × | | | × | |
| | Mean | ×.× | | | × | | | ×.<br>× | |
| | Median | ×. | | | ×. | | | ×.<br>× | |
| | SD | ×.<br>× | | | ×. | | | ×.<br>× | |
| | Minimum | × | | | × | | | × | |
| | Maximum | × | | | × | | | × | |
| | CV% | ×. | | | ×. | | | ×. | |
| | BLQ | ( xx.x%) | | | ( XX . X%) | | | (×x.x%) | |
| 5 to 10 mins post | п | × | × | × | × | × | × | × | × |
| | Mean | ×.<br>× | ×.<br>× | ×× | ×. | × : | ×.× | ×.<br>× | ××× |
| | SD | ×.× | ×.× | ×.× | ×. × | ×.× | ×.× | ×. × | ×.× |
| | Minimum | ×.× | ×.× | ×.× | ×. × | × :× | ×.× | ×.× | ×.× |
| | Median | × | × | × | × | × | × | × | × |
| | Maximum | × | × | × | × | × | × | × | × |
| | CV% | ×. | ×.× | ×.× | ×. | ×.* | ×.× | ×. × | ××× |
| | BLQ | (XX.X%) | | | ( XX . X%) X | | | ( XX . X%) X | |

<sup>...</sup> SD: Standard Deviation; BLQ: Below Limit of Quantification

Clinical cut-off date: DDMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:MM

Programming Note: Repeat for all timepoints.

Table 14.2.1.4 Day 1: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint (continued) Protocol: BTI-201 PK Population

| | | | MAD<br>rhu-pGSN | | | |
|---|---|---|---|---|---|---|
| | | | 24 mg/kg | | Д | Placebo |
| Time Point | | | (N=XX) | | ) | (N=xx) |
| | | Actual Value | Change from<br>Pre-Injection | (Change from Pre-<br>Injection) -<br>(Mean Placebo<br>Change from Pre-<br>Injection) | Actual Value | Change<br>from Pre-Injection |
| Pre-Injection | п | × | | | × | |
| | Mean | × : | | | ×.× | |
| | Median | * * * | | | × × | |
| | SD | * * * | | | × × | |
| | Minimum | × | | | × | |
| | Maximum | × | | | × | |
| | CV% | × :× | | | ×:× | |
| | BLQ | x (xx.x%) | | | x (xx.x%) | |
| 5 to 10 mins post | ជ | × | × | × | × | × |
| | Mean | × · × | ×.× | ×.× | ×.× | ×.× |
| | SD | * * * | ×.× | ×.× | ×.× | ×.× |
| | Minimum | ××× | ×. × | × : × | ×.× | ×.× |
| | Median | × | × | × | × | × |
| | Maximum | × | × | × | × | × |
| | CV% | ×.× | ×.× | ×.× | × · × | ×.× |
| | BLQ | ( XX.X%) X | | | (×x.x%) x | |
| • | | | | | | |

SD: Standard Deviation; BLQ: Below Limit of Quantification

Clinical cut-off date: DDMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:MM

Programming Note: Repeat for all timepoints.


Table 14.2.1.5 Day 2: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint Protocol: BTI-201 PK Population

| Time Point | | | MAD<br>rhu-pGSN<br>6 mg/kg<br>(N=xx) | | | MAD<br>rhu-pGSN<br>12 mg/kg<br>(N=xx) | | P1<br>(N | Placebo<br>(N=xx) |
|---|---|---|---|---|---|---|---|---|---|
| | | Actual<br>Value | Change<br>from Pre-<br>Injection | (Change from Pre- Injection) - (Mean Placebo Change from Pre- Injection) | Actual<br>Value | Change<br>from Pre-<br>Injection | (Change from Pre- Injection) - (Mean Placebo Change from Pre- Injection) | Actual<br>Value | Change<br>from Pre-<br>Injection |
| 77<br>77<br>77<br>77<br>77<br>77 | ۶ | > | | | > | | | ٥ | |
| | Mean | ×× | | | < × | | | × × | |
| | Median | ×.× | | | ×. × | | | ×.× | |
| | SD | ×.× | | | ×. × | | | ×.× | |
| | Minimum | × | | | × | | | × | |
| | Maximum | × | | | × | | | × | |
| | CV% | ×. | | | ×. × | | | ×. | |
| | BLQ | ( XX.X%) X | | | ( XX.X%) | | | (XX.X%) | |
| 5 to 10 mins post | п | × | × | × | × | × | × | × | × |
| | Mean | ×. × | ×. | ×. | × : | × : | ×.× | × : | ×.× |
| | SD | ×. × | ×. | ×. | × : | × : | ×.× | × : | ×.× |
| | Minimum | ×.× | ×.× | ×.× | ×.× | ×.× | ×.× | ×.× | ×.× |
| | Median | × | × | × | × | × | × | × | × |
| | Maximum | × | × | × | × | × | × | × | × |
| | CV% | ×.× | ××× | ×.× | ×.<br>× | ×.× | ×.× | ×. | ×.× |
| | BLQ | x (xx.x%) | | | X (XX.X%) | | | ( ××. ×%) × | |
| : | | | | | | | | | |

SD: Standard Deviation; BLQ: Below Limit of Quantification

Clinical cut-off date: DDMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:MM

Table 14.2.1.5 Day 2: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint (continued) Protocol: BTI-201
PK Population

| Time Point | | MAD<br>rhu-pGSN<br>24 mg/kg<br>(N=xx) | | P. | Placebo<br>(N=xx) |
|---|---|---|---|---|---|
| | Actual Value | Change from<br>Pre-Injection | (Change from Pre-Injection) - (Mean Placebo Change from Pre-Injection) | Actual Value | Change<br>from Pre-Injection |
| | | ١ | | | n |

| | | | | | | | | × | ×.× | ×.× | × :× | × | × | ×.× | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| × | * * | ×.× | ×.× | × | × | × :× | x (xx.x%) | × | ×.× | ×.× | × :× | × | × | × : | x (xx.x%) |
| | | | | | | | | × | ×:× | ×:× | × :× | × | × | ×:× | |
| | | | | | | | | × | ×.× | ×.× | ×.× | × | × | ×.× | |
| × | ×.× | × : | × : | × | × | × : | x (xx.x%) | × | ×:× | ×:× | × : | × | × | ×:× | (XX.X%) |
| ជ | Mean | Median | SD | Minimum | Maximum | CV% | BLQ | ជ | Mean | SD | Minimum | Median | Maximum | CV% | BLQ |
| Pre-Injection | 1 | | | | | | | 5 to 10 mins post | | | | | | | |

... SD: Standard Deviation; GeoMean: Geometric Mean; GeoCV%: Geometric CV%; BLQ: Below Limit of Quantification

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat for all timepoints.

2018-12-03

Table 14.2.1.6 Day 3: Summary of Estimated Plasma rhu-pGSN Concentrations (unit) by Timepoint Protocol: BTI-201 PK Population

Programming Note: Repeat Table 14.2.1.5 for Day 3.


Table 14.2.2.1 Day 1: Summary of Plasma pGSN PK Parameters Protocol: BTI-201 PK Population

| Parameter (unit) | | SD/MAD $IDSN$ $G mg/kg$ $(N=xx)$ | MAD<br>rhu-pGSN<br>12 mg/kg<br>(N=xx) | MAD rhu-pGSN $24 \text{ mg/kg}$ (N=xx) | Placebo<br>(N=xx) |
|---|---|---|---|---|---|
| AUC <sub>0-t</sub> (unit) | ч | × | × | × | × |
| | Mean | × . × | ××× | ××× | ×:× |
| | SD | × : | × : | ××× | ×.× |
| | Minimum | ×.× | × : | × : × | ×.×. |
| | Median | × | × | × | × |
| | Maximum | × | × | × | × |
| | CV% | ×.× | × : | ×.× | ×. × |
| | GeoMean | ×.× | ×.× | ×.× | ×.×. |
| | GeoCV% | ×. × | ×. × | ×.× | ×.<br>× |
| C <sub>max</sub> (unit) | П | × | × | × | × |
| | Mean | ×: × | × | ××× | ×:× |
| | SD | ×.× | × : | × : | ×.× |
| | Minimum | ×.× | × : | ×.× | ×. × |
| | Median | × | × | × | × |
| | Maximum | × | × | × | × |
| | CV% | ×.× | ×.× | ×.× | ×. × |
| | GeoMean | ×.× | × : | × : × | ×.×. |
| | %/1\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | > | > | > | > |

SD: Standard Deviation; GeoMean: Geometric Mean; GeoCV%: Geometric CV%

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat for all PK parameters.

Table 14.2.2.2 Day 2: Summary of Plasma pGSN PK Parameters Protocol: BTI-201 PK Population

| Parameter (unit) | | MAD<br>rhu-pgsN<br>6 mg/kq | MAD<br>rhu-pGSN<br>12 mg/kg | MAD<br>rhu-pGSN<br>24 mg/kg | Placebo |
|---|---|---|---|---|---|
| | | (N=XX) | (N=XX) | (N=XX) | (N=xx) |
| AUC <sub>0-t</sub> (unit) | g | × | × | × | × |
| | Mean | ×.× | × : | ×: × | ××× |
| | SD | ×:× | × : × | ×: × | ×: × |
| I | Minimum | ×:× | × : × | ×.× | ×: × |
| I | Median | × | × | × | × |
| I | Maximum | × | × | × | × |
| | CV% | ×:× | × : × | ×.× | ×: × |
| | GeoMean | × : | × : × | ×: × | ××× |
| | GeoCV% | ×.* | ×.× | ×. × | ×.× |
| C <sub>max</sub> (unit) | ч | × | × | × | × |
| | Mean | × : | × : × | ×: × | ××× |
| | SD | ×.× | × : × | ×: × | ×: × |
| I | Minimum | ×:× | ×.× | ×.× | × :× |
| I | Median | × | × | × | × |
| I | Maximum | × | × | × | × |
| | CV% | ×:× | × · × | ×.× | ×: × |
| | GeoMean | ×:× | ×.× | ×.× | ×. × |
| | GeoCV% | ×:× | ×.× | ×.× | × :× |

SD: Standard Deviation; GeoMean: Geometric Mean; GeoCV%: Geometric CV%

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat for all PK parameters.

Table 14.2.2.3 Day 3: Summary of Plasma pGSN PK Parameters PK Population

| pulation |
|----------|
| K Po |

| | | MAD<br>rhu-pgsN<br>6 ma/ka | MAD<br>rhu-pgsN<br>12 mg/kg | MAD<br>rhu-pGSN<br>24 mg/kg | ر<br>دره م |
|---|---|---|---|---|---|
| Parameter (unit) | | (X=N) | (N=XX) | (XX=N) | (N=XX) |
| AUC <sub>0-t</sub> (unit) | ជ | × | × | × | × |
| | Mean | ×.× | ×.× | ×: × | ××× |
| | SD | ×.× | ×.× | *: | ×.× |
| | Minimum | ×.× | ×.× | ×: × | ×.× |
| | Median | × | × | × | × |
| | Maximum | × | × | × | × |
| | CV% | ×.× | ×.× | *: | ×.× |
| | GeoMean | ×.× | ×.× | *: | ×.× |
| | GeoCV% | ×.× | ×.× | ×.× | × . × |
| C <sub>max</sub> (unit) | ជ | × | × | × | × |
| | Mean | ×.× | ×.× | ×:× | ×.× |
| | SD | ×.× | ×.× | *: | ×.× |
| | Minimum | ×.× | ×.× | ×: × | ×.× |
| | Median | × | × | × | × |
| | Maximum | × | × | × | × |
| | CV% | ×.× | ×.× | ×:× | ×.× |
| | GeoMean | × :× | ×.× | × : × | ×. × |
| | SPOCV* | ××× | ×·× | ××× | ××× |

SD: Standard Deviation; GeoMean: Geometric Mean; GeoCV%: Geometric CV%

Programming Note: Repeat for all PK parameters.

Clinical cut-off date: DDMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:MM

Table 14.2.3.1 Day 1: Summary of Estimated Plasma rhu-pGSN PK Parameters Protocol:  ${\tt BTI-201}$  PK Population

| | | SD/MAD<br>rhu-pGSN<br>6 mg/kg<br>(N=xx) | IAD<br>ogsn<br>/kg<br>:*) | MAD<br>rhu-pGSN<br>12 mg/kg<br>(N=xx) | D<br>ogsn<br>g/kg | MAD<br>rhu-pGSN<br>24 mg/kg<br>(N=xx) | LD<br>pgsn<br>g/kg |
|---|---|---|---|---|---|---|---|
| Parameter (unit) | | Change from Pre-Injection | Double Delta<br>Analysis | Change from<br>Pre-Injection | Double Delta<br>Analysis | Change from | Double Delta<br>Analysis |
| AUC <sub>0-t</sub> (unit) | ជ | × | × | × | × | × | × |
| | Mean | ××× | ×.× | ×.× | ×.× | ×× | × × |
| | SD | ×.× | ×.× | ×.× | ×.× | ××× | × × |
| | Minimum | ×.× | ×.× | ×.× | ×.× | ××× | × × |
| | Median | × | × | × | × | × | × |
| | Maximum | × | × | × | × | × | × |
| | CV% | ×.× | × | ×.× | ×. × | ×. × | ×. × |
| C <sub>max</sub> (unit) | น | × | × | × | × | × | × |
| | Mean | ×.× | ×.× | ×.× | ×.× | ××× | × × |
| | SD | ×.× | ×.× | ×.× | ×.× | ×.× | ×.× |
| | Minimum | ×.× | ×.× | ×.× | ×.× | ××× | ×.× |
| | Median | × | × | × | × | × | × |
| | Maximum | × | × | × | × | × | × |
| | CV% | ×.× | ××× | ×. × | ×. × | ×. × | ×. × |

SD: Standard Deviation;

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Include the following: PK parameters (including dose normalized parameters):

- AUC<sub>0-t</sub>
- AUC<sub>0-8h</sub>

Table 14.2.3.2 Day 2: Summary of Estimated Plasma rhu-pGSN PK Parameters Protocol: BTI-201 PK Population

| MAD | rhu-pgsN | 24 mg/kg | (X=X) |
|-----|----------|-----------------|--------------------------------|
| MAD | rhu-pgsN | 12 mg/kg | (N=XX) |
| MAD | rhu-pgsN | 6 mg/kg | (N=XX) |
| | MAD | MAD<br>rhu-pgsn | MAD SN rhu-pGSN cg 12 mg/kg 24 |

| Parameter (unit) | | Change from<br>Pre-Injection | Double Delta<br>Analysis | Change from<br>Pre-Injection | Double Delta<br>Analysis | Change from<br>Pre-Injection | Double Delta<br>Analysis |
|---|---|---|---|---|---|---|---|
| AUC <sub>0-t</sub> (unit) | и | × | × | × | × | × | × |
| | Mean | × : | ××× | ×.× | ×. × | ×× | ××× |
| | SD | × : | ××× | ×.× | ×.× | ××× | ×.× |
| | Minimum | ×.× | ×.× | ×.× | ×.× | ×.× | ×.× |
| | Median | × | × | × | × | × | × |
| | Maximum | × | × | × | × | × | × |
| | CV% | ×. × | × . | ×. | × | × . × | × . × |
| C <sub>max</sub> (unit) | п | × | × | × | × | × | × |
| | Mean | × : | ××× | ×.× | ×.× | ××× | ×.× |
| | SD | ×.× | ×.× | ×.× | ×.× | ×.× | ×.× |
| | Minimum | ×: × | ×.× | ×.× | ×.× | ××× | ×.× |
| | Median | × | × | × | × | × | × |
| | Maximum | × | × | × | × | × | × |
| | CV% | ×.× | ×.× | ×. × | ×.× | ×.× | ×.× |

SD: Standard Deviation;

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Include the following: PK parameters (including dose normalized parameters):

- AUC<sub>0-t</sub>
- AUC<sub>0-8h</sub>

Table 14.2.3.3 Day 3: Summary of Estimated Plasma rhu-pGSN PK Parameters Protocol: BTI-201 PK Population

| Parameter (unit) | | Change from<br>Pre-Injection | Double Delta<br>Analysis | Change from<br>Pre-Injection | Double Delta<br>Analysis | Change from<br>Pre-Injection | Double Delta<br>Analysis |
|---|---|---|---|---|---|---|---|
| AUCo-+ (unit) | ٤ | × | × | × | × | × | × |
| | Mean | ×.× | × | ×× | × | ×.× | ××× |
| | SD | ×.× | ×.× | ×.× | ×.× | ×× | ×.× |
| | Minimum | × : | ×.× | ×.× | ×.× | ×× | ××× |
| | Median | × | × | × | × | × | × |
| | Maximum | × | × | × | × | × | × |
| | CV% | ×. × | × . × | × . | × : | × . × | × : |
| C <sub>max</sub> (unit) | ជ | × | × | × | × | × | × |
| | Mean | × : | ×.× | ×.× | ××× | ××× | ××× |
| | SD | ×.× | ×.× | ×.× | ×.× | ×.× | ××× |
| | Minimum | ×: × | ×.× | ×.× | ×. × | ××× | ×.× |
| | Median | × | × | × | × | × | × |
| | Maximum | × | × | × | × | × | × |
| | CV% | ×.× | ×.× | ×.× | ×. × | ×.× | ×.× |

SD: Standard Deviation;

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Include the following: PK parameters (including dose normalized parameters):

- AUC<sub>0-t</sub>
- AUC<sub>0-8h</sub>

Table 14.2.4.1 SD: Summary of PD Parameters Protocol: BTI-201
Intent-to-Treat Population

| | | | rhu-pGSN 6 mg/kg | 6 mg/kg | д ` | Placebo | Overall | all<br>> |
|---|---|---|---|---|---|---|---|---|
| | | | | AA)<br>Ratio from | | (N-AA)<br>Ratio from | ( | A)<br>Ratio from |
| Parameter | Visit | | Actual Value | Baseline1 | Value | Baseline $^1$ | Actual Value | Baseline1 |
| - | | | | | | | | |
| Procalcitonin (unit) | Baseline⊥ | п | × | | × | | × | |
| | | Mean | ××××. | | ××××. | | ×.xx | |
| | | Median | ×××.× | | ××××× | | ××××× | |
| | | SD | ××××× | | ×××××× | | xxx.x | |
| | | Minimum | ××.× | | × | | ××.× | |
| | | Maximum | ××.× | | ×. × | | XX.X | |
| | | GeoMean | X.XXX | | xxx.x | | X.XXX | |
| | Day 2 | Ş | × | × | × | × | × | > |
| | | 11 : | h | | h | | | h h |
| | | Mean | ××××× | ××××× | ××××× | ××××× | ××××× | ××××× |
| | | SD | XXXX.X | XXXX.X | XXXX.X | XXXX.X | X.XXX | XXXX.X |
| | | Minimum | ×××.× | xxxxx | ××××× | ×. x x | xxx.x | xxxxx |
| | | Median | ××.× | ××.× | ××.× | ××.× | XX.X | x.xx |
| | | Maximum | ××.× | ××.× | ××.× | ××.× | ××.× | ××.× |
| | | ln SD | | ××××× | | ×××.× | | ××××× |
| | | GeoMean | X.XX. | x.xx | ×××. | x x x x | x.xx | x.xx |
| | ( | | | | | | | |
| | Day 3 or 4 | п | × | × | × | × | × | × |
| | | Mean | X.XXX | XXXX.X | XXXX.X | XXXX.X | X.XXX | XXXX.X |
| | | SD | ×.xxx | ××××× | ××××. | ×. ××× | ×××××× | ×.xxx |
| | | Minimum | ××××× | xxx.x | ××××. | ×××.× | xxx.x | ×.xxx |
| | | Median | ××.× | ××.× | ×. × | ××.× | ××.× | ××.× |
| | | Maximum | ××.× | ××.× | ××.× | ××.× | ××.× | ×× |
| | | ln SD | | xxx.x | | ×. x x | | xxxxx |
| | | GeoMean | ×××.× | xxx.x | ××××× | ×. x x | XXXX.X | xxxxx |
| etc. | etc. | | | | | | | |

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM Novotech - Strictly Confidential Clinical cut-off date: DDMMMYYYY

Programming Note: Repeat for all PD parameters and all scheduled post baseline timepoints.

Note: SD: Standard Deviation

Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Unscheduled visits not included in post baseline assessments.

2018-12-03

Table 14.2.4.2 MAD: Summary of PD Parameters Protocol: BTI-201 Intent-to-Treat Population

Programming Note:
Repeat Table 14.2.4.1
Include: rhu-pGSN 6 mg/kg;
rhu-pGSN 12 mg/kg;
rhu-pGSN 24 mg/kg;
Combined Active; Combined Placebo; Overall

Table 14.2.5.1 SD: Summary of PD Parameters Protocol: BTI-201
Per Protocol Population

| | | | rhu-pGSN 6 mg/kg | 6 mg/kg | P | Placebo (N=v*) | Overall | (11) |
|---|---|---|---|---|---|---|---|---|
| | | | 7 | Ratio from | \ | Ratio from | 77 17 | Ratio from |
| Parameter | Visit | | Actual Value | Baseline $^1$ | Value | Baseline $^1$ | Actual Value | Baseline <sup>1</sup> |
| Procalcitonin (unit) | ${\tt Baseline}^1$ | п | × | | × | | × | |
| | | Mean | ××××× | | ×××××× | | xxx.x | |
| | | Median | ××××× | | ××××× | | xxx.x | |
| | | SD | xxx.x | | ××××× | | XXXX.X | |
| | | Minimum | ××.× | | ××.× | | xx.x | |
| | | Maximum | ××.× | | × . × | | x. xx | |
| | | GeoMean | X.XXX | | x.xx | | X.XXX | |
| | Day 2 | ٤ | × | × | × | × | × | × |
| | | Mean | ×.xxx | ××××× | xxx.x | ×.xx | xxx.x | ×××.× |
| | | SD | XXXX.X | XXXX.X | xxx.x | XXXX.X | XXXX.X | XXXX.X |
| | | Minimum | XXXX.X | XXXX.X | xxx.x | XXXX.X | XXXX.X | XXXX.X |
| | | Median | ××.× | ××.× | ××. | XX.X | XX.X | XX.X |
| | | Maximum | ××.× | ×. x | ××.× | ×. × | x.xx | ××.× |
| | | ln SD | | XXXX.X | | x.xxx | | ×××××× |
| | | GeoMean | ××××× | ×××.× | xxx.x | ×××. | × × × × | × × × × |
| | ( | | : | : | ; | ; | : | : |
| | Day 3 or 4 | п | × | × | × | × | × | × |
| | | Mean | XXXX.X | XXXX.X | XXXX.X | X.XXX | XXXX.X | XXXX.X |
| | | SD | ×.xxx | ×××××× | ×××××× | ×. xxx | x.xxx | ××××× |
| | | Minimum | ××××× | ××××× | ××××× | ×. ×. × | x.xx | ××××× |
| | | Median | ××.× | ××.× | ××.× | ×× | xx.x | ××.× |
| | | Maximum | ××.× | ××.× | ××.× | ×× | xx.x | ××.× |
| | | ln SD | | xxx.x | | x.xx | | xxx.x |
| | | GeoMean | xxx.x | xxx.x | ××××× | XXXX.X | X.XXX | xxx.x |
| etc. | etc. | | | | | | | |

Programming Note: Repeat for all PD parameters and all scheduled post baseline timepoints. Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Note: SD: Standard Deviation

Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Unscheduled visits not included in post baseline assessments.

2018-12-03

Table 14.2.5.2 MAD: Summary of PD Parameters Protocol: BTI-201
Per Protocol Population

Programming Note:
Repeat Table 14.2.5.1
Include: rhu-pGSN 6 mg/kg;
rhu-pGSN 12 mg/kg;
rhu-pGSN 24 mg/kg;
Combined Active;

Overall

Table 14.3.1.1 SD: Summary of Concomitant Medication Protocol: BTI-201 Safety Population

| Anatomic Therapeutic Classification (ATC3) | r] | rhu-pGSN<br>6 mg/kg<br>(N=xx) | 7. | | Placebo<br>(N=xx) | 0 | | Overall (N=xx) | xx) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term (PT) | Д | M (%) u | | | M (%) M | Į | | M (%) u | M (3 | |
| Subjects with at least one Concomitant Medication | ×× | xx (%x.xx) xx | × | × | xx (%x.xx) xx | × | × | ××) | xx (%x.xx) xx | × |
| ATC3/1 | ×× | xx (%x.xx) xx | × | × | xx (%x.xx) xx | × | × | ××) | xx (%x.xx) xx | × |
| PT1 | ×× | xx (xx.x%) | ×× | X | XX (XX.X%) | × | X | XX) | xx (%x.xx) xx | × |
| PT2 | ×× | xx (xx.x%) | × | × | xx (%x.xx) xx | ×× | × | XX) | xx (%x.xx) | × |
| ATC3/2 | ×× | XX (XX.X%) | × | × | XX (XX.X%) | × | × | XX (XX.X%) | | ×× |
| PT1 | ×× | (%x.xx) xx | × | × | xx (xx.x%) | × | × | (XX.X%) | | × |
| PT2 | ×× | xx (xx.x%) | ×× | X | xx (xx.x%) | × | X | xx (xx.x%) | | × |
| PT3 | ×× | (××.××) | × | × | (××.×%) | ×× | × | (××.××) | | × |
| ATC3/3 | ×× | xx (%x.xx) xx | ×× | × | xx (%x.xx) xx | × | × | ××) | xx (%x.xx) xx | × |
| PT1 | ×× | xx (xx.x%) | ×× | ×× | xx (%x.xx) xx | ×× | × | XX) | xx (%x.xx) xx | × |

Note: If a subject has multiple occurrences of a medication, the subject is presented only once in the subject count (N).

Occurrences are counted each time in the mentions/Occurrence (M) column.

WHO-DD, XXXX

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Table 14.3.1.2 MAD: Summary of Prior and Concomitant Medication Protocol:  ${\tt BTI-201}$  Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:
Repeat Table 14.3.1.1
Include: rhu-pGSN 6 mg/kg;
rhu-pGSN 12 mg/kg;
Combined Active;
Combined Placebo;
Overall


Table 14.3.3.1.1 SD: Overall Summary of Treatment-Emergent Adverse Events Protocol: BTI-201 Safety Population

| | rhu-pgsN<br>6 mg/kg | Placebo | Overall |
|---|---|---|---|
| | (N=XX) | (N=xx) | (N=xx) |
| | M (%) M | M (%) n | M (%) u |
| Number of subjects reporting at least: | | | |
| One TEAE | ×× (%ו××) ×× | ×× (%×.××) ×× | ×× (%×.××) ×× |
| One NCI-CTEAE Grade 3 TEAE | (XX.XX) | (××. ××) | (XX.XX) |
| One Serious TEAE | xx (%x.xx) xx | xx (%x.xx) xx | xx (%x.xx) xx |
| One Drug Related TEAE | xx (%x.xx) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| TEAE Leading to Death | xx (%x.xx) xx | xx (%x.x%) xx | xx (xx.x%) xx |
| One Procedure Related TEAE | xx (%x.xx) xx | xx (%x.xx) xx | xx (xx.x%) xx |
| One TEAE leading to study treatment discontinuation | xx (xx.x%) xx | xx (%x.xx) xx | xx (xx.x%) xx |
| Number of subjects reporting TEAEs by NCI-CTEAE Grade | | | |
| Grade 1 | xx (xx.x%) xx | xx (%x.x%) xx | xx (xx.x%) xx |
| Grade 2 | xx (%x.xx) xx | xx (%x.xx) xx | xx (xx.x%) xx |
| Grade 3 | xx (%x.xx) xx | xx (%x.xx) xx | xx (xx.x%) xx |
| Grade 4 | xx (%x.xx) xx | xx (%x.xx) xx | xx (xx.x%) xx |
| Grade 5 | xx (%x.xx) xx | xx (%x.xx) xx | xx (%x.xx) xx |
| אויייסיס ייליייסיס ייליייסיס יילייסיס ואבי האי הפוקעה הסיסיסיסיסיסיסיסיסיסיסיסיסיסיסיסיסיסיס | | | |
| TABLE TO STATE THE PROPERTY OF | (0: | (0: | , 0 / |
| Definitely not Kelated | ( ×× ·× × ) | (%X.X%) | (%X · X%) |
| Probably not Related | xx (%x.xx) xx | xx (%x.xx) xx | xx (%x.xx) xx |
| Possibly Related | xx (%x.xx) xx | xx (%x.xx) xx | xx (%x.xx) xx |
| Probably Related | xx (%x.xx) xx | xx (%x.xx) xx | xx (%x.xx) xx |
| Definitely Related | | | |
| Number of subjects reporting TEAEs by relationship to study procedure | | | |
| Definitely not Related | xx (%x.x%) xx | xx (%x.x%) xx | xx (%x.xx) xx |
| Probably not Related | xx (%x.xx) xx | xx (%x.xx) xx | xx (%x.xx) xx |
| Possibly Related | xx (%x.xx) xx | xx (%x.xx) xx | xx (%x.xx) xx |
| Probably Related | xx (xx.x%) xx | xx (%x.x%) xx | xx (%x.xx) xx |
| Definitely Related | | | |

in the Patient count (n) column for a given System Organ Class and Preferred Term. Occurrences are counted each time in the mentions/occurrence (M) column. Related TEAE = A Possibly, Probably related TEAE or Definitely Related.MedDRA Version xx.x the first administration of study drug. If a subject has multiple occurrences of a TEAE, the subject is presented only once Note: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurred or worsened following

Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x)

Table 14.3.3.1.2 MAD: Overall Summary of Treatment-Emergent Adverse Events Protocol:  $\rm BTI-201$  Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Include: rhu-pGSN 6 mg/kg; Repeat Table 14.3.3.1.1

rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg;

Combined Placebo; Combined Active;

Overall


Table 14.3.3.2.1 SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT) Protocol: BTI-201 Safety Population

| Subjects with at least one TEAE (N=xX) (N=XX) | | rhu-pgsN | | |
|---|---|---|---|---|
| N=xx N N N N N N N N N | | 6 mg/kg | Placebo | Overall |
| ccts with at least one TEAE xx (xx.x\$) xx xx (xx.x\$) xx | | (N=XX) | (N=xx) | (N=XX) |
| TTL XX (XX.X\$) XX | | M (%) M | | M (%) M |
| 2T1 XX (XX.X\$) XX | Subjects with at least one TEAE | xx (xx.x%) xx | xx (%x.xx) xx | xx (xx.x%) xx |
| 271 XX (XX,X\$) XX XX (X | SOC1 | | | (××.×%) |
| XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) <td>PT1</td> <td>(XX.X%)</td> <td>(XX.X%)</td> <td>(xx.x%)</td> | PT1 | (XX.X%) | (XX.X%) | (xx.x%) |
| PT1 XX (XX, X\$) XX < | SOC2 | | | (××.×%) |
| PT2 XX (XX, X\$) XX (XX, X\$) XX (XX, X\$) PT3 XX (XX, X\$) XX XX (XX, X\$) PT4 XX (XX, X\$) XX XX (XX, X\$) XX (XX, X\$) XX (XX, X\$) XX | PT1 | (××.××) | | (××.××) |
| PT3 XX (XX.X.X.\$) XX (XX.X.\$) XX (XX.X.\$) PT4 XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) PT1 XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) PT2 XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) PT3 XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) PT4 XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) PT4 XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) PT4 XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) PT4 XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) PT4 XX (XX.X.\$) XX (XX.X.\$) XX (XX.X.\$) | PT2 | (×x.x%) | (××·××) | (××.×%) |
| PT4 XX (XX, X\$) XX XX (XX, X\$) XX XX (XX, X\$) XX (XX, X\$) XX XX (XX, X\$) XX XX (XX, X\$) PT1 XX (XX, X\$) XX XX (XX, X\$) PT2 XX (XX, X\$) XX XX (XX, X\$) PT3 XX (XX, X\$) XX XX (XX, X\$) PT4 XX (XX, X\$) XX XX (XX, X\$) PT5 XX (XX, X\$) XX XX (XX, X\$) PT4 XX (XX, X\$) XX XX (XX, X\$) PT5 XX (XX, X\$) XX XX (XX, X\$) PT5 XX (XX, X\$) XX XX (XX, X\$) PT5 XX (XX, X\$) XX XX (XX, X\$) | PT3 | (××.××) | (xx.x%) | (xx.x%) |
| PT1 XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) PT2 XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) PT3 XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) PT4 XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) PT5 PT7 PT7 PT7 PT7 PT7 PT7 PT7 | PT4 | (XX.X%) | (XX.X%) | (XX.X%) |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | SOC3 | (xx.x%) | | (××.×%) |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | PT1 | (××.××) | (××.××) | (××.×%) |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | PT2 | | (××.××) | (××.×%) |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | PT3 | (×x.x%) | (××.×%) | (XX.X%) |
| xx (xx.x\$) xx | PT4 | (xx.x%) | (××·×%) | (xx.x%) |
| | PT5 | (XX.X%) | (××·×%) | (XX.X%) |

Note: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurred or worsened following the first administration of study drug. If a subject has multiple occurrences of a TEAE, the subject is presented only once in the Patient count (n) column for a given System Organ Class and Preferred Term. Occurrences are counted each time in the mentions/Occurrence (M) column. MedDRA Version xx.x

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Table 14.3.3.2.2 MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT) Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Repeat Table 14.3.3.2.1 Programming Note:

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active;

Combined Placebo;

Overall

Table 14.3.3.3.1 SD: Summary of Treatment-Emergent Deaths (Summary by SOC, PT) Protocol: BII-201 Safety Population

| | rhu-pgsN | | | |
|---|---|---|---|---|
| | 6 mg/kg | Placebo | Overall | |
| | (N=XX) | (N=XX) | (N=XX) | |
| | M (%) u | M (%) u | M (%) M | |
| Subjects with at least one TEAE leading to Death | xx (xx.x%) xx | xx (%x.x%) xx | xx (%x.xx) xx | × |
| SOCI | xx (xx.x%) xx | xx (%x.xx) xx | xx (xx.x%) xx | × |
| PT1 | xx (xx.x%) xx | xx (%x.xx) xx | xx (xx.xx) xx | XX |
| SOC2 | xx (%x.xx) xx | xx (%x.xx) xx | x (%x.x%) xx | ×× |
| PT1 | xx (%x.xx) xx | xx (%x.xx) xx | xx (%x.xx) xx | XX |
| PT2 | XX (XX.X%) XX | xx (xx.x%) xx | XX (XX.X%) XX | XX |
| PT3 | xx (xx.x%) xx | xx (%x.xx) xx | xx (%x.xx) xx | ×× |
| PT4 | xx (%x.xx) xx | xx (%x.xx) xx | xx (%x.xx) xx | × |
| 8003 | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx | × |
| PT1 | XX (XX.X%) XX | xx (xx.x%) xx | XX (XX.X%) XX | XX |
| PT2 | xx (xx.x%) xx | xx (%x.xx) xx | XX (%X.X%) XX | × |
| PT3 | xx (%x.xx) xx | xx (xx.x%) xx | xx (%x.xx) xx | XX |
| PT4 | xx (xx.x%) xx | xx (%x.xx) xx | xx (%x.xx) xx | ×× |
| PT5 | xx (xx.x%) xx | xx (xx.x%) xx | XX (%X.XX) XX | × |

Note: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurred or worsened following the first administration of study drug. If a subject has multiple occurrences of a TEAE, the subject is presented only once in the Patient count (n) column for a given System Organ Class and Preferred Term. Occurrences are counted each time in the mentions/Occurrence (M) column. MedDRA Version xx.x

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Clinical cut-off date: DDMMMYYYY

Table 14.3.3.3.2 MAD: Summary of Treatment-Emergent Deaths (Summary by SOC, PT) Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.3.3.1

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active; Combined Placebo;

Overall

Table 14.3.3.4.1 SD: Summary of Serious Treatment-Emergent Adverse Events (Summary by SOC, PT) Protocol: BTI-201 Safety Population

| | | rh | rhu-pgsN | | | ק<br>הלם<br>הלם | Ç | | Overall | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 5cts with at least one Serious TEAE xx (xx.x%) xx | | , <sup>–</sup> | N=XX) | | | (N=XX | 2 | | (N=X) | . × | |
| | | ¤ | (%) W | | | (%) | M | | n (%) | | |
| 271 XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) <td>Subjects with at least one Serious TEAE</td> <td>×)<br/>×</td> <td>(% x . x)</td> <td>×</td> <td>×</td> <td>(xx.x)</td> <td>××</td> <td>×</td> <td>x.xx)</td> <td></td> <td>×</td> | Subjects with at least one Serious TEAE | ×)<br>× | (% x . x) | × | × | (xx.x) | ×× | × | x.xx) | | × |
| 7.1 XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) <td>SOC1</td> <td>××</td> <td>(% X . X)</td> <td>×</td> <td>×</td> <td>(xx.xx)</td> <td>××</td> <td>×</td> <td>XXXXX</td> <td></td> <td>×</td> | SOC1 | ×× | (% X . X) | × | × | (xx.xx) | ×× | × | XXXXX | | × |
| XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) XX (XX,X\$) <td>PT1</td> <td></td> <td>(%x.x%)</td> <td>××</td> <td>×</td> <td>(XX.XX)</td> <td></td> <td>×</td> <td></td> <td></td> <td>×</td> | PT1 | | (%x.x%) | ×× | × | (XX.XX) | | × | | | × |
| PT1 XX (XX, X\$) XX (XX, X\$) XX (XX, X\$) PT2 XX (XX, X\$) XX XX, X\$ XX XX< | SOC2 | | ×. ×. | ×× | × | (xx.xx) | | × | XXXX) | | × |
| PTZ XX (XX, X\$) XX (XX, X\$) XX (XX, X\$) XX (XX, X\$) XX XX, X\$ XX XX XX, X\$ XX X | PT1 | XX (X | (% X . X | ×× | × | (xx.xx) | | × | x.xx) | | × |
| PT3 XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) XX (XX.X\$) <td>PT2</td> <td>XX (X</td> <td>(% X . X</td> <td>××</td> <td>×</td> <td>(xx.x%)</td> <td></td> <td>×</td> <td>x.xx)</td> <td></td> <td>×</td> | PT2 | XX (X | (% X . X | ×× | × | (xx.x%) | | × | x.xx) | | × |
| PT4 XX (XX.X\$) | PT3 | | (% X . X) | ×× | × | (xx.xx) | | × | | | × |
| PT1 XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) XX XX (XX.X\$) PT2 XX (XX.X\$) XX XX (XX.X\$) XX (XX.X\$) XX XX (XX.X\$) PT3 XX (XX.X\$) XX XX (XX.X\$) XX (XX.X\$) XX XX (XX.X\$) PT4 XX (XX.X\$) XX XX (XX.X\$) XX (XX.X\$) XX XX (XX.X\$) PT5 PT6 PT7 PT7 PT7 PT7 PT7 PT7 PT7 | PT4 | | (×.x%) | ×× | × | (XX.XX) | | × | | | × |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | SOC3 | | ×. ×. | ×× | × | (xx.x) | | × | ×. ××) | | × |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | PT1 | | (% X · X) | ×× | × | (xx.xx) | | × | x. xx) | | × |
| $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | PT2 | ×× | (% X . X %) | ×× | × | (xx.xx) | | × | x.xx) | | × |
| $(x \times x \times x) \times x \times (x \times x \times x) \times x \times x \times x \times x \times x \times x \times x \times$ | PT3 | | (% X · X | ×× | × | (xx.x%) | | × | | | × |
| xx (xx.x\$) xx | PT4 | | (% X . X | ×× | × | (xx.xx) | | × | | | × |
| | PT5 | | (% X · X) | ×× | × | (xx.xx) | | × | x.xx) | | × |

Note: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurred or worsened following the first administration of study drug. If a subject has multiple occurrences of a TEAE, the subject is presented only once in the Patient count (n) column for a given System Organ Class and Preferred Term. Occurrences are counted each time in the mentions/Occurrence (M) column. MedDRA Version xx.x

Program: filepath name, Output: filepath name (version x.x) Created: DDMMMYYYY HH:NM Clinical cut-off date: DDMMMYYYY

Table 14.3.3.4.2 MAD: Summary of Serious Treatment-Emergent Adverse Events (Summary by SOC, PT) Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:MM

Programming Note: Repeat Table 14.3.3.4.1

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg;

rhu-pGSN 24 mg/kg; Combined Active; Combined Placebo;

Overall

Table 14.3.3.5.1 SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and NCI-CTCAE Grade) Protocol: BTI-201 Safety Population

| | r | rhu-pgsN | 7 | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | • | 6 mg/kg | | 1 | Placebo | | 0 | Overall | |
| | | (N=XX) | | | (N=XX) | | $\Box$ | (N=XX) | |
| | ľ | n (%) M | 1 | - | n (%) M | | п | n (%) M | |
| Subjects with at least one TEAE | × | xx (xx.x%) xx | ×× | × | xx (xx.x%) | × | × | xx (%x.x%) xx | ×× |
| SOCI | × | (×x.x%) | ×× | × | (×x.x%) xx | ×× | ( ××. ××) ×× | ×. X. | ×× |
| PT1 | × | (××.×%) | × | × | xx (xx.x%) | ×× | ×)<br>×× | (xx.x%) | ×× |
| Grade 1 | × | (×x.x%) | ×× | × | (××.×%) | XX | X) XX | (×x.x×) | ×× |
| Grade 2 | × | (×x.x%) | ×× | × | (××.×%) | ×× | X) XX | (xx.x%) | XX |
| Grade 3 | × | (×x.x%) | ×× | × | XX (XX.X%) | XX | X) XX | (××.××) | ×× |
| Grade 4 | × | (××.×%) | ×× | × | (××.×%) | ×× | X) XX | (××.××) | ×× |
| Grade 5 | × | (××.×%) | ×× | × | (xx.xx) | ×× | XX XX | (xx.xx) | ×× |
| SOC2 | × | xx (xx.x%) | ×× | × | xx (xx.x%) | ×× | xx (xx.x%) | X.X%) | ×× |
| PT1 | × | (XX.X%) | ×× | × | xx (xx.x%) | ×× | X) XX | (XX.X%) | XX |
| Grade 1 | × | (××.××) | × | × | xx (xx.x%) | ×× | ×)<br>×× | (××·××) | ×× |
| Grade 2 | × | (XX.X%) | ×× | × | xx (xx.x%) | ×× | X) XX | (XX.X%) | XX |
| Grade 3 | × | (×x.x%) | ×× | × | xx (xx.x%) | ×× | X) XX | (XX.X%) | XX |
| Grade 4 | × | (×x.x%) | ×× | × | (××.×%) | ×× | X) XX | (××.×%) | ×× |
| Grade 5 | × | (××.×%) | ×× | × | XX (XX.X%) | XX | XX XX | (××.××) | ×× |

Note: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurred or worsened following the first administration of study drug. If a subject has multiple occurrences of a TEAE, the subject is presented only once in the Patient count (n) column for a given System Organ Class and Preferred Term. Occurrences are counted each time in the mentions/Occurrence (M) column. MedDRA Version xx.x

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY

Table 14.3.3.5.2 MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and NCI-CTCAE Grade) Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat Table 14.3.3.5.1 Include: rhu-pGSN 6 mg/kg

rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg;

Combined Active;

Combined Placebo;

Overall

Table 14.3.1.6.1 SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study Drug) Protocol: BTI-201 Safety Population

| | rhu-pGSN<br>6 mg/kg<br>(N=xx) | Placebo<br>(N=xx)<br>n (%) M | Overa<br>(N=X) | Overall (N=xx) | |
|---|---|---|---|---|---|
| Subjects with at least one TEAE | xx (%x.xx) xx | xx (%x.xx) xx | (X) XX | xx (%x.xx) xx | × |
| SOC1 | xx (xx.x%) xx | xx (%x.xx) xx | xx) xx | x (%x.xx) | ×× |
| PT1 | xx (xx.x%) xx | xx (%x.xx) xx | XX) XX | x (%x.xx) | ×× |
| Definitely not Related | xx (xx.x%) xx | xx (%x.xx) xx | XX) XX | x (%x.xx) | ×× |
| Probably not Related | XX (XX.X%) XX | xx (%x.xx) xx | XX) XX | x (%x.xx) | XX |
| Possibly Related | XX (XX.X%) XX | xx (%x.xx) xx | XX) XX | x (%x.xx) | XX |
| Probably Related | XX (XX.X%) XX | xx (%x.xx) xx | XX) XX | x (%x.xx) | ×× |
| Definitely Related | xx (xx.x%) xx | xx (%x.xx) xx | xx) xx | x (%x.xx) | ×× |
| SOC2 | xx (xx.x%) xx | xx (%x.xx) xx | XX) XX | X (%X.XX) | × |
| PT1 | xx (xx.x%) xx | xx (%x.xx) xx | XX) XX | x (%x.xx) | ×× |
| Definitely not Related | xx (xx.x%) xx | xx (%x.xx) xx | XX) XX | ( %x.xx) | ×× |
| Probably not Related | XX (%X.X%) XX | xx (%x.xx) xx | XX) XX | x (%x.xx) | ×× |
| Possibly Related | XX (%X.X%) XX | xx (%x.xx) xx | XX) XX | ( %x.xx) | ×× |
| Probably Related | XX (XX.X%) XX | xx (%x.xx) xx | XX) XX | ( %x.xx) | ×× |
| Definitely Related | XX (XX.X%) XX | xx (%x.xx) xx | xx) xx | (xx.x%) xx | × |

Note: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurred or worsened following the first administration of study drug. If a subject has multiple occurrences of a TEAE, the subject is presented only once in the Patient count (n) column for a given System Organ Class and Preferred Term. Occurrences are counted each time in the mentions/Occurrence (M) column. MedDRA Version  $xx\,.\,x$ 

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Table 14.3.3.6.2 MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study Drug) Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.3.6.1 Include: rhu-pGSN 6 mg/kg;

rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg;

Combined Placebo; Combined Active;

Overall

Table 14.3.3.7.1 SD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study Procedure) Protocol: BTI-201 Safety Population

| | rhu-pGSN<br>6 mg/kg | Placebo | Overall |
|---|---|---|---|
| | (X)=N) (%) u | (N=XX)<br>M (%) u | (N=xx) |
| | | 11 / ) 11 | |
| Subjects with at least one TEAE | xx (xx.x%) xx | xx (%x.xx) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (%x.xx) xx | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (%x.xx) xx | xx (%x.xx) xx |
| Definitely not Related | xx (xx.x%) xx | xx (%x.xx) xx | xx (%x.xx) xx |
| Probably not Related | XX (XX.X%) XX | xx (%x.xx) xx | XX (%X.XX) XX |
| Possibly Related | XX (XX.X%) XX | xx (%x.x%) xx | XX (%X.X%) XX |
| Probably Related | XX (XX.X%) XX | xx (%x.xx) xx | XX (%X.X%) XX |
| Definitely Related | xx (xx.x%) xx | XX (XX.X%) XX | xx (xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |
| | XX (XX.X%) XX | xx (%x.xx) xx | XX (%X.X%) XX |
| Definitely not Related | xx (%x.x%) xx | xx (%x.xx) xx | XX (XX.X%) XX |
| Probably not Related | xx (xx.x%) xx | xx (%x.xx) xx | xx (xx.x%) xx |
| Possibly Related | XX (XX.X%) XX | xx (%x.xx) xx | xx (%x.xx) xx |
| Probably Related | XX (%X.X%) XX | xx (%x.xx) xx | XX (%X.XX) XX |
| Definitely Related | XX (%X.XX) XX | xx (%x.xx) xx | xx (%x.xx) xx |

Note: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurred or worsened following the first administration of study drug. If a subject has multiple occurrences of a TEAE, the subject is presented only once in the Patient count (n) column for a given System Organ Class and Preferred Term. Occurrences are counted each time in the mentions/Occurrence (M) column. MedDRA Version  $xx\,.\,x$ 

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM Clinical cut-off date: DDMMMYYYY

Table 14.3.3.7.2 MAD: Summary of Treatment-Emergent Adverse Events (Summary by SOC, PT and Relationship to Study Procedure)
Protocol: BTI-201
Safety Population

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.3.7.1 Include: rhu-pGSN 6 mg/kg;

rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg;

Combined Placebo; Combined Active;

Overall

Table 14.3.3.8.1 SD: Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation (Summary by SOC, PT)
Protocol: BTI-201
Safety Population

| | Н | rhu-pgsN | Z | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | • | 6 mg/kg | - | Д | Placebo | | Overall | 111 | |
| | | (N=XX) | | | (N=XX) | | (N=XX) | × | |
| | r | n (%) M | Ţ | п | n (%) M | | M (%) u | Σ | |
| Subjects with at least one TEAE Leading to Treatment Discontinuation | × | xx (%x.xx) xx | ×× | ×× | xx (%x.x%) xx | | xx (%x.x%) xx | %<br>× | × |
| SOC1 | × | (%X : XX) | × | ×× | x (%x.xx) xx | × | (%X.XX) | %<br>% | × |
| PT1 | × | xx (xx.x%) | | ×× | | | xx (xx,x%) | | × |
| PT2 | × | (×x.x%) | ×× | ×× | | XX | XX (XX.X%) | %) XX | × |
| PT3 | × | xx (xx.x%) | ×× | ×× | | XX | xx (xx.x%) | %) XX | × |
| PT4 | × | (××.×%) | ×× | ×× | x (%x.xx) xx | × | xx (xx.x%) | %) XX | × |
| PT1 | × | (××.×%) | × | ×× | (×x.x%) | ×× | xx (xx.x%) | (%) XX | × |
| SOC2 | × | xx (xx.x%) | × | ×× | xx (%x.xx) xx | | xx (xx.x%) | (%) XX | × |
| PT1 | × | xx (xx.x%) | ×× | ×× | x (%x.xx) xx | ×× | xx (xx.x%) | | XX |
| PT2 | × | xx (xx.x%) | × | ×× | x (%x.xx) xx | ××× | xx (xx.x%) | | ×× |
| PT3 | × | (××.×%) | × | ×× | x (%x.xx) xx | ××× | xx (xx.x%) | | ×× |
| PT4 | × | (××.×%) | ×× | ×× | x (%x.xx) xx | ×× | xx (xx.x%) | | ×× |
| PT5 | × | xx (xx.x%) | ×× | ×× | x (%x.xx) xx | XX | XX (XX.X%) | | ×× |
| PIG | × | xx (xx.x%) | ×× | ×× | xx (%x.xx) xx | | xx (xx.x%) | xx (%) | × |

Note: A treatment-emergent adverse event (TEAE) is defined as an adverse event that occurred or worsened following the first administration of study drug. If a subject has multiple occurrences of a TEAE, the subject is presented only once in the Patient count (n) column for a given System Organ Class and Preferred Term.

Occurrences are counted each time in the mentions/Occurrence (M) column. MedDRA Version xx.x

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY

Table 14.3.3.8.2 MAD: Summary of Treatment-Emergent Adverse Events Leading to Treatment Discontinuation (Summary by SOC, PT) Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.3.8.1

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg;

rhu-pGSN 24 mg/kg; Combined Active;

Combined Placebo;

Overall


Table 14.3.3.9.1 SD: Summary of Overall Survival Protocol: BTI-201 Safety Population

| | rhu-pgsn: | | |
|---|---|---|---|
| | 6 mg/kg | Placebo | Overall |
| | (N=XX) | (N=xx) | (N=xx) |
| Deaths | | | |
| Number of Subjects that Died | xx (xx.x%) | xx (xx.x%) | (×x.x%) |
| Number of Subjects that did not Die | XX (XX.X%) | XX (XX.X%) | (XX.X%) |
| Survival Time (days) (95% $\mathrm{CI}^1$ ) | | | |
| 25th Percentile | $\times \times $ | $\times \times $ | XX (XX.X, XX.X) |
| Median | $\times \times $ | xx (xx.x, xx.x) | xx (xx.x, xx.x) |
| 75th Percentile | (xxx, xxxx) xx | (x.x, xx, xx) xx | (x, x, x, x, x) |

Note: CI = Confidence Interval; <sup>1</sup>Brookmeyer and Crowley method (1982. Log-log transformation); Overall Survival is defined as the difference (in days) between the time of first study drug administration to the date of death + 1 (Include the day of the study drug administration.) Subjects who did not die will be censored at the study exit visit.

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY

Table 14.3.3.9.2 MAD: Summary of Overall Survival Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat Table 14.3.3.9.1

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active; Combined Placebo; Overall Novotech – Strictly Confidential


Table 14.3.4.1.1.1 SD: Summary of CBC (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

| | | | rhu-pgsN: 6 mg/kg | 6 mg/kg | Placebo (N=xx) | (ebo | Overall (N=xx) | all<br>(x) |
|---|---|---|---|---|---|---|---|---|
| | | | | Change from | | Change from | | Change from |
| Parameter | Visit | | Actual Value | Baseline1 | Actual Value | $Baseline^1$ | Actual Value | Baseline1 |
| Hemoglobin $(g/L)$ | $Baseline^1$ | ч | × | | × | | × | |
| | | Mean | xxx.x | | XXX.X | | x.xxx | |
| | | Median | X.XXX | | XXXX.X | | XXX.X | |
| | | SD | ×.xxx | | xxx.x | | ×××××××××××××××××××××××××××××××××××××× | |
| | | Minimum | ××.× | | XX.X | | ×.×. | |
| | | Maximum | ××.× | | × × × | | × × × | |
| | Day 2 | п | × | | × | | × | |
| | | Mean | XXX.X | | XXX.X | | xxx.x | |
| | | Median | xxx.x | | XXX.X | | x.xxx | |
| | | SD | XXX.X | | XXXX.X | | x.xxx | |
| | | Minimum | ××.× | | ××.× | | ××.× | |
| | | Maximum | ××.× | | ××. | | ××.× | |
| | Day 3 or 4 | ជ | × | × | × | × | × | × |
| | | Mean | XXXX.X | X.XXX | XXXX.X | X.XXX | XXX.X | XXXX.X |
| | | Median | XXX.X | x.xx | XXXX.X | xxxx.x | x.xxx | X.XX.X |
| | | SD | xxx.x | ×.xx | XXX.X | xxx.x | xxx.x | XXX.X |
| | | Minimum | xx.x | xx.x | xx | xx.x | xx.x | x.xx |
| | | Maximum | ××.× | ×. × | ××.× | ××.× | ××.× | xx.x |
| etc. | etc. | | | | | | | |

Include all CBC Parameters and all scheduled time points. Programming Note:

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Table 14.3.4.1.1.2 MAD: Summary of CBC (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.4.1.1.1 Include all CBC Parameters and all scheduled time points.

Include: rhu-pGSN 6 mg/kg;

rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg;

Combined Placebo; Combined Active;

Overall


Table 14.3.4.1.2.1 SD: Summary of CBC Shifts from Baseline (Low, Normal, High) Protocol: BTI-201 Safety Population

| | | | | ${\tt Baseline}^1$ | | |
|---|---|---|---|---|---|---|
| | | | | rhu-pGSN: 6 mg/kg<br>(N=xx) | ۵ | |
| Parameter | Result<br>Classification | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) | Missing<br>n (%) | Total<br>n (%) |
| Hemoglobin (g/L) Day 2 | Low | | | | | |
| | Normal | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | High | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| | Missing | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Total | XX (XX.X%) | (%x.x%) xx | (×x.x%) | (×x.x%) xx | XX (XX.X%) |
| Day 3 or 4 | Low | XX (XX.X%) | (%x.xx) xx | (xx.x%) | (XX.X%) | XX (XX.X%) |
| | Normal | XX (XX.X%) | (×x.x%) xx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | High | XX (XX.X%) | (×x.x%) xx | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| | Missing | xx (xx.x%) | (×.x.) xx | XX (XX.X%) | (%x.xx) xx | XX (XX.X%) |
| | Total | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |

Note <sup>1</sup>Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. Unscheduled visits not included in post baseline assessments.

etc.

etc.

Programming Note: Also Include: Placebo, Overall Include all CBC Parameters and all scheduled time points.

Clinical cut-off date: DDMMMYYYY Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYY HH:MM

Table 14.3.4.1.2.2 MAD: Summary of CBC Shifts from Baseline (Low, Normal, High) Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:
Repeat Table 14.3.4.1.2.1
Include all CBC Parameters and all scheduled time points.

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active; Combined Placebo;

Overall


Table 14.3.4.2.1.1 SD: Summary of Coagulation (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201

Safety Population

| | | | rhu-pgsN: 6 mg/kg | 6 mg/kg | Placebo | sebo | Overall | all |
|---|---|---|---|---|---|---|---|---|
| | | | (X=X) | (x) | (X=X) | (×× | (X=X) | (XX) |
| | | | | Change from | | Change from | | Change from |
| Parameter | Visit | | Actual Value | $Baseline^1$ | Actual Value | $Baseline^1$ | Actual Value | $Baseline^1$ |
| PT/INR (unit) | Baseline¹ | п | × | | × | | × | |
| | | Mean | x.xxx | | XXXX.X | | x.xxx | |
| | | Median | X.XXX | | XXXX.X | | XXXX.X | |
| | | SD | X.XXX | | XXX.X | | XXXX.X | |
| | | Minimum | ××.× | | ××.× | | ××.× | |
| | | Maximum | xx.x | | ××.× | | × × × | |
| | Day 2 | ជ | × | | × | | × | |
| | | Mean | X.XXX | | XXXX.X | | XXXX.X | |
| | | Median | X.XXX | | xxx.x | | ×.xxx | |
| | | SD | X.XXX | | XXXX.X | | X.XXX | |
| | | Minimum | ××.× | | ××.× | | ××.× | |
| | | Maximum | ××.× | | ××. | | × × × | |
| | Dav 3 or 4 | Д | × | × | × | × | × | × |
| | 1 | Mean | XXX.X | ×.xx | xxx.x | ×.×× | ××××× | X.XXX |
| | | Median | x.xx | ×.xxx | XXX.X | ×.xx | x.xxx | XXX.X |
| | | SD | XXXX.X | x.xx | XXXX.X | XXXX.X | xxxx.x | X.XX.X |
| | | Minimum | xx.x | XX.X | ××.× | ××.× | xx.x | XX.X |
| | | Maximum | xx.x | xx.x | ××.× | ××.× | xx.x | x.xx |
| etc. | etc. | | | | | | | |

Include all Coagulation Parameters and all scheduled time points. Programming Note:

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Table 14.3.4.2.1.2 MAD: Summary of Coagulation (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.4.2.1.1

Include all Coagulation Parameters and all scheduled time points.

Include: rhu-pGSN 6 mg/kg;

rhu-pGSN 12 mg/kg;

rhu-pGSN 24 mg/kg;

Combined Active;

Combined Placebo;

Overall

Table 14.3.4.2.2.1 SD: Summary of Coagulation Shifts from Baseline (Low, Normal, High) Protocol: BTI-201 Safety Population

| | | | | | | $Baseline^1$ | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | , I | | | rhu | rhu-pGSN: 6 mg/kg<br>(N=xx) | 1/kg | | |
| Parameter | | Result<br>Classification | Low<br>n (%) | Normal<br>n (%) | al (5) | High<br>n (%) | Missing<br>n (%) | Tota.<br>n (%) | Total<br>n (%) |
| PT/INR (unit) | Day 2 | Low<br>Normal | (×x.xx) xx | (%x.xx) xx | (% X | XX (XX.X%) | (%x.x%) xx | XX (XX.X%) | (% X X |
| | | Hıgh<br>Missing | XX (XX. X%)<br>XX (XX. X%) | xx | √ √ √ √ × | XX (XX. X%) XX (XX. XX. X%) XX (XX. XX. | XX | XX (XX. XX)<br>(% X . XX) XX (%) | X X X X X X X X X X X X X X X X X X X |
| | | Total | XX (XX.X%) | (xx.x%) | % X . | xx (xx.x%) | xx (xx.x%) | xx (xx. x%) | ×. ×. |
| | Day 3 or 4 | Low | XX (XX, X%) | (×.xx) xx | (% X. | xx (xx.x%) | (XX.X%) | (%x.xx) xx | x.x%) |
| | | Normal | XX (XX, XX) XX (X, XX, XX) XX (X, XX, | (XX.X%) XX XX (XX.X%) XX | ○/o o/o | (xx.x%) xx | XX (XX.X%) XX (XX.X%) XX (XX.XX) XX | XX (XX.X%) XX (XX.X%) | (xx.x%)<br>(xx.x%) |
| | | Missing | (%x.xx) xx | (%x.xx) xx | . (%X. | xx (xx.x%) | (%x.xx) xx | ×× | (XX.X%) |
| | | Total | xx (xx.x%) | xx (xx.x%) | . X % | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | X.X%) |
| etc. | etc. | | | | | | | | |

Note 'Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. Unscheduled visits not included in post baseline assessments.

Also Include: Placebo, Overall Programming Note:

Include all Coagulation Parameters and all scheduled time points.

Clinical cut-off date: DDMMMYYYY Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Table 14.3.4.2.2.2 MAD: Summary of Coagulation Shifts from Baseline (Low, Normal, High) Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:
Repeat Table 14.3.4.2.2.1
Include all Coagulation Parameters and all scheduled time points.
Include: rhu-pGSN 6 mg/kg;
rhu-pGSN 12 mg/kg;
rhu-pGSN 24 mg/kg;
Combined Active;
Combined Placebo;

Table 14.3.4.3.1.1 SD: Summary of Comprehensive Metabolic Profile (Summary of Actual and Change from Baseline Values) by Timepoint

Protocol: BTI-201 Safety Population


| | | | rhu-pGSN: 6 mg/kg | 6 mg/kg | Plac | Placebo | Overall | all |
|---|---|---|---|---|---|---|---|---|
| | | | (X=XX) | (X) | (N=XX) | (XX) | (N=XX) | (x) |
| | | | | Change from | | Change from | | Change from |
| Parameter | Visit | | Actual Value | ${\tt Baseline}^1$ | Actual Value | ${\tt Baseline}^1$ | Actual Value | Baseline1 |
| Sodium (unit) | $Baseline^1$ | п | × | | × | | × | |
| | | Mean | XXXX.X | | X.XXX | | X.XXX | |
| | | Median | X.XXX | | X.XXX | | XXX.X | |
| | | SD | XXXX.X | | X.XXX | | X.XXX | |
| | | Minimum | XX.X | | ××.× | | ×.×. | |
| | | Maximum | × × × | | × × × | | × × × | |
| | | 1 | : | | ; | | ; | |
| | Day 2 | п | × | | × | | × | |
| | | Mean | XXXX.X | | ×.xx | | ×.xx | |
| | | Median | XXXX.X | | X.XXX | | X.XXX | |
| | | SD | XXXX.X | | x.xx | | x.xxx | |
| | | Minimum | XX.X | | ××.× | | ××.× | |
| | | Maximum | × × × | | ××.× | | × × × | |
| | Day 3 or 4 | ч | × | × | × | × | × | × |
| | | Mean | XXXX.X | X.XXX | X.XXX | XXXX.X | XXXX.X | XXXX.X |
| | | Median | xxx.x | x.xx | xxxx.x | xxx.x | x.xxx | XXXX.X |
| | | SD | XXXX.X | x.xx | x.xx | XXXX.X | XXX.X | X.XX.X |
| | | Minimum | xx.x | xx.x | ××.× | ××.× | ××.× | x.xx |
| | | Maximum | ××.× | ×. × | ××.× | ××.× | ××.× | ××.× |
| etc. | etc. | | | | | | | |

Note: SD: Standard Deviation

Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Unscheduled visits not included in post baseline assessments.

Programming Note: Include all Comprehensive Metabolic Profile Parameters and all scheduled time points.

Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMYYYY Program: filepath\_name, Output: filepath\_name (version x.x) Table 14.3.4.3.1.2 MAD: Summary of Comprehensive Metabolic Profile (Summary of Actual and Change from Baseline Values) by Timepoint

Protocol: BTI-201 Safety Population

Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x)

Programming Note:

Repeat Table 14.3.4.3.1.1

Include all Comprehensive Metabolic Profile Parameters and all

scheduled time points.

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg;

Combined Active;

Combined Placebo;

Overall

Table 14.3.4.3.2.1 SD: Summary of Comprehensive Metabolic Profile Shifts from Baseline (Low, Normal, High) Protocol: BTI-201 Safety Population

| | | | | | Baseline. | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | H | rhu-pGSN: 6 mg/kg<br>(N=xx) | / kg | | |
| Parameter | | Result<br>Classification | Low<br>n (%) | Normal<br>n (%) | High<br>n (%) | Missing<br>n (%) | Total<br>n (%) | |
| Sodium (unit) | Day 2 | Low | | | | | | |
| | | Normal | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | 00 |
| | | High | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%) |
| | | Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | (%) |
| | | Total | xx (xx.x%) | (xx.x%) | xx (xx.x%) | (XX.X%) | (%x.x%) xx | 0/0 |
| Ι | Day 3 or 4 | Low | xx (xx.x%) | (×x.x%) | (××.×%) | (××.××) ×× | xx (xx.x%) | 0/0 |
| | | Normal | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | 00 |
| | | High | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | 00 |
| | | Missing | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | (%)<br>(%) |
| | | Total | (%x.xx) xx | (%X.XX) XX | (%x.x%) xx | (×x.x%) xx | xx (xx.x%) | (lo |
| etc. | etc. | | | | | | | |

Note 'Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. Unscheduled visits not included in post baseline assessments.

Programming Note: Also Include: Placebo, Overall Include all Comprehensive Metabolic Profile Parameters and all scheduled time points.

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Table 14.3.4.3.2.2 MAD: Summary of Comprehensive Metabolic Profile Shifts from Baseline (Low, Normal, High) Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.4.3.2.1

Include all Comprehensive Metabolic Profile Parameters and all

scheduled time points.

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg;

rhu-pGSN 24 mg/kg;

Combined Active;

Combined Placebo;

Overall


Table 14.3.4.4.1 SD: Summary of Vital Signs (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201

Safety Population

| | | | rhu-pGSN | rhu-pGSN: 6 mg/kg | Д | Placebo | Overall | :a11 |
|---|---|---|---|---|---|---|---|---|
| | | | =N) | (N=xx) | | (N=XX) | (N=XX) | (xx) |
| | | | | Change from | Actual | Change from | | Change from |
| Parameter | Visit | | Actual Value | Baseline <sup>1</sup> | Value | $Baseline^1$ | Actual Value | Baseline1 |
| ()<br>()<br>()<br>()<br>()<br>() | ()<br>()<br>()<br>() | Ş | : | | ; | | | |
| Systemate brood | DASGLLIG- | 11 | × | | × | | | |
| pressure (mmHg) | | Mean | X.XXX | | xxx.x | | | |
| | | Median | x.xxx | | ××××× | | | |
| | | SD | ×.xxx | | ×××. | | | |
| | | Minimum | xx.x | | ××.× | | | |
| | | Maximum | ×.×. | | ××.× | | | |
| | Day 1: End of<br>Infusion | п | × | × | × | × | × | × |
| | | Mean | ×.xxx | ×.xxx | ×××. | ×.xx | xxx.x | ×.xx |
| | | Median | X.XXX | X.XX.X | ×××××× | xxx.x | x.xxx | XXXX.X |
| | | SD | XXXX.X | ×.xxx | ×××××× | xxx.x | XXXX.X | ×.xx |
| | | Minimum | XX.X | XX.X | ××.× | XX.XX | X. XX | XX.X |
| | | Maximum | × × × | ×××× | ××. | ×× × | × × × | × × × × |
| | Day 1: 30 mins | п | × | × | × | × | × | × |
| | | Mean | X.XXX | X.XX.X | xxx.x | XXXX.X | XXXX.X | X.XXX |
| | | Median | x.xxx | x.xxx | xxx.x | x.xx | XXXX.X | x.xx |
| | | SD | X.XXX | X.XXX | xxx.x | XXXX.X | XXXX.X | X.XXX |
| | | Minimum | XX.X | XX.X | ××.× | XX.XX | X.XX | XX.X |
| | | Maximum | ××.× | × . × | ××.× | XX.XX | X. XX | ×.xx |
| etc. | etc. | | | | | | | |

Note: SD: Standard Deviation

1-Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Unscheduled visits not included in post baseline assessments.

Include all Vital Signs Parameters and all time points. Programming Note:

Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Table 14.3.4.4.2 MAD: Summary of Vital Signs (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.4.4.1 Include all Vital Sign Parameters and all scheduled time points.

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg;

rhu-pGSN 24 mg/kg; Combined Active;

Combined Placebo;

Overall
Table 14.3.4.5.1 SD: Summary of Vital Signs Interpretation by Timepoint Protocol: BTI-201 Safety Population

| Visit | | rhu-pGSN: 6 mg/kg<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| ${\tt Baseline}^1$ | n<br>Normal | (% X X X X X X X X X X X X X X X X X X X | ( | (% X X X X X X X X X X X X X X X X X X X |
| | Abnormal NCS<br>Abnormal CS | XX (XX.X%)<br>XX (XX.X%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
| Day 1: 30 mins | n<br>Lama | ×× × · · · · | X X X | (%: :::) ::: |
| | Abnormal NCS<br>Abnormal CS | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | (\$x.xx)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| Day 2 | n<br>Normal | xx<br>xx (xx.x%) | xx<br>xx (xx.x%) | xx<br>xx (xx.x%) |
| | Abnormal NCS<br>Abnormal CS | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
| etc. | etc. | | | |

Note: SD: Standard Deviation

 $<sup>^{1}</sup>$ Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. NCS = Not Clinically Significant, CS = Clinically Significant. Unscheduled visits not included in post baseline assessments.

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMYYYY

Table 14.3.4.5.2 MAD: Summary of Vital Signs Interpretation by Timepoint Protocol:  ${\tt BTI-201}$  Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat Table 14.3.4.5.1 Include all scheduled time points. Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active; Combined Placebo;


Table 14.3.4.6.1 SD: Summary of Mean EKG (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BII-201

Safety Population

| | | | rhu-pgsN | rhu-pGSN: 6 mg/kg | Д | Placebo | Overall | all |
|---|---|---|---|---|---|---|---|---|
| | | | =N) | (N=XX) | | (N=xx) | (N=XX) | (×× |
| | | | | Change from | Actual | Change from | | Change from |
| Parameter | Visit | | Actual Value | ${\tt Baseline}^1$ | Value | ${\tt Baseline}^1$ | Actual Value | Baseline <sup>1</sup> |
| Heart Rate (unit) Baseline | Baseline¹ | ជ | × | | × | | | |
| | | Mean | X.XX.X | | ×.xxx | | | |
| | | Median | X.XXX | | ×.xxx | | | |
| | | SD | X.XXX | | ×.xxx | | | |
| | | Minimum | X.XX | | ××.× | | | |
| | | Maximum | ×<br>×<br>× | | ××. | | | |
| | Day 28 / Early<br>Termination | п | × | × | × | × | × | × |
| | | Mean | X.XXX | XXXX.X | ×.xxx | XXXX.X | XXXX.X | X.XXX |
| | | Median | X.XXX | X.XXX | ×.xxx | XXXX.X | XXXX.X | X.XXX |
| | | SD | X.XXX | x.xx | ×.xxx | XXXX.X | xxx.x | XXXX.X |
| | | Minimum | xx.x | x.xx | ××.× | x.xx | xx.x | ××.× |
| | | Maximum | ××. | ×. ×× | ×. × | ×. × | × × × | ××.× |
| PR Interval (unit) Baseline <sup>1</sup> | $Baseline^1$ | п | × | | × | | × | |
| | | Mean | xxx.x | | ×××××× | | xxx.x | |
| | | Median | X.XXX | | ××××. | | ×.xxx | |
| | | SD | X.XXX | | ×.xxx | | x.xxx | |
| | | Minimum | XX.X | | ××.× | | XX.X | |
| | | Maximum | XX.X | | ××.× | | XX.X | |
| etc. | etc. | | | | | | | |

Note: SD: Standard Deviation

1-Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Unscheduled visits not included in post baseline assessments.

Include all EKG Parameters and all time points. Programming Note:

Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Table 14.3.4.6.2 MAD: Summary of Mean EKG (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.4.6.1 Include all EKG Parameters and all scheduled time points.

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active;

Combined Placebo;

Overall


Table 14.3.4.7.1 SD: Summary of EKG Interpretation (Worst) by Timepoint Protocol: BTI-201

Safety Population

| Placebo Overall (N=xx) (N=xx) | xx | XX XX XX (XX.X%) |
|---|---|---|
| rhu-pGSN: 6 mg/kg<br>(N=xx) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | ( |
| | n<br>Normal<br>Abnormal NCS<br>Abnormal CS | n<br>Normal<br>Abnormal NCS<br>Abnormal CS |
| Visit | Baseline <sup>1</sup> | Day 28 / Early<br>Termination |

Note: SD: Standard Deviation

Clinical cut-off date: DDMMMYYYY Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

 $<sup>^{1}</sup>$ Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. NCS = Not Clinically Significant, CS = Clinically Significant. Unscheduled visits not included in post baseline assessments.

Table 14.3.4.7.2 MAD: Summary of EKG Interpretation (Worst) by Timepoint Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat Table 14.3.4.7.1 Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active; Combined Placebo; Novotech – Strictly Confidential


Table 14.3.4.8.1 SD: Summary of CURB-65 Score(Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201

Safety Population

| | | rhu-pGSN<br>(N= | rhu-pGSN: 6 mg/kg<br>(N=xx) | Д | Placebo (N=xx) | Overall (N=xx) | all<br>(x) |
|---|---|---|---|---|---|---|---|
| | | | | Actual | Change from | | $\circ$ |
| Visit | | Actual Value | $Baseline^1$ | Value | ${\tt Baseline}^1$ | Actual Value | Baseline <sup>1</sup> |
| $Baseline^1$ | п | × | | × | | | |
| | Mean | xxx.x | | x.xx | | | |
| | Median | xxx.x | | x.xx | | | |
| | SD | XXX.X | | xxx.x | | | |
| | Minimum | XX.X | | ××.× | | | |
| | Maximum | XX.X | | ×.xx | | | |
| Day 3 or 4 | ជ | × | × | × | × | × | × |
| | Mean | ××××× | XXX.X | x.xx | XXX.X | X.XXX | XXXX.X |
| | Median | xxx.x | XXXX.X | x.xx | x.xxx | x.xx | XXXX.X |
| | SD | xxx.x | XXXX.X | XXXX.X | XXX.X | X.XXX | XXXX.X |
| | Minimum | ××.× | ××.× | ××.× | XX.X | x.xx | XX.XX |
| | Maximum | x. x | ××.× | × × × | xx.x | ××.× | ×. xx |
| Day 7 | п | × | × | × | × | × | × |
| | Mean | xxx.x | xxx.x | x.xx | XXX.X | x.xx | XXXX.X |
| | Median | ××××× | XXX.X | x.xx | XXX.X | X.XXX | XXXX.X |
| | SD | ××××× | XXX.X | x.xx | XXX.X | X.XXX | XXXX.X |
| | Minimum | ××.× | ××.× | ××.× | XX.X | x.xx | XX.XX |
| | Maximum | ××.× | ××.× | ×. × | ××.× | xx.x | XX.X |
| etc. | | | | | | | |

Note: SD: Standard Deviation

Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Unscheduled visits not included in post baseline assessments.

Include all scheduled time points. Programming Note:

Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMYYYY Program: filepath\_name, Output: filepath\_name (version x.x) Table 14.3.4.8.2 MAD: Summary of CURB-65 Score (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.4.8.1 Include all scheduled time points.

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg;

rhu-pGSN 24 mg/kg; Combined Active;

Combined Placebo;

Overall


Table 14.3.4.9.1 SD: Summary of PSI Score (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

| | | rhu-pGSN | rhu-pgsN: 6 mg/kg | | Placebo | Overall | all |
|---|---|---|---|---|---|---|---|
| | | =X) | (N=XX) | | (N=XX) | (x=N) | (× |
| | | | Change from | Actual | Change from | | $\mathcal{O}$ |
| Visit | | Actual Value | Baseline1 | Value | Baseline1 | Actual Value | Baseline <sup>1</sup> |
| Baseline <sup>1</sup> | ۵ | × | | × | | | |
| | Mean | ×××××××××××××××××××××××××××××××××××××× | | × × × × | | | |
| | Median | ××××× | | ×××.× | | | |
| | SD | XXX.X | | ×××.× | | | |
| | Minimum | XX.X | | ×. × | | | |
| | Maximum | x. x | | ×. × | | | |
| Day 3 or 4 | п | × | × | × | × | × | × |
| | Mean | XXXX.X | X.XXX | ×.xxx | X.XXX | X.XXX | XXXX.X |
| | Median | XXXX.X | X.XXX | ×.xxx | X.XXX | X.XXX | XXXX.X |
| | SD | XXX.X | X.XXX | XXX.X | X.XXX | XXXX.X | XXXX.X |
| | Minimum | XX.X | ××.× | ××.× | xx.x | xx.x | XX.X |
| | Maximum | x.xx | xx.x | ××.× | ××.× | xx.x | x.xx |
| Day 7 | п | × | × | × | × | × | × |
| | Mean | ×××××× | xxxx.x | xxx.x | xxx.x | xxxx.x | xxx.x |
| | Median | xxx.x | x.xx | xxx.x | x.xxx | XXXX.X | xxx.x |
| | SD | XXX.X | XXXX.X | x.xx | X.XXX | XXXX.X | XXXX.X |
| | Minimum | x.xx | X.XX | ××.× | × × | XX.X | xx.x |
| | Maximum | XX.X | XX.XX | ××.× | ××.× | XX.X | ××.× |
| etc. | | | | | | | |

Note: SD: Standard Deviation

1-Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Unscheduled visits not included in post baseline assessments.

Include all scheduled time points. Programming Note:

Clinical cut-off date: DDMMMYYYY Program: filepath\_name, Output: filepath\_name (version x.x)

Created: DDMMMYYYY HH:MM

Table 14.3.4.9.2 MAD: Summary of PSI Score (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.4.9.1 Include all scheduled time points.

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active;

Combined Placebo;

Overall


Table 14.3.4.10.1 SD: Summary of PSI Risk Class by Timepoint Protocol: BTI-201 Safety Population

| Visit | Risk Class | ho = ho | Placebo (N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| | | | (1) | |
| $Baseline^1$ | п | ×× | ×× | ×× |
| | Class I | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Class II | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Class III | (%x.x%) xx | xx (xx.x%) | xx (xx.x%) |
| | Class IV | (%x.xx) xx | (×x.x%) xx | xx (xx.x%) |
| | Class V | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| Day 28 / Early Termination | ч | ×× | ×× | × |
| | Class I | (XX.X%) | (xx.x%) | xx (xx.x%) |
| | Class II | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Class III | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| | Class IV | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| | Class V | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Note: SD: Standard Deviation

 $^{1}$ Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. NCS = Not Clinically Significant, CS = Clinically Significant. Unscheduled visits not included in post baseline assessments.

Clinical cut-off date: DDMMYYYY
Program: filebath name, Outbut: filebath name (versi

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Table 14.3.4.10.2 MAD: Summary of PSI Risk Class by Timepoint Protocol:  $\rm BTI-201$  Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat Table 14.3.4.10.1 Include all scheduled time points. Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active; Combined Placebo; Overall Novotech – Strictly Confidential


Table 14.3.4.11.1 SD: Summary of SOFA Score (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

| | | | ., | | | ( | r |
|---|---|---|---|---|---|---|---|
| | | rhu-pgsn | rhu-pGSN: 6 mg/kg | ш | Placebo | Overall | all |
| | | =Z) | (N=xx) | | (N=XX) | (x=x) | (X) |
| | | | Change from | Actual | Change from | | Change from |
| Visit | | Actual Value | $Baseline^1$ | Value | $Baseline^1$ | Actual Value | Baseline <sup>1</sup> |
| $Baseline^1$ | n | × | | × | | | |
| | Mean | xxx.x | | xxx.x | | | |
| | Median | XXXX.X | | x.xx | | | |
| | SD | XXX.X | | xxx.x | | | |
| | Minimum | X.XX | | ××.× | | | |
| | Maximum | XX.X | | ××.× | | | |
| Day 3 or 4 | п | × | × | × | × | × | × |
| | Mean | XXX.X | XXXX.X | ×.×× | x.xxx | ××××× | XXX.X |
| | Median | XXX.X | XXXX.X | ×.×× | x.xxx | ××××× | XXX.X |
| | SD | XXX.X | XXXX.X | xxx.x | XXXX.X | xxx.x | XXXX.X |
| | Minimum | X.XX | X. XX | ××.× | xx.x | ××.× | X.xx |
| | Maximum | XX.X | ××.× | × × × | × × × | ××.× | ×.xx |
| Day 7 | п | × | × | × | × | × | × |
| | Mean | x.xx | XXXX.X | ×.xx | x.xxx | xxx.x | x.xxx |
| | Median | x.xx | XXXX.X | ×.xx | X.XXX | xxx.x | XXXX.X |
| | SD | XXXX.X | X.XXX | x.xx | XXXX.X | XXXX.X | XXXX.X |
| | Minimum | X.XX | ×.xx | ××.× | XX.X | ××.× | X.XX |
| | Maximum | xx.x | x.xx | ×××× | x.xx | xx.x | x.xx |

etc.

Include all scheduled time points. Programming Note:

Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMYYYY Program: filepath\_name, Output: filepath\_name (version x.x)

Note: SD: Standard Deviation

Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Unscheduled visits not included in post baseline assessments.

Table 14.3.4.11.2 MAD: Summary of SOFA Score (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat Table 14.3.4.11.1 Include all scheduled time points.

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg;

rhu-pGSN 24 mg/kg; Combined Active;

Combined Placebo;

Overall


Table 14.3.4.12.1 SD: Summary of MMSE Score (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

| | | rhu-pgsN | rhu-pGSN: 6 mg/kg | Н | Placebo | Overall | 111 |
|---|---|---|---|---|---|---|---|
| | | =N) | (N=XX) | | (N=xx) | (x=N) | (X) |
| | | | Change from | Actual | Change from | | Change from |
| Visit | | Actual Value | Baseline1 | Value | $Baseline^1$ | Actual Value | Baseline1 |
| ${	t Baseline}^1$ | п | × | | × | | | |
| | Mean | XXXX.X | | x.xx | | | |
| | Median | XXXX.X | | xxx.x | | | |
| | SD | XXXX.X | | ××××× | | | |
| | Minimum | X. XX | | ××.× | | | |
| | Maximum | X. XX | | ××.× | | | |
| Day 3 or 4 | п | × | × | × | × | × | × |
| | Mean | XXXX.X | xxx.x | xxx.x | x.xxx | xxx.x | xxx.x |
| | Median | XXXX.X | xxx.x | xxx.x | x.xxx | xxx.x | xxx.x |
| | SD | XXXX.X | XXXX.X | XXXX.X | X.XXX | XXX.X | XXXX.X |
| | Minimum | X.XX | ××.× | ××. × | ××.× | ××.× | xx.x |
| | Maximum | XX.X | × × × | ××.× | × . × | × × × | ×. ×. |
| Day 7 | п | × | × | × | × | × | × |
| | Mean | XXXX.X | xxx.x | x.xx | x.xxx | ××××× | xxx.x |
| | Median | XXXX.X | xxx.x | xxx.x | x.xxx | xxx.x | xxx.x |
| | SD | XXXX.X | XXX.X | XXXX.X | X.XXX | XXXX.X | XXXX.X |
| | Minimum | X.XX | ××.× | ××. × | ××.× | ××.× | xx.x |
| | Maximum | X.XX | x.xx | ××.× | ×. × | xx.x | XX.X |
| etc. | | | | | | | |

Include all scheduled time points. Programming Note:

Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY Program: filepath\_name, Output: filepath\_name (version x.x)

Note: SD: Standard Deviation

1-Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Unscheduled visits not included in post baseline assessments.

Table 14.3.4.12.2 MAD: Summary of MMSE Score (Summary of Actual and Change from Baseline Values) by Timepoint Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note:

Repeat Table 14.3.4.12.1 Include all scheduled time points.

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg;

rhu-pGSN 24 mg/kg; Combined Active;

Combined Placebo;

Overall


| Hospitalization | | |
|-----------------------|-------------------|-------------------|
| Summary of F | | |
| Table 14.3.4.13.1 SD: | Protocol: BTI-201 | Safety Population |

| Parameter (Kaplan-Meier Estimates) | rhu-pGSN: 6 mg/kg<br>(N=xx) | Placebo<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|
| Hospital Stay<br>Number of Subjects Discharged | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of Subjects not Discharged | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Length of Stay in Hospital (hours) (95% $\mathrm{CI}^1$ ) | | | |
| 25th Percentile | xx (xx.x, xx.x) | (x.x., x.x) $xx$ | xx (xx.x, xx.x) |
| Median | xx (xx.x, xx.x) | (x, x, x, x, x) | xx (xx.x, xx.x) |
| 75th Percentile | XX (XX.X, XX.X) | xx (xx.x, xx.x) | XX (XX.X, XX.X) |
| ICU Stay | | | |
| Number of Subjects in ICU | xx (xx.x%) | (×x.x%) | xx (xx.x%) |
| Number of Subjects not in ICU | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) |
| Length of Stay in ICU (days) (95% $\mathrm{CI}^1$ ) | | | |
| 25th Percentile | XX (XX.X, XX.X) | (x, x, x, x, x) | $\times \times $ |
| Median | xx (xx.x, xx.x) | $\times \times (\times \times $ | $\times \times (\times \times $ |
| 75th Percentile | XX (XX.X, XX.X) | XX (XX.X, XX.X) | XX (XX.X, XX.X) |
| Intubation | | | |
| Number of Subjects Intubated | xx (xx.x%) | (×x.x%) | xx (xx.x%) |
| Number of Subjects not Intubated | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Length of Intubation (days) (95% $\mathrm{CI}^1$ ) | | | |
| 25th Percentile | xx (xx.x, xx.x) | xx (xx.x, xx.x) | $x \times (x \times x, x \times x)$ |
| Median | (x.x. (x.x. x) xx.x) | (x, x, x, x, x) | xx (xx.x, xx.x) |
| 75th Percentile | xx (xx.x, xx.x) | XX (XX.X, XX.X) | XX (XX.X, XX.X) |

Note: CI = Confidence Interval; <sup>1</sup>Brookmeyer and Crowley method (1982. Log-log transformation); Length of stay in hospital is defined as the date and time of discharge/date of study exit (23:59 PM) - date and time of hospitalization admission due to CAP in hours

Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x)

Table 14.3.4.13.2 MAD: Summary of Hospitalization Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: Repeat Table 14.3.4.13.1 Include all scheduled time points.

Include: rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg; Combined Active; Combined Placebo; Overall Novotech – Strictly Confidential


## BTI-201: Mock Listings: Table of Contents

## Listings

| TO A A LA LA LA CARACTER TOOK | × |
|---|---|
| Listing 16.2.4.4.1 SD: Pregnancy Test Results | 18 |
| | 101 |
| 10.2.4.4.2 MAD: FIEGIICY 1ESC | T3 |
| Listing 16.2.4.5.1 SD: Confirmation of CAP | 20 |
| Listing 16.2.4.5.2 MAD: Confirmation of CAP | 21 |
| Listing 16.2.4.6.1 SD: Eligibility Assessment | 22 |
| 16.2.4.6.2 MAD: | 23 |
| 16.2.4.7.1 SD: P | 24 |
| 16.2.4.7.2 | 25 |
| Listing 16.2.5.1.1 SD: Randomization | 26 |
| 16.2.5.1.2 | 27 |
| Listing 16.2.5.2.1 SD: Study Drug Administration | 28 |
| Listing 16.2.5.2.2 MAD: Study Drug Administration | 29 |
| Listing 16.2.5.3.1 SD: Study Drug Interruption | 30 |
| Listing 16.2.5.3.2 MAD: Study Drug Interruption | 31 |
| 16.2.6.1.1 SD: Individual pGSN | 32 |
| 16.2.6.1.2 MAD: Individual | 33 |
| Listing 16.2.6.2.1 SD: Individual Estimated Plasma rhu-pGSN Concentrations (unit) | 34 |
| Listing 16.2.6.2.2 MAD: Individual Estimated Plasma rhu-pGSN Concentrations (unit) | 35 |
| Listing 16.2.6.3.1 SD: Individual pGSN Plasma PK Parameters | 36 |
| Listing 16.2.6.3.2 MAD: Individual pGSN Plasma PK Parameters by Day | 37 |
| 16.2.6.4.1 SD: Individual Estimated Plasma rhu-pGSN PK E | 38 |
| Listing 16.2.6.4.2 MAD: Individual Estimated Plasma rhu-pGSN PK Parameters by Day | 39 |

| Listing 16.2.6.5.1 SD: Anti-rhu-pGSN Antibodies | . 40 |
|---------------------------------------------------------------|------|
| 16.2.6.5.2 MAD: Ant | 41 |
| Listing 16.2.6.6.1 SD: Biomarkers | 42 |
| 16.2.6.6 | 43 |
| 16.2.6.7. | . 44 |
| 16.2.6.7.2 MAD: | 45 |
| 16.2.7.1.1 SD: Adverse Events | 46 |
| Listing 16.2.7.1.2 MAD: Adverse Events | 47 |
| 16.2.7.2.1 SD: Serious A | 48 |
| 16.2.7.2.2 | 49 |
| 16.2.7.3.1 | 50 |
| sting 16.2.7.3.2 | 51 |
| isting 16 | 52 |
| 16.2.7.4.2 | 53 |
| Listing 16.2.8.1.1.1 SD: CBC | 54 |
| $\vdash$ | 55 |
| 16.2.8.1.2.1 SD: A | 56 |
| 16.2.8.1.2 | 57 |
| 16.2.8.2 | 58 |
| 16.2.8.2.1.2 MAD: | 59 |
| 16.2.8.2.2.1 SD: A | 60 |
| 16.2.8.2.2.2 MAD: Abnormal | 61 |
| 16.2.8.3.1.1 SD: Comprehensive | 62 |
| 16.2.8.3.1.2 | 63 |
| 16.2.8.3 | 64 |
| .8.3.2 | 65 |
| Listing 16.2.9.1 SD: Vital Signs | 66 |
| 16.2.9.2 MAD: Vital | 67 |
| 16.2.10.1 SD: EKG | . 68 |
| 16.2.10.2 MAD: | 69 |
| Listing 16.2.11.1 SD: Physical Examination | 70 |
| 16.2.11.2 | 71 |
| Listing 16.2.12.1.1 SD: Outcome Prediction Models CURB-65 | 72 |
| 16.2.12.1.2 MAD: Outcome Predic | 73 |
| sting 16.2.12.2.1 SD: Outcome Predict | 74 |
| 16.2.12 | . 75 |
| 16.2.12 | 76 |
| Listing 16.2.12.3.2 MAD: Outcome Prediction Models SOFA Score | 77 |
| 16.2.12.4. | . 78 |
| Listing 16.2.12.4.2 MAD: Outcome Prediction Models MMSE Score | 79 |

## **GENERAL COMMENTS**

```
Unless otherwise states, parameters will be listed in alphabetical order
```

Change from Baseline:

Change from Baseline will be calculated as:

Change from baseline = new value - baseline value

Names and order of Treatment Groups

Cohort 1: rhu-pGSN 6 mg/kg;

Cohort 1: Placebo

MAD:

Cohort 2: rhu-pGSN 6 mg/kg;

Cohort 2: Placebo

Cohort 3: rhu-pGSN 12 mg/kg;

Cohort 3: Placebo

Cohort 4: rhu-pGSN 24 mg/kg;

Cohort 4: Placebo

Names of visits

SD:

Screening

Day 1 Day 2

Day 3/4

Day 7

Day 14

Day 28 / Early Termination (Combined visit for safety and efficacy)

Unscheduled

MAD:

Screening

Day 1

Day 2

Day 3

Day 4

Day 7

Day 14

Novotech - Strictly Confidential

- Day 28 / Early Termination (Combined visit for safety and efficacy)
  - Unscheduled

- Column widths and text-wrapping may be altered in final output in order to best present the data Footnotes may be added/amended if required

| 0 |
|-----------------------|
| V1.0 |
| <u>_</u> |
| eu |
| Ξ |
| pu |
| ē |
| ¥ |
| 0 |
| 2 |
| 2 |
| , Final V2.0 Amendmer |
| := |
| tings, F |
| 200 |
| Sti |
| $\Box$ |
| EOS Listings, |
| Ы |
| 쏭 |
| ě |
| 2 |
| S |
| atı |
| t stat |
| $\overline{}$ |
| je |
| _ |
| ⋾ |
| noc |
| Docume |

2018-12-03

Listing 16.2.1.2.1 SD: Subject Disposition Protocol: BTI-201 Intent-to-Treat Population


Cohort 1: rhu-pGSN 6 mg/kg

| Subject | Final Disposition | Reason for Discontinuation | Date of Study Exit (DDMMYYYY) | Date of Last Contact (DDMMMYYYY) |
|---|---|---|---|---|
| | | Due to Adverse Event: | | |
| XXX | Withdrawn | AE#: XXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY |
| XXX | Completed | | DDMMMYYYY | |
| XXX | Completed | | DDMMMXXXX | |
| XXX | Withdrawn | Other: XXXXXXXXXXXX | DDMMMYYYY | |
| etc. | | | | |

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM


Listing 16.2.1.2.2 MAD: Subject Disposition Protocol: BTI-201 Intent-to-Treat Population Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.1.2.1 for MAD.

| Protocol No: BTI-201 | Document status: Mock EOS L | Document status: Mock EOS Listings, Final V2.0 Amendment V1.0 | 2018-12-0 |
|---|---|---|---|
| Listing 16.2.2.1 SD: Protocol Deviation<br>Protocol: BTI-201<br>Intent-to-Treat Population | eviations | | |
| Cohort 1: rhu-pGSN 6 mg/kg | | | |
| Subject | Type of Deviation | Date of Deviation (DDWMMYYYY) | Description of Deviation |
| XXX | ABCD | DDMMMYYYY | ABCD |
| | ABCD | DDMMYYYY | ABCD |
| : | | | |
| XXX | ABCD | DDMMMYYYY | ABCD |
| | ABCD | DDMMMYYYY | ABCD |
| : | | | |
| XXX | ABCD | DDMMMXXXX | ABCD |
| | ABCD | DDMMMYYY | ABCD |
| i | | | |
| XXX | ABCD | DDMMMYYYY | ABCD |
| XXX | ABCD | DDMMMYYY | ABCD |

2018-12-03

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMNYYYY HH:MM

Clinical cut-off date: DDMMMYYYY

Page x of x

Listing 16.2.2.2 MAD: Protocol Deviations Protocol: BTI-201 Intent-to-Treat Population


Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.2.1 for MAD.

Listing 16.2.3.1 SD: Analysis Populations Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| ocol | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Per Protocol<br>Population | Yes | Yes | Yes | Yes | Yes | Yes | Yes | |
| PK<br>Population | Yes | Yes | Yes | Yes | Yes | Yes | Yes | |
| Safety<br>Population | Yes | Yes | Yes | Yes | Yes | Yes | Yes | |
| Intent-to-Treat<br>Population | Yes | Yes | Yes | Yes | Yes | Yes | Yes | |
| Subject | XXX | XXX | XXX | XXX | XXX | XXX | XXX | Etc. |

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:MM

2018-12-03

Listing 16.2.3.2 MAD: Analysis Populations Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.3.1 for MAD.


Listing 16.2.4.1.1 SD: Demographics and Baseline Characteristics Protocol:  $\mathtt{BTI-201}$ 

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | Date of<br>Informed<br>Consent | Protocol | Date of<br>Birth | Age at<br>Informed | | Child<br>Bearing | Contraceptive | | Height | Weight |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | (DDMMMXXXX) | Version | (DDMMMYYYY) | Consent | S e x | Potential | | Race | (cm) | (kg) |
| XXX | DDMMMYYYY | Amendment 1 | DDMMMXYYY | ×× | Male | | | White | ××× | ×. × |
| XXX | DDMMMXXXX | Amendment 1 | DDMMMYYYY | ×× | Female | No | | White | XXX | ××.×× |
| XXX | DDMMMXYYY | Amendment 1 | DDMMMXXXX | ×× | Male | | | White | XXX | x.xx |
| | | | | | | | Hormonal | Other: | | |
| XXX | DDMMMXXXX | Amendment 1 | DDMMMXXXX | ×× | Female | Yes | methods | XXXXXXXXX | ××× | ×.×× |
| etc. | | | | | | | | | | |

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Listing 16.2.4.1.2 MAD: Demographics and Baseline Characteristics Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.4.1.1 for MAD.


Listing 16.2.4.2.1 SD: Viral Serology Protocol: BTI-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Subject | Visit | Visit Date (DDMMMYYYY | Test | Result | Most Recent<br>Viral Load<br>(unit) | Most Recent<br>CD4 Count<br>(unit) |
|---|---|---|---|---|---|---|
| XXX | Screening | DDMMYYYYY | HIV<br>Hepatitis B | Negative<br>Negative | ×××××× | ×:<br>×:<br>×: |
| | | | Surrace Antigen<br>Hepatitis C | Negative | | |
| XXX | Screening | DDMMMYYYY | HIV | Negative | XXXXXX | x.xx |
| | | | Hepatitis B | Negative | | |
| | | | Hepatitis C | Negative | | |
| etc. | | | | | | |

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Listing 16.2.4.2.2 MAD: Viral Serology Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.4.2.1 for MAD.

Listing 16.2.4.3.1 SD: Medical History Protocol: BTI-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Subject | Condition/<br>Body System | System Organ Class /<br>Preferred Term | Date of<br>Diagnosis<br>(DDMMMYYYY) | Resolution Date (DDMMMYYYY) | Concomitant<br>Medication<br>Taken | Ongoing |
|---|---|---|---|---|---|---|
| XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX YYYYYYYY/<br>ZZZZZZZZ | DDMMMYYYY | DDMMMYYYY | No | No |
| | XXXXXXXXXXXXXXX/ | XXXXXXXXX/ YYYYYYYY/ ZZZZZZZZZ | DDMMMYYYY | DDMMMYYYY | Yes | Yes |
| <br>XXX | /XXXXXXXXXXX | XXXXXXXXX/ YYYYYYYY/ | DDMMMYYYY | DDMMMXXXX | No | NO |
| XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXX YYYYYXX<br>ZZZZZZZZZZZZZZZ | DDMMMYYYY | DDMMMYYYY | | |
| XXX | /XXXXXXXXXXXX | /XXXXXXXX/ XXXXXXXXX | DDMMMYYYY | ZZZZMMMQQ | No | No |
| XXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXX YXXYYYYX XXXXXXXXXXXXXXXXXX | DDMMMYYYY | DDMMMYYYY | No | No |

Note: MedDRA Version XX.X

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

2018-12-03

Listing 16.2.4.3.2 MAD: Medical History Protocol: BTI-201
Intent-to-Treat Population
Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.4.3.1 for MAD.

Listing 16.2.4.4.1 SD: Pregnancy Test Results Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Sample Date/ Time (DDMMMYYY/ HH:MM) Sample Type Result | DDMMMYYY/HH:MM Urine Negative DDMMMYYY/HH:MM Urine Negative | DDMMMYYY/ HH:MM Serum Negative DDMMMYYY/ HH:MM Urine Negative DDMMMYYY/ HH:MM Urine | DDMMMYYY/ HH:MM Serum Negative DDMMMYYY/ HH:MM Urine Negative DDMMMYYY/ HH:MM Urine |
|---|---|---|---|
| Visit | Screening<br>Day 1<br>Day 28 / Early<br>Termination | Screening<br>Day 1<br>Day 28 / Early<br>Termination | Screening<br>Day 1<br>Day 28 / Early<br>Termination |
| Assessment Performed -<br>Reason Not Performed Vi | Yes Solater Parameters | Yes Sc<br>Da | Yes<br>Da<br>Da |
| Subject | XXX | XXX | XXX |

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Clinical cut-off date: DDMMMYYYY
Listing 16.2.4.4.2 MAD: Pregnancy Test Results Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.4.4.1 for MAD. 2018-12-03

Listing 16.2.4.5.1 SD: Confirmation of CAP Protocol: BTI-201 Intent-to-Treat Population

| | , | | à |
|---|------|---|---------------|
| | 3 | | |
| | ٥ | | ) |
| | Z | 2 | 4 |
| į | j | ( | ) |
| į | | 1 | ) |
| | 5 | | 2 |
| | 1 | | |
| | 1111 | | |
| | 2 | | 1111 |
| , | | | |
| | | | 111 |
| | 1505 | | 111 |
| | ( | | 110101 |
| | | | OTION OT OTTO |
| | ( | | OTION OT OTTO |

| | | | | | Was CXR or | | | Date and Time of | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Was there | CT Scan | | Date and Time of | Hospitalization | |
| | | | Was there | radiological | Performed: | | presentation to | Admission due to | |
| | | | clinical | confirmation | Date | CXR or CT | the hospital | CAP | |
| | | Visit Date | confirmation | of CAP (CXR | Performed | Scan | /AAAWWWQQ) | /XXXWWWQQ) | Subject |
| Subject Visit | Visit | (DDMMMYYY) | of CAP | or CT) | (DDMMMYYY) | Findings | HH: MM) | HH: MM) | Randomized |
| | | | | | Yes: | | | | |
| XXX | Screening | DDMMMYYYY | Yes | Yes | DDMMMXXXX | XXXXXXXXX | DDMMYYYY/ HH:MM | DDMMYYYY/ HH:MM | Yes |
| | | | | | Yes: | | | | |
| XXX | Screening | DDMMMYYYY | Yes | Yes | DDMMMXXXX | XXXXXXXXX | DDMMYYYYY/ HH:MM | DDMMYYYYY/ HH:MM | Yes |
| | | | | | Yes: | | | | |
| XXX | Screening | DDMMMYYYY | Yes | Yes | DDMMMXXXX | XXXXXXXXX | DDMMYYYYY HH:MM | DDMMMYYYY HH:MM | Yes |
| etc. | | | | | | | | | |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.4.5.2 MAD: Confirmation of CAP Protocol: BTI-201
Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.4.5.2 for MAD.

Listing 16.2.4.6.1 SD: Eligibility Assessment Protocol: BTI-201


Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Subject | Eligibility Assessment Date (DDWMWYYYY) | Did the patient meet all inclusion criteria? | Inclusion<br>criterion<br>not met | Did the patient meet all exclusion criteria? | Exclusion<br>Criterion<br>not met |
|---|---|---|---|---|---|
| XXX | DDMMMXXXX | Yes | | X<br>& O | |
| XXX | DDMMMXXXX | Yes | | Yes | |
| XXX | DDMMMXXXX | Yes | | Yes | |
| XXX | DDMMMAXXX | Yes | | Yes | |
| XXX | DDMMMXXXX | Yes | | Yes | |
| XXX | DDMMMXXXX | Yes | | Yes | |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.4.6.2 MAD: Eligibility Criteria Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.4.6.1 for MAD.


2018-12-03

Listing 16.2.4.7.1 SD: Prior Medications Protocol: BTI-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Route | 2222 | 22222 | 22222 | 22222 | 2222 | |
|---|---|---|---|---|---|---|
| Frequency | XXXXXX | YYYYY | XXXXXX | YYYYY | XXXXXX | |
| Unit | Unit | Unit | Unit | Unit | Unit | |
| Dose | XX | × | × | × | × | |
| Ongoing | ON | No | O N | No | O<br>N | |
| Start Date/<br>Stop Date<br>(DDMMMYYYY) | DDMMAXXXX<br>/ XXXX | DDMMMYYYY / | DDMMMYYYY / | DDMMMYYYY / | DDMMMYYYY / | |
| Indication | Pre-existing<br>condition: MH# | Other: YYYYYY | Other: YYYYYY | Other: YYYYYY | Pre-existing condition: MH# | |
| Drug Name/ATC3/PT | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| CM# | Π | 0 | П | 0 | Н | |
| Subject<br>Number | ××× | | XXX | | XXX | Etc. |

Note: Prior medications are defined as any medication where the use was stopped prior to the first administration of the study medication.

WHO-DD, XXXXXXXXX

Clinical cut-off date: DDMMMYYYY

Listing 16.2.4.7.2 MAD: Prior Medications
Protocol: BTI-201
Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.4.7.1 for MAD.

| 0 |
|------------------------|
| V1.0 |
| `>' |
| <b>–</b> |
| $\subseteq$ |
| ഉ |
| ≽ |
| Þ |
| - |
| Ĕ |
| 5 |
| V2.0 / |
| 0. |
| 7 |
| > |
| æ |
| , Final V2.0 , |
| gs, |
| ΞĘ |
| istii |
| Listin |
| <b>JS Listin</b> |
| EOS Listin |
| EOS Listings, Fin |
| ck EOS Listin |
| lock EOS Listin |
| <b>Mock EOS Listin</b> |
| : Mock EOS Listin |
| us: Mock EOS Listin |
| tus: Mock |
| tus: Mock |
| tus: Mock |
| it status: Mock |
| it status: Mock |
| it status: Mock |
| it status: Mock |
| it status: Mock |
| ocument status: Mock |
| it status: Mock |

2018-12-03

| : Randomization | | Population |
|--------------------|-------------------|---------------------|
| SD: | | 11/2 |
| Listing 16.2.5.1.1 | Protocol: BTI-201 | Intent-to-Treat Por |


Cohort 1: rhu-pGSN 6 mg/kg

| Subject | Date /Time of<br>Randomization<br>(DDMMYYYY/ HH:MM) | Randomization Number | Date /Time of<br>Emergency Unblinding<br>(DDWMMYYYY/ HH:MM) | Reason for Emergency Unblinding |
|---|---|---|---|---|
| XXX | DDMMYYYYY/ HH:MM | XXXXX | | |
| XXX | DDMMMYYYYY/ HH:MM | XXXXX | | |
| XXX | DDMMMXXXX HH: MM | XXXXX | | |
| XXX | DDMMMYYYYY/ HH:MM | XXXXX | DDMMMYYYY/ HH:MM | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX | DDMMMXXXX HH: MM | XXXXX | | |
| XXX | DDMMMYYYY/ HH:MM | XXXXX | | |
| etc. | | | | |

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:MM


Listing 16.2.5.1.2 MAD: Randomization Protocol: BTI-201 Intent-to-Treat Population


Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.5.1.1 for MAD.

Listing 16.2.5.2.1 SD: Study Drug Administration Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | | | | | | | | No - XXXXXXXXX | Day 1 | XXX |
|---|---|---|---|---|---|---|---|---|---|---|
| ×× | ×× | | Yes | HH:MM | DDMMMYYYY/ HH:MM | HH:MM | DDMMMYYYY/ HH:MM | Yes | Day 1 | XXX |
| ×× | ×× | | Yes | HH:MM | DDMMMYYYY/ HH:MM | HH: MM | DDMMYYYYY HH:MM | Yes | Day 1 | XXX |
| | ×× | XXXXXXXXXXX | No | HH:MM | DDMMMYYYY/ HH:MM | HH: MM | /XXXXWWWQQ | Yes | Day 1 | XXX |
| ×× | ×× | | Yes | HH:MM | DDMMMYYYY/ HH:MM | HH: MM | /XXXXWWQQ | Yes | Day 1 | XXX |
| ×× | ×× | | Yes | HH:MM | DDMMMYYYY HH: MM | HH:MM | DDMMYYYYY HH: MM | Yes | Day 1 | XXX |
| - minutes) | - (mr) | Administered | Prescribed | | HH:MM) | HH:MM) | (DDMMYYYYY HH:MM) | reason) | Visit | Subject Visit |
| Interruptions | red | Successfully | per Dose | / X X / | / XXXXWWWQQ) | cion | of Injection | no, provide | | |
| (Including | Volume (1 | Reason not | Administered | tion | of Injection | / Time | Start Date, | Administered? (If Start Date/ Time | | |
| of Injection | of | | Study Drug | Time, | Stop Date/ Time | | | Was Study Drug | | |
| Total Duration | Tota | | | | | | | | | |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.5.2.2 MAD: Study Drug Administration Protocol: BTI-201
Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

| | | | | | | | | Total Duration |
|---|---|---|---|---|---|---|---|---|
| | | Was Study Drug | | Stop Date/ Time | Study Drug | | | of Injection |
| | | Administered? (If | Administered? (If Start Date/ Time of | of Injection | Administered | Reason not | Volume | (Including |
| | | no, provide | Injection | /XXXXMMDD) | per Dose | Successfully | Administered | Interruptions |
| Subject Visit | Visit | reason) | (DDMMMYYYY/ HH:MM) | HH:MM) | Prescribed | Administered | (mT) | - minutes) |
| XXX | Day 1 | Yes | DDMMMYYYY/ HH:MM | DDMMYYYY/ HH:MM | Yes | | XX | XX |
| | Day 2 | Yes | DDMMMXXXX/ HH:MM | DDMMMYYYY HH: MM | Yes | | ×× | ×× |
| | Day 3 | Yes | DDMMMYYYY/ HH:MM | DDMMYYYYY HH:MM | No | XXXXXXXXXXXX | XX | XX |
| XXX | Day 1 | Yes | DDMMMYYYY HH: MM | DDMMYYYY/ HH:MM | Yes | | XX | ×× |
| | Day 2 | Yes | DDMMMYYYY/ HH:MM | DDMMYYYY/ HH:MM | Yes | | XX | XX |
| | Day 3 | No - XXXXXXXXX | | | | | | |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.5.3.1 SD: Study Drug Interruption Protocol: BTI-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Reason for Interruption | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|
| Date and Time of Date and Time of Interruption Injection Re-start (DDMMMYYYY/ HH:MM) (DDMMMYYYY/ HH:MM) | DDMMMYYYY HH:MM | DDMMMYYYY/ HH:MM<br>DDMMMYYYY/ HH:MM<br>DDMMMYYYY/ HH:MM |
| Date and Time of Interruption (DDMMMYYYY/ HH:MM) | DDWMYYYY/ HH:MM<br>DDWMYYYY/ HH:MM | DDWMYYYY/ HH:MM<br>DDWMYXYY/ HH:MM<br>DDWMYXYY/ HH:MM |
| Interruption | П П О | н н н |
| Visit | Day 1<br>Day 1 | Day 1<br>Day 1<br>Day 1 |
| Subject Visit | ×××<br>××× | XXX<br>XXX<br>XXX |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.5.3.2 MAD: Study Drug Interruption Protocol: BII-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Reason for Interruption | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|
| Date and Time of<br>Injection Re-start<br>(DDWMMYYYY/ HH:MM) | DDMMYYYYY HH:MM DDMMYYYYY HH:MM DDMMYYYYY HH:MM DDMMYYYYY HH:MM |
| Date and Time of Interruption (DDWMMYYYY/ HH:MM) | DDWMYYYYY HH: MM DDWMYYYYY HH: MM DDWMYYYYY HH: MM DDWMYYYYY HH: MM |
| Interruption | |
| Visit | Day 1<br>Day 2<br>Day 1<br>Day 3<br>Day 1 |
| Subject Visit | × |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.6.1.1 SD: Individual pGSN Plasma Concentrations (unit) Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

Comments from Pre-Injection / Placebo Ratio Injection from Pre-Ratio from Pre-Injection Ratio Day 1 tration Concen-(ng/mL) Deviation Time of PK Sample Collection (HH:MM) PK Sample Collection (DDMMMYYYY) Date of Collected? Was PK Sample Sampling Time of Dose on Dosing Day /XXXXWWWQQ) Date/Time HH:MM) Day Subject Number

| XXXXXXX | | | | | | | | XXXXXXXX | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | ×.×. | XX.X | XX.X | ××.× | ××.× | ×.×× | | ×.×. | XX.X | XX.X | XX.X | XX.XX | XX.XX |
| | XX.X | xx.x | XX.X | ××.× | ××.× | ××.× | | ×.×. | ××.× | ×.xx | XX.X | XX.X | XX.X |
| XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| xx mins | suim xx | xx hours | xx hours | xx hours | xx hours | xx hours | xx mins | xx mins | xx hours | xx hours | xx hours | xx hours | xx hours |
| HH: MM | HH: MM | HH: MM | HH: MM | HH: MM | HH: MM | HH: MM | нн: мм | HH: MM | HH: MM | HH: MM | HH: MM | HH: MM | HH: MM |
| DDMMMXXX | XXXXMMMQQ | DDMMMYYYY | DDMMMXXXX | DDMMMXXXX | DDMMMXXXX | DDMMMXXXX | DDMMMXXXX | DDMMMXYYY | DDMMMYYYY | DDMMMXXXX | DDMMMXXXX | DDMMMXXXX | DDMMMXXXX |
| Yes | Yes | Yes | Yes | Yes | Yes | Yes | Y<br>es | Yes | Yes | Yes | Yes | Yes | Yes |
| Pre-Injection | 5 to 10 mins | 2 hours post | 8 hours post | 12 hours post | 16 hours post | 24 hours post | Pre-Injection | 5 to 10 mins post | 2 hours post | 8 hours post | 12 hours post | 16 hours post | 24 hours post |
| DDMMMYYYY/<br>HH:MM | | | | | | | DDMMMYYYY/<br>HH:MM | | | | | | |
| $\vdash$ | | | | | | | П | | | | | | |
| XXX | | | | | | | XXX | | | | | : | |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.6.1.2 MAD: Individual pGSN Plasma Concentrations (unit) Protocol: BTI-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Comments | XXXXXXX | | | | | | | XXXXXXXX | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Ratio<br>from Pre-<br>Injection<br>/ Placebo<br>Ratio<br>from Pre-<br>Injection | >> | < × | ××.× | XX.X | ××.× | ×.×. | | XX. | XX.X | XX.X | XX.X | XX.X | ×.×. |
| Ratio<br>from Pre-<br>Injection<br>Day 1 | >> | < ×: ×: | XX.X | XX.X | ××.× | XX.XX | | XX.X | ×.×. | XX.X | XX.X | XX.X | X.XX |
| Concentration (ng/mL) | XXX | S X | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Time<br>Deviation | xx mins | xx hours | xx hours | xx hours | xx hours | xx hours | xx mins | xx mins | xx hours | xx hours | xx hours | xx hours | xx hours |
| Time of PK Sample Collection (HH:MM) | HH: MM | . нн<br>НН: ММ | HH: MM | HH: MM | HH: MM | HH: MM | нн: мм | HH:MM | HH: MM | HH: MM | HH: MM | HH: MM | HH: MM |
| Date of PK Sample Collection | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMXXXX | DDMMMYYYY | DDMMMXXXX | DDMMMYYYY | DDMMMXXXX | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY |
| Was PK<br>Sample<br>Collected? | Z S | v v v | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| Sampling Time | Pre-Injection | post<br>2 hours post | 8 hours post | 12 hours post | 16 hours post | 24 hours post | Pre-Injection | 5 to 10 mins post | 2 hours post | 8 hours post | 12 hours post | 16 hours post | 24 hours post |
| Date/Time of Dose on Dosing Day (DDMMMYYYY/ HH:MM) | DDMMMYYYY/<br>HH:MM | | | | | | DDMMMYYYY/<br>/YYYYY | | | | | | |
| Day | Н | | | | | | 7 | | | | | | |
| Subject<br>Number | ××× | | | | | | | | | | | : | |

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMNYYYY HH:MM

Listing 16.2.6.2.1 SD: Individual Estimated Plasma rhu-pGSN Concentrations (unit) Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

× Placebo Change from from Pre-Injection) Thiertion) (Change - (Mean Pre-Injection from Pre-Change tration (ng/ml.) Concen-Deviation Time Time of
PK Sample
Collection
(HH:MM) Date of PK Sample Collection (DDMMMYYYY) Collected? Was PK Sample Sampling Time of Dose on Dosing Day /XXXXWWMQQ) Date/Time HH:MM) 727 Subject

| Comments | XXXXXXXX | | | | | | | | | XXXXXXXX | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Deviation (ng/mL) Day 1 Injection) Comments | | ××.× | | XX.X | ×.xx | XX.X | XX.X | ××.× | | X.X | ××.× | XX.X | XX.X | ×.×× | XX.X |
| Day 1 | | ××.× | | XX.X | ××.× | ×.×× | ×.×× | ××.× | | ××.× | ××.× | ×.×× | XX.X | ××.× | ××.× |
| (ng/mr) | XXX | XXX | | XXX | XXX | XXX | XXX | XXX | XXX | ××× | XXX | XXX | XXX | XXX | XXX |
| | xx mins | xx mins | | xx hours | xx hours | xx hours | xx hours | xx hours | xx mins | xx mins | xx hours | xx hours | xx hours | xx hours | xx hours |
| (HH:MM) | HH: MM | HH:MM | | HH: MM | HH: MM | HH: MM | HH: MM | HH:MM | HH: MM | HH: MM | HH: MM | HH: MM | HH: MM | HH: MM | HH:MM |
| COTTECTED? (DUMMMYYYY) (HH:MM) | DDMMMYYYY | DDMMMYYYY | | DDMMMYYYY | DDMMMXXXX | DDMMMXXXX | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMXXXX | DDMMMXXXX | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY |
| | Yes | Yes | | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| Sampling Time | Pre-Injection | 5 to 10 mins | post | 2 hours post | 8 hours post | 12 hours post | 16 hours post | 24 hours post | Pre-Injection | 5 to 10 mins post | 2 hours post | 8 hours post | 12 hours post | 16 hours post | 24 hours post |
| | DDMMMYYYYY/<br>HH:MM | | | | | | | | DDMMMYYYY/<br>/YYYYMM | | | | | | |
| Day | $\vdash$ | | | | | | | | П | | | | | | |
| Number | ××× | | | | | | | | XXX | | | | | : | |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.6.2.2 MAD: Individual Estimated Plasma rhu-pGSN Concentrations (unit) Protocol: BTI-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Comments | XXXXXXXX | | | | | | | | XXXXXXXX | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (Change<br>from Pre-<br>Injection)<br>- (Mean<br>Placebo<br>Change from<br>Pre-<br>Injection) | | ××.× | XX.X | XX.X | XX.X | XX.X | ××.× | | X.XX | ×.×. | XX.X | XX.X | XX.X | ××.× |
| Change<br>from Pre-<br>Injection<br>Day 1 | | ××.× | ×.×. | XX.X | XX.X | XX.X | ××.× | | XX.X | ×.xx | XX.X | XX.X | XX.X | XX.X |
| Concentration (ng/mL) | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| Time<br>Deviation | xx mins | xx mins | xx hours | xx hours | xx hours | xx hours | xx hours | suim xx | xx mins | xx hours | xx hours | xx hours | xx hours | xx hours |
| Time of<br>PK Sample<br>Collection<br>(HH:MM) | HH: MM | HH: MM | HH: MM | HH: MM | HH: MM | HH: MM | HH:MM | HH: MM | HH: MM | HH:MM | HH: MM | HH: MM | HH: MM | HH:MM |
| Date of<br>PK Sample<br>Collection<br>(DDMMMYYYY) | DDMMMXYYY | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMXXXX | DDMMMYYYY | DDMMMXYYY | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMXXXX |
| Was PK<br>Sample<br>Collected? | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| Sampling Time | Pre-Injection | 5 to 10 mins | post<br>2 hours post | 8 hours post | 12 hours post | 16 hours post | 24 hours post | Pre-Injection | 5 to 10 mins post | 2 hours post | 8 hours post | 12 hours post | 16 hours post | 24 hours post |
| Date/Time of Dose on Dosing Day (DDMMMYYYY/ HH:MM) | DDMMMYYYY/<br>/YYYYYHH: | | | | | | | DDMMMYYYY/<br>HH:MM | | | | | | |
| Subject<br>Number Day | XXX 1 | | | | | | | 7 | | | | | • | |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.6.3.1 SD: Individual pGSN Plasma PK Parameters Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

Day 1

| DN Cmax | ×. × | ×. × | ×. ×. | ×. ×. | × × × | × · × × | |
|---|---|---|---|---|---|---|---|
| Tmax kel t <sub>14</sub> CL/F V <sub>Z</sub> /F (unit) (unit) (unit) %AUC <sub>ext</sub> DN_AUC <sub>O-t</sub> DN_AUC <sub>O-8</sub> DN_AUC <sub>O-inf</sub> DN_C <sub>max</sub> | × × × | × · × × | × | × × × | × × × | ×. × | |
| DN_AUC <sub>0-8</sub> | ×.× | ×. × | ×. ×× | × × × | × × × | ×. × | |
| DN_AUC <sub>0-t</sub> | × × × | × × × | × × × | × × × | × × × | × · × | |
| %AUC <sub>ext</sub> | ×. × | ××.× | ××.× | ××.× | ××. | x . x | |
| $V_z/F$ (unit) | ×. ×. | ×.× | ×.× | ×××× | ×.× | x.xx | |
| CL/F<br>(unit) | ×.<br>×. | ×.× | ××.× | ××.× | ××.× | xx.x | |
| th (unit) | ×. ×× | ××.× | ××.× | ××.× | ××.× | XX.X | |
| k <sub>el</sub><br>(unit) | ×. × | ××.× | ××.× | ××.× | ××.× | XX.X | |
| T <sub>max</sub><br>(unit) | ×.× | ××.× | ××.× | xx.x | ××.× | xx.x | |
| C <sub>max</sub> (unit) | ×. ×× | ××.× | ××.× | ××.× | ××.× | XX.X | |
| AUC <sub>0-inf</sub><br>(unit) | ×. ×× | ××.× | ××.× | ××.× | ××.× | xx.x | |
| AUC <sub>0-8h</sub> / | × × × | ×.× | ××.× | ××.× | ××.× | xx.x | |
| AUC <sub>0-t</sub><br>(unit) | ×.× | ××.× | ××.× | ××.× | ××.× | x . x | |
| Subject<br>Number | XXX | XXX | XXX | XXX | XXX | XXX | : |

Clinical cut-off date: DDMMMYYYY

2018-12-03

Listing 16.2.6.3.2 MAD: Individual pGSN Plasma PK Parameters by Day Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

Day 1

| N Gmax | ×.× | ××.× | ××.× | ××.× | ××.× | xx.x | |
|---|---|---|---|---|---|---|---|
| Tmax kel th CL/F Vz/F (unit) (unit) (unit) %AUCext DN_AUCO-t DN_AUCO-8 DN_AUCO-inf DN_Cmax | ×. ×. | ××.× | ××.× | ××.× | × × × | × × × | |
| DN_AUC <sub>0-8</sub> | ×. × | ×. × | ×. × | ×. × | × × × | × × × | |
| DN_AUC <sub>0-t</sub> | ××. | ×. × | ×.× | ×.× | ×.× | ×.× | |
| %AUC <sub>ext</sub> | ××. | × × × | × × × | ××.× | × × × | ××. | |
| $V_z/F$ (unit) | ×××× | ×.× | ×.× | ×.× | ×.× | ××. | |
| CL/F<br>(unit) | ××. | ××.× | ××.× | ××.× | ××.× | ××.× | |
| tي<br>(unit) | ×. ×× | ×.× | ××.× | ××.× | ××.× | ××.× | |
| k <sub>el</sub><br>(unit) | ××. | ××.× | ××.× | ××.× | ××.× | ××.× | |
| T <sub>max</sub><br>(unit) | ××. | ××.× | ××.× | ××.× | ××. | ××. | |
| C <sub>max</sub> (unit) | ××. | ××.× | ××.× | ××.× | ××. | ××. | |
| AUC <sub>0-inf</sub> C <sub>max</sub> (unit) | ×. ×× | ××.× | ××.× | ××.× | ××.× | ××. | |
| AUC <sub>0-8h</sub> & (unit) | ××. | ××.× | ××.× | ××.× | ××.× | ××.× | |
| AUC <sub>0-t</sub><br>(unit) | × × × | ××.× | ××.× | ××.× | ××.× | ××.× | |
| Subject<br>Number | XXX | XXX | XXX | XXX | XXX | XXX | : |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.6.4.1 SD: Individual Estimated Plasma rhu-pGSN PK Parameters Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

Day 1

| | 8 DN C <sub>max</sub> | × × × | ×.×. | ××. | ××. | ×. ×. | × . × | |
|---|---|---|---|---|---|---|---|---|
| | DN_AUC <sub>0-8</sub> | ×. ×. | ×.× | × × × | × × × | ××. | × × × | |
| a Analysis | DN_AUC <sub>0-t</sub> | × × × | ×. ×. | ××. | ××. | × × × | × | |
| Double Delta Analysis | C <sub>max</sub> (unit) DN AUC <sub>0-t</sub> DN AUC <sub>0-8</sub> | XX.X | ××.× | ××. | ××. | ××. | ×.× | |
| | AUC <sub>0-8h</sub><br>(unit) | ×.×× | ×.× | × × × | × × × | ×.× | × × × | |
| | AUC <sub>0-t</sub><br>(unit) | ×.× | ××.× | ××. | ××. | ××. | × × × | |
| | DN C <sub>max</sub> | ×.× | ×.× | × × × | × × × | ×. × | × . × | |
| ion | DN_AUC0-8 | x. xx | ××.× | × × × | × × × | × × × | × × | |
| Change from Pre-Injection | DN_AUC <sub>0-t</sub> | ×. ×. | ×.×× | xx.x | xx.x | ×. ×× | ×.×× | |
| thange fro | C <sub>max</sub><br>(unit) | x.xx | ×. ×× | ××. | ××. | ×. ×× | ×. ×× | |
| 0 | AUC <sub>0-8h</sub><br>(unit) | x.xx | ×. ×× | ××. | ××. | ××. | ×. ×× | |
| | AUC <sub>0-t</sub><br>(unit) | ×.× | ××.× | ××. | ××. | ××. | × × × | |
| | Subject<br>Number | XXX | XXX | XXX | XXX | XXX | XXX | : |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.6.4.2 MAD: Individual Estimated Plasma rhu-pGSN PK Parameters by Day Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

Day 1

| | 0-8 DN C <sub>max</sub> | ×.×. | ××.× | | × × × | | |
|---|---|---|---|---|---|---|---|
| <br>S | DN AUC | × × × | x.xx | ×××× | × × × | x.xx | × |
| ta Analysi | DN_AUC0-t | ×<br>×<br>× | ××.× | ×. × | × × × | ××. | ××.× |
| Double Delta Analysis | AUC <sub>0-8h</sub><br>(unit) C <sub>max</sub> (unit) DN_AUC <sub>0-t</sub> DN_AUC <sub>0-8</sub> | × × × | ××.× | ×. × | × × × | × × × | × |
| | | × × × | ×. ×× | ×. × | × × × | × × × | ××. |
| | AUC <sub>0-t</sub><br>(unit) | × | × × × | ×.×× | × × × | × × × | ××. |
| | DN C <sub>max</sub> | × × × | × × × | × × × | × × × | × × × | × × × |
| tion | DN_AUC <sub>0-t</sub> DN_AUC <sub>0-8</sub> | ×. × | x.xx | ×.× | × × × | × × × | × × × |
| Change from Pre-Injection | DN_AUC <sub>0-t</sub> | ×.× | x.xx | ×.×× | ××. | x.xx | ×. ×× |
| Change fro | C <sub>max</sub> (unit) | ×. ×× | ×.× | ×. × | ×. ×× | ×.× | ×. ×. |
| 0 | AUC <sub>0-8h</sub><br>(unit) | ×. ×× | x.xx | ×. ×× | ×. ×× | x.xx | ×.×× |
| | AUC <sub>0-t</sub><br>(unit) | × × × | × × × | × . × | × × × | ××. | × |
| | Subject<br>Number | XXX | XXX | XXX | XXX | XXX | XXX |

Clinical cut-off date: DDMMMYYYY

Listing 16.2.6.5.1 SD: Anti-rhu-pGSN Antibodies Protocol: BTI-201
Intent-to-Treat Population Cohort 1: rhu-pGSN 6 mg/kg

Programming Note: Listing shell will be updated once data transfer agreement is available.

Listing 16.2.6.5.2 MAD: Anti-rhu-pGSN Antibodies Protocol: BTI-201
Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note:
Repeat Listing 16.2.6.5.1 for MAD.
Include all time points and all parameters.

Listing 16.2.6.6.1 SD: Biomarkers Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Subject | Parameter (Unit) | Study Visit | Sample Date/ Time (DDMMMXYYY/<br>HH:MM) | Actual<br>Value | Change from<br>Baseline | Reference<br>Ranges | High/ Low<br>Flag | Comments |
|---|---|---|---|---|---|---|---|---|
| XXX | Procalcitonin (unit) | Day $1^*$ | ММ:НН /ХХХХМММОО | × | | xx , xx | | |
| | | Day 2 | DDMMMYYYY/ HH:MM | × | | XX, XX | | |
| | | Day 3 | DDMMMYYYY/ HH:MM | × | × | xx, xx | н | |
| | | Day 4 | DDMMYYYYY/ HH:MM | × | ×× | XX, XX | L | |

Etc. Etc.

Note: \*Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. L = Below Normal Range, H = Above Normal Range

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x)

Programming Note: Include all time points and all parameters.

Created: DDMMMYYYY HH:MM

Listing 16.2.6.6.2 MAD: Biomarkers Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note:
Repeat Listing 16.2.6.6.1 for MAD.
Include all time points and all parameters.

Listing 16.2.6.7.1 SD: Sputum and Blood Culture Protocol: BII-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | Result | | | |
|---|---|---|---|---|
| Genomic | Immunoassay Diagnostic Test | | | |
| Results | Immunoassay | | | |
| Antigen | Detection | | | |
| | Gram-Stains | | | |
| Date/Time of | Collection | DDMMMYYYY/ | /XXXXWWMQQ | |
| Sputum Culture<br>Collected - Reason | Subject Study Visit Not Performed | Yes | Yes | |
| | Study Visit | Screening | Screening | |
| | Subject | XXXXX | XXXXX | etc. |

Clinical cut-off date: DDMMMYYYY

Programming Note: Include all time points and all parameters.

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM


Listing 16.2.6.7.2 MAD: Sputum and Blood Culture Protocol: BTI-201
Intent-to-Treat Population
Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.6.7.1 for SD.

Listing 16.2.7.1.1 SD: Adverse Events Protocol: BTI-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| TEAE | K e s | Yes | ON | Yes | |
|---|---|---|---|---|---|
| Outcome | Recovered /<br>Resolved | Recovered /<br>Resolved | Recovered /<br>Resolved | Recovered /<br>Resolved | |
| Other<br>Action | None | None | None | None | |
| Action<br>Taken<br>with<br>Study<br>Drug | None | None | None | Drug<br>withdrawn | |
| Relationship<br>to Study<br>Procedure | Possibly<br>Related | Definitely<br>not Related | Definitely<br>not Related | Definitely<br>not Related | |
| Relationship<br>to Study Drug | Possibly<br>Related | Definitely<br>not Related | Definitely<br>not Related | Definitely<br>not Related | |
| Severity<br>(NCI-<br>CTCAE) | Grade 1 | Grade 1 | Grade 1 | Grade 1 | |
| SAE | Yes | Y<br>e<br>s | N | No | |
| Start Date/<br>Stop Date/<br>(DDMMMYYYY/<br>DDMMMYYYY) | DDMMMYYYYY/<br>HH:MM<br>DDMMMYYYY/<br>DDMMMYYYYY/ | DDMMMYYYYY/<br>HH: MM<br>DDMMMYYYY/<br>DDMMMYYYY/ | DDWMMYYYYY/<br>HH:MM<br>DDMMYYYY/<br>DDMMYYYY/<br>DDMMYYYYY/ | DDMMMYYYY /<br>Ongoing | |
| Adverse Event Verbatim/<br>System Organ Class/<br>Preferred Term | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| AE# | $\vdash$ | 0 | $\vdash$ | ~ | |
| Subject<br>Number | XXX | | XXX | | etc. |

Note: TEAE = A treatment-emergent adverse event. MedDRA Version xx.x

Clinical cut-off date: DDMMMYYYY

Listing 16.2.7.1.2 MAD: Adverse Events Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.7.1.1 for MAD.


Listing 16.2.7.2.1 SD: Serious Adverse Events Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Subjec<br>t<br>Number AE# | Adverse Event Verbatim/<br>System Organ Class/<br># Preferred Term | Start Date/<br>Stop Date/<br>(DDMMMYYYY/<br>DDMMMYYYY) | SAE<br>Criteria | Severity<br>(NCI-<br>CTCAE) | Severity Relationship Relationship<br>(NCI- to Study to Study<br>CTCAE) Drug Procedure | Relationship<br>to Study<br>Procedure | Action<br>Taken<br>with<br>Study<br>Drug | Other<br>Action | Outcome | TEAE |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX 1 | /xxxxxxxxxxxxxxxxxxxxx/x/x/x/x/xxxxxxxx | DDMMMYYYYY<br>HH:MM<br>DDMMMYYYYY<br>/YYYYY | Is Life<br>Threatening | Grade 1 | Possibly<br>Related | Possibly<br>Related | None | None | Recovered /<br>Resolved | Yes |
| N | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/<br>HH:MM<br>DDMMMYYYY/<br>HH:MM | Is Life<br>Threatening | Grade 1 | Definitely<br>not Related | Definitely<br>not Related | None | None | Recovered /<br>Resolved | Yes |
| XXX 1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYYY / YYYYYY HH: MM H: MM / HH: | Is Life<br>Threatening | Grade 1 | Definitely<br>not Related | Definitely<br>not Related | None | None | Recovered /<br>Resolved | N |
| ~ | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY / | Is Life<br>Threatening | Grade 1 | Definitely<br>not Related | Definitely<br>not Related | Drug<br>withdrawn | None | Recovered /<br>Resolved | Yes |
| etc. | | | | | | | | | | |

Note: TEAE = A treatment-emergent adverse event. MedDRA Version xx.x

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Listing 16.2.7.2.2 MAD: Serious Adverse Events Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.7.2.1 for MAD.

Listing 16.2.7.3.1 SD: Adverse Events Leading to Study Medication Discontinuation Protocol:  $\mathtt{BTI}-201$ 

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| TEAE | Yes | Yes | | O<br>N | ₹<br>es | |
|---|---|---|---|---|---|---|
| Outcome | Recovered /<br>Resolved | Recovered /<br>Resolved | | Recovered /<br>Resolved | Recovered /<br>Resolved | |
| Other | None | None | | None | None | |
| Action<br>Taken<br>with<br>Study<br>Drug | Drug<br>withdrawn | Drug<br>withdrawn | Drug<br>withdrawn | Drug<br>withdrawn | Drug<br>withdrawn | |
| Relationship<br>to Study<br>Procedure | Possibly<br>Related | Definitely<br>not Related | | Definitely<br>not Related | Definitely<br>not Related | |
| Relationship<br>to Study Drug | Possibly<br>Related | Definitely<br>not Related | | Definitely<br>not Related | Definitely<br>not Related | |
| Severity<br>(NCI-<br>CTCAE) | Grade 1 | Grade 1 | | Grade 1 | Grade 1 | |
| SAE | Yes | Yes | | No | NO | |
| Start Date/<br>Stop Date/<br>(DDMMMYYYY/<br>DDMMMYYYY) | DDWMYYYYY/<br>HH:WM<br>DDWMYYYYY/<br>HH:WM | DDMMMYYYY/<br>HH:MM<br>DDMMYYYYY/<br>HH:MM | | DDMMMYYYY/<br>HH:MM<br>DDMMYYYY/<br>HH:MM | DDMMMYYYY / | |
| Adverse Event Verbatim/<br>System Organ Class/<br>Preferred Term | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXX/ | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| AE# | П | ~ | | $\vdash$ | 2 | |
| Subject<br>Number | XXX | | | XXX | | etc. |

Note: TEAE = A treatment-emergent adverse event. MedDRA Version xx.x

Clinical cut-off date: DDMMMYYYY

Listing 16.2.7.3.2 MAD: Adverse Events Leading to Study Medication Discontinuation Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.7.3.1 for MAD.

Listing 16.2.7.4.1 SD: Overall Survival Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Subject | Date of First Study Drug<br>Administration<br>(DDMMMYYYY) | Event/Censoring<br>Date<br>DDMMYYYY) | Event or Censoring<br>Description | Days to Event |
|---|---|---|---|---|
| XXX | DDMMMXXXX | DDMMMYYYY | Death | XXX |
| XXX | DDMMMYYYY | DDMMMXXXX | Last assessment date | XXX |
| XXX | DDMMMYYYY | DDMMMXXXX | Last assessment date | XXX |
| XXX | DDMMYYYY | DDMMMXXXX | Death | XXX |
| (<br>+<br>( | | | | |
| יייי. | | | | |

Note: Overall Survival is defined as the difference (in days) between the the day of the study drug administration.)

Subjects who did not die will be censored at the study exit visit.

Clinical cut-off date: DDMMMYYYY

```
Listing 16.2.7.4.2 MAD: Overall Survival Protocol: BTI-201 Intent-to-Treat Population
```

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.7.4.1 for MAD.

Listing 16.2.8.1.1.1 SD: CBC Protocol: BTI-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Subject | Parameter (Unit) Study Visit | nit) | | Sample Date/<br>Time<br>(DDMMMYYYY/<br>HH:MM) | Actual<br>Value | Actual Change from Reference<br>Value Baseline <sup>1</sup> Ranges | Reference<br>Ranges | High/ Low<br>Flag | Clinical<br>Significance | Abnormality<br>Description |
|---|---|---|---|---|---|---|---|---|---|---|
| | Haemoglobin (unit) Screening | unit) | Screening | DDMMMYYYY/ | XX | | XX, XX | | | |
| | | | Day $1^1$ | /XXXXWIMID | × | | xx, xx | | | |
| | | | Day 2 | HH:MM<br>DDMMMYYYY/ | × | × | xx, xx | 田 | NCS | |
| | | | Day 3 or 4 | HH:MM<br>DDMMYYYY/<br>HH:MM | × | ×× | xx, xx | Ы | S. | ××××××××××××××××××××××××××××××××××××××× |

て 十 丘

Etc.

Note: <sup>1</sup>Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. L = Below Normal Range, H = Above Normal Range, NCS = Not Clinically Significant, CS = Clinically Significant.

Clinical cut-off date: DDMMMYYYY

Programming Note:

Include all time points and all parameters.
Listing 16.2.8.1.1.2 MAD: CBC Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.8.1.1.1 for MAD.

Include all time points and all parameters.

Listing 16.2.8.1.2.1 SD: Abnormal CBC Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | | | Sample Date/ | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Time | | | | | | |
| | | | /XXXXWWWQQ) | Actual | Actual Change from | Reference | High/ Low | Clinical | Abnormality |
| Subject | Parameter (Unit) Study Visit | Study Visit | HH:MM) | Value | Baseline <sup>1</sup> Ranges | Ranges | Flag | Significance | Description |
| XXX | Haemoglobin (unit) | Day 2 | /XXXXWWMQQ | × | XX | XX, XX | н | NCS | |
| | | | HH:MM | | | | | | |
| | | Day 3 or 4 | /XXXXWWMQQ | ×× | ×× | XX, XX | IJ | CS | XXXXXXXXXXXXXXX |
| | | | HH:MM | | | | | | |

E (

Etc.

Note: <sup>1</sup>Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. L = Below Normal Range, H = Above Normal Range, NCS = Not Clinically Significant, CS = Clinically Significant.

Clinical cut-off date: DDMMMYYYY

Programming Note:

Include all time points and all parameters.

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:NM


Listing 16.2.8.1.2.2 MAD: Abnormal CBC Protocol: BTI-201 Intent-to-Treat Population Cohort 2: rhu-pGSN 6 mg/kg


Programming Note:
Repeat Listing 16.2.8.1.2.1 for MAD.
Include all time points and all parameters.

Listing 16.2.8.2.1.1 SD: Coagulation Protocol: BTI-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | | | Sample Date/<br>Time | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Parameter (Unit) Study Visit | Study Visit | (DDMMMYYYY/) | | Actual Change from Reference<br>Value Baseline <sup>1</sup> Ranges | Reference<br>Ranges | High/ Low<br>Flag | Clinical<br>Significance | Abnormality<br>Description |
| XXX | PT/INR (unit) | Screening | / XXXXMMMQQ | ×× | | xx, xx | | | |
| | | | нн:мм | | | | | | |
| | | Day $1^1$ | /XXXXWWWQQ | ×× | | xx, xx | | | |
| | | | HH:MM | | | | | | |
| | | Day 2 | DDMMMXXXX/ | × | ×× | xx, xx | н | NCS | |
| | | | HH: MM | | | | | | |
| | | Day 3 or 4 | DDMMMXXXX/ | ×× | XX | xx, xx | Ц | CS | XXXXXXXXXXXXXX |
| | | | HH:MM | | | | | | |

Etc.

Note: <sup>1</sup>Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. L = Below Normal Range, H = Above Normal Range, NCS = Not Clinically Significant, CS = Clinically Significant.

Clinical cut-off date: DDMMMYYYY

Programming Note:

Include all time points and all parameters.

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM


Listing 16.2.8.2.1.2 MAD: Coagulation Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.8.2.1.1 for MAD.

Include all time points and all parameters.

Listing 16.2.8.2.2.1 SD: Abnormal Coagulation Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| Subject | Parameter (Unit) Study Visit | Study Visit | Sample Date/<br>Time<br>(DDMMMYYYY/<br>HH:MM) | Actual<br>Value | Change from Referenc<br>Baseline <sup>1</sup> Ranges | Reference<br>Ranges | High/ Low<br>Flag | Clinical<br>Significance | Abnormality<br>Description |
|---|---|---|---|---|---|---|---|---|---|
| XXX | PT/INR (unit) | Day 2<br>Day 3 or 4 | DDMMMYYYYY / HH:MM DDMMMYYYYY / HH:MM | × ×<br>× × | × × | xx 'xx xx | н н | NCS<br>CS | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Etc. Etc.

Note: <sup>1</sup>Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. L = Below Normal Range, H = Above Normal Range, NCS = Not Clinically Significant, CS = Clinically Significant.

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x)

Programming Note:

Include all time points and all parameters.

Created: DDMMMYYYY HH:MM


Listing 16.2.8.2.2.2 MAD: Abnormal Coagulation Protocol: BTI-201 Intent-to-Treat Population Cohort 2: rhu-pGSN 6 mg/kg


Include all time points and all parameters. Programming Note: Repeat Listing 16.2.8.2.2.1 for MAD.

Listing 16.2.8.3.1.1 SD: Comprehensive Metabolic Profile Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | | | Sample Date/<br>Time | r<br>- | ( | ſ | | - | - |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Parameter (Unit) Study Visit | Study Visit | (DDMMMYYYY/<br>HH:MM) | Actual<br>Value | Actual Change from Reference<br>Value Baseline <sup>1</sup> Ranges | Reterence<br>Ranges | Hıgh/ Low<br>Flag | Clinical<br>Significance | Abnormalıty<br>Description |
| XXX | Sodium (unit) | Screening | /XXXXMMQQ | × | | XX, XX | | | |
| | | $	extsf{Day} 1^1$ | /XXXXMMMQQ | × | | xx, xx | | | |
| | | Day 2 | HH:MM<br>DDMMMXYYY/ | × | × | xx, xx | н | NCS | |
| | | Day 3 or 4 | HH:MM DDMMMAXYY | × | ×× | XX, XX | ы | S | ××××××××××××××××××××××××××××××××××××××× |
| | | | HH: MM | | | | | | |

Etc.

Note: <sup>1</sup>Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. L = Below Normal Range, H = Above Normal Range, NCS = Not Clinically Significant; CS = Clinically Significant.

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Include all time points and all parameters. Programming Note:

Listing 16.2.8.3.1.2 MAD: Comprehensive Metabolic Profile Protocol: BTI-201
Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Include all time points and all parameters. Repeat Listing 16.2.8.3.1.1 for MAD. Programming Note:

Listing 16.2.8.3.2.1 SD: Abnormal Comprehensive Metabolic Profile Protocol: BII-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | | | Sample Date/ | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Time | | | | | | |
| | | | /XXXXWWMQQ) | Actual | Actual Change from Reference | Reference | High/ Low | Clinical | Abnormality |
| Subject | Parameter (Unit) Study Visit | Study Visit | HH:MM) | Value | $Baseline^1$ | Ranges | Flag | Significance | Description |
| XXX | Sodium (unit) | Day 2 | / XXXXWWMQQ | ×× | ×× | XX, XX | н | NCS | |
| | | | HH:MM | | | | | | |
| | | Day 3 or 4 | /XXXXWWMQQ | × | ×× | XX, XX | ı | CS | XXXXXXXXXXXXXX |
| | | | HH:MM | | | | | | |

Etc.

Note: <sup>1</sup>Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. L = Below Normal Range, H = Above Normal Range, NCS = Not Clinically Significant; CS = Clinically Significant.

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x)

Programming Note:

Include all time points and all parameters.

Created: DDMMMYYYY HH:MM


Listing 16.2.8.3.2.2 MAD: Abnormal Comprehensive Metabolic Profile Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note:

Repeat Listing 16.2.8.3.2.1 for MAD.

Include all time points and all parameters.


Listing 16.2.9.1 SD: Vital Signs Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| 1 | | | | |
|---|---|---|---|---|
| If Abnormal, specify | | XXXXXXXX | XXXXXXXXX | |
| Change Investigator's<br>from Overall If<br>Baseline <sup>1</sup> Interpretation | Normal | Abnormal NCS | Abnormal NCS | |
| | | | ×× | |
| Actual<br>Value | × | × | × | |
| Time<br>(HH:MM) | HH: MM | HH: MM | HH:MM | |
| Timepoint | | $Pre-dose^1$ | End of<br>Infusion | |
| Assessment<br>Date<br>(DDMMMYYYY) | DDMMMYYYY | AXXXMMDO | | |
| Study Visit | Screening | Day 1 | | |
| Assessment Performed - arameter Reason Not (Unit) Performed | X<br>⊕<br>S | Yes | | |
| Subjec Parameter<br>t (Unit) | Systolic<br>Blood | Fressure<br>(mmHg) | | Etc. |
| Subjec | × | | | Etc. |

Note: 'Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration. NCS = Not Clinically Significant, CS = Clinically Significant

Clinical cut-off date: DDMMMYYYY

Include all time points and all parameters.

Programming Note:

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM


Listing 16.2.9.2 MAD: Vital Signs Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.9.1.1 for the MAD.

Programming Note: Repeat Listing 16.2.9.1 for MAD.

Include all time points and all parameters.


Intent-to-Treat Population Listing 16.2.10.1 SD: EKG Protocol: BII-201

Cohort 1: rhu-pGSN 6 mg/kg

| If<br>Abnormal,<br>specify | | XXXXXXXXX | XXXXXXXX | | XXXXXXXXX |
|---|---|---|---|---|---|
| Worst<br>Investigator's<br>Overall<br>Interpretation | | Abnormal NCS | Abnormal NCS | | Abnormal NCS |
| Worst Mean Mean Change Investigator's Investigator's ctual from Overall Overall Value Baseline¹ Interpretation Interpretation | Normal | Abnormal NCS | Abnormal NCS<br>Abnormal NCS | Abnormal NCS | Abnormal CS |
| Mean Change<br>from<br>Baseline <sup>1</sup> | | | | | × × × |
| Mean<br>Actual<br>Value | | ××. | × × × | | ×.<br>× |
| Mean<br>Actual Actual<br>Value Value | × | × | × ×<br>× × | × | × |
| Time<br>(HH:MM) | нн:мм | нн:мм | HH:MM<br>HH:MM | нн:мм | нн:мм |
| Timepoint | EKG 1 | EKG 2 | EKG 1<br>EKG 2 | EKG 1 | EKG 2 |
| Assessment<br>Date<br>(DDMMMYYYY) | DDMMMYYYY | | ZYYYMMMQQ | DDMMMYYYY | |
| Assessment Performed - Assessment Mean Lrameter Reason Not Date Time Actual Actual (Unit) Performed Study Visit (DDMMMYYYY) Timepoint (HH:MM) Value Value | Screening DDMMMYYYY | | Day $1^1$ | Day 28 /<br>Early | Termination |
| Assessment Performed - Subjec Parameter Reason Not t (Unit) Performed | Yes | | Yes | Yes | |
| Parameter<br>(Unit) | Heart<br>Rate | (unit) | | | |
| Subjec I | ××× | | | | |

etc.

Note: <sup>1</sup>Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

NCS = Not Clinically Significant, CS = Clinically Significant

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Include all parameters. Programming Note:

Listing 16.2.10.2 MAD: EKG Protocol: BTI-201 Intent-to-Treat Population


Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.10.1 for MAD. Include all parameters.

Listing 16.2.11.1 SD: Physical Examination Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| <pre>If Abnormal,</pre> | 222222222222222222222222222222222222222 | 22222222222 | | | |
|---|---|---|---|---|---|
| Result | Normal<br>Normal<br>Abnormal NCS<br>Abnormal NCS | Normal<br>Normal<br>Abnormal NCS<br>Abnormal NCS | Normal<br>Normal | | Normal |
| Body System | Skin<br>HEENT<br><br>Musculoskeletal | Skin<br>HEENT<br><br>Musculoskeletal | Skin<br>HEENT | į | Musculoskeletal |
| Date/Time Physical Examination performed (DDMMMYYYYY) | DDMMXXXXX HH:MM | DDMMYYYY HH:MM | DDMMYYYY/ HH:MM<br> | | |
| Visit | Screening | Day 1 | Day 2 | | |
| Assessment Performed - Reason Not Performed | Yes | ⊗<br>O | K & K | NO -<br>ZZZZZZZZ | |
| Subject | ×× | | | XXX | ÷ |

Note: NCS = Not Clinically Significant, CS = Clinically Significant

Include all time points and all parameters. Programming Note:

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

2018-12-03

Listing 16.2.11.2 MAD: Physical Examination Protocol: BTI-201 Intent-to-Treat Population Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.9.11.1 for MAD. Include all time points and all parameters.

Listing 16.2.12.1.1 SD: Outcome Prediction Models CURB-65 Protocol: BII-201


Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | | Test | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Performed - | | | | Respiratory | Systolic/ | | CURB- | CURB-65 Score |
| | | Reason Not | | Confusion of Blood Urea | Blood Urea | Rate | Diastolic | Age | Actual | Actual Change from |
| Subject | Subject Study Visit | Performed | Visit Date | New Onset | Nitrogen ( | (breaths/min) | BP (mmHg) (years) | (years) | Value | $Baseline^1$ |
| XXXXX | $Screening^1$ | Yes | DDMMMXXXX | XX | xx (unit) | ×× | xx /xxx | × | ×× | |
| | Day 3/4 | Yes | DDMMMXXXX | ×× | xx (unit) | ×× | xx /xxx | × | × | ×× |
| | Day 7 | Yes | DDMMMXXXX | ×× | xx (unit) | ×× | xx /xxx | ×× | X | ×× |
| | Day 14 | Yes | DDMMMXYYY | ×× | xx (unit) | ×× | xx /xxx | × | × | ×× |
| | Day 28 / | Yes | DDMMMXYYY | ×× | xx (unit) | ×× | xx /xxx | × | × | ×× |
| | Early | | | | | | | | | |
| | Termination | | | | | | | | | |

Etc.

Note: <sup>1</sup>Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Listing 16.2.12.1.2 MAD: Outcome Prediction Models CURB-65 Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Repeat Listing 16.2.12.1.1 for MAD. Programming Note:


Listing 16.2.12.2.1 SD: Outcome Prediction Models PSI (Port Score) Protocol: BII-201

Intent-to-Treat Population

.

Cohort 1: rhu-pGSN 6 mg/kg

| | | Test Performed - | | | | |
|---|---|---|---|---|---|---|
| | | Reason Not | | PSI Score | core | |
| Subject | Study Visit | Performed | Visit Date | Actual Value | Change from ${\sf Baseline}^1$ | PSI Class |
| XXXXX | $Screening^1$ | Yes | DDMMMXXXX | ×× | | Н |
| | Day 3/4 | Yes | DDMMMXXXX | ×× | XX | II |
| | Day 7 | Yes | AXXXMMMQQ | ×× | ×× | III |
| | Day 14 | Yes | AXXXMMMQQ | ×× | ×× | IV |
| | Day 28 / Early | Yes | DDMMMXXXX | ×× | XX | $\wedge$ |
| | Termination | | | | | |

Etc.

Note: 'Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:MM

Listing 16.2.12.2.2 MAD: Outcome Prediction Models PSI (Port Score) Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Repeat Listing 16.2.12.2.1 for MAD. Programming Note:

Listing 16.2.12.3.1 SD: Outcome Prediction Models SOFA Score Protocol:  $\mathtt{BTI}-201$ 

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | | Host Dorformed - | | SOFA Score | |
|---|---|---|---|---|---|
| Subject | Study Visit | | Visit Date | Actual Value | Change Irom<br>Baseline <sup>1</sup> |
| XXXXX | $Screening^1$ | Yes | DDMMMYYYY | XX | |
| | Day 3/4 | Yes | DDMMMXXXX | ×× | ×× |
| | Day 7 | Yes | DDMMMXXXX | ×× | ×× |
| | Day 14 | Yes | DDMMMXXXX | ×× | ×× |
| | Day 28 / Early | Yes | DDMMMYYYY | ×× | ×× |
| | Termination | | | | |

Etc.

Note: <sup>1</sup>Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Listing 16.2.12.3.2 MAD: Outcome Prediction Models SOFA Score Protocol: BTI-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.12.3.1 for MAD.

Listing 16.2.12.4.1 SD: Outcome Prediction Models MMSE Score Protocol:  $\mathtt{BTI}-201$ 

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | | | | MMSE | Score | |
|---|---|---|---|---|---|---|
| Subject | Study Visit | Test Performed -<br>Reason Not Performed | Visit Date | Actual Value | Change from<br>Baseline <sup>1</sup> | ı |
| XXXXX | $Screening^1$ | Yes | DDMMMXYYY | ×× | | |
| | Day 3/4 | Yes | ZZZZMMMQQ | ×× | ×× | |
| | Day 7 | Yes | ZZZZMMMQQ | ×× | ×× | |
| | Day 14 | Yes | ZZZZMMMQQ | ×× | ×× | |
| | Day 28 / Early | Yes | ZZZZMMMQQ | ×× | ×× | |
| | Termination | | | | | |

etc.

Note: <sup>1</sup>Baseline. Baseline is defined as the last valid, non-missing assessment prior to first study drug administration.

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Listing 16.2.12.4.2 MAD: Outcome Prediction Models MMSE Score Protocol: BTI-201
Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Repeat Listing 16.2.12.4.1 for MAD. Programming Note:

Listing 16.2.13.1 SD: Concomitant Medications Protocol: BTI-201 Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | Route | 22222 | Z Z Z Z Z Z Z | 22222 | Z Z Z Z Z Z Z | 22222 | |
|---|---|---|---|---|---|---|---|
| | Frequency | XXXXXX | YYYYY | XXXXXX | YYYYY | XXXXXX | |
| | Unit | Unit | Unit | Unit | Unit | Unit | |
| | Dose | × | × | × | × | × | |
| | Ongoing | O<br>N | N | O<br>Z | Y<br>e<br>s | N | |
| Start Date/<br>Stop Date | (DDMMMXYYY) | DDMMMYYYY / | DDMMMYYYY / | DDMMMYYYY / | DDMMMYYYY /<br>Ongoing | DDMMMYYYY / | |
| | Indication | To treat AE: AE# | Other: YYYYY | Other: YYYYYY | Other: YYYYY | To treat AE: AE# | |
| | Drug Name/ATC3/PT | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | CM# | Н | N | Н | N | Н | |
| Subject | Number | XXX | | XXX | | XXX | Etc. |

Note: Concomitant medications are medications taken at least once after first study-drug administration. WHO-DD, xxxxxxxxxxx

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMYYYY HH:NM


Listing 16.2.13.2 MAD: Concomitant Medication Protocol: BTI-201 Intent-to-Treat Population


Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.9.13.1 for MAD.


Listing 16.2.14.1 SD: Hospitalization Follow-Up Protocol: BTI-201

Intent-to-Treat Population

Cohort 1: rhu-pGSN 6 mg/kg

| | | | | Require | Vasopressors | No | No | No | No | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Administered F | Antibiotics Vas | Yes | No | No | No | |
| Intubation | | | | Number of | Days | ×× | | | | |
| Intuk | | | | | Yes/No | Yes | No | No | No | |
| ICU Stay | | | | Number of | Days | ×× | XX | | | |
| ICU | | | | | Yes/No | Yes | Yes | No | No | |
| | | | Number | of | Hours | × | ×× | ×× | ×× | |
| Length of Hospital Stay | Date and Time of Date/ Time of | Jace, Illie or<br>ischarge/ Study | Hospitalization Discharge/ Study Admission due to Exit | Exit | (DDMMMXYYY/ | HH:MM) | DDMMYYYYY HH:MM DDMMMYYYY HH:MM | MM:HH / XXXXMMMOO | DMMMYYYY/ HH:MM | DMMMYYYY/ HH:MM |
| ngth of | ime of | ation D | Discharged Admission due to | CAP (DDMMMYYYY/ | ) | HH:MM | HH: MM | HH:MM | HH:MM D | |
| Le | Date and T | Date and I<br>Hospitaliz | | | HH: MM) | /XXXXMMMQQ | /XXYMMMDDMM:HH /YYYYYY/ | DDMMMYYYY HH: MM DDMMMYYYY / | DDMMMYYYY, HH:MM DDMMMYYYY/ | |
| | | | Discharged | from | Hospital | Yes | Yes | Yes | No | |
| | | | | | Subject | XXX | XXX | XXX | XXX | etc. |

Note: Length of stay in hospital is defined as the date and time of discharge/date of study exit (23:59 PM) date and time of hospitalization admission due to CAP in hours

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:NM

Listing 16.2.14.2 MAD: Hospitalization Follow-Up Protocol: BII-201 Intent-to-Treat Population

Cohort 2: rhu-pGSN 6 mg/kg

Programming Note: Repeat Listing 16.2.14.1 for MAD.


# **BTI-201: Mock Figures: Table of Contents**

#### Figures

## **GENERAL COMMENTS**


Names of Treatment Groups: SD:

rhu-pGSN 6 mg/kg.

MAD:

rhu-pGSN 6 mg/kg; rhu-pGSN 12 mg/kg; rhu-pGSN 24 mg/kg.

Names of PK sampling times: Day 1 (SD and MAD) & Day 3 (MAD)

Pre-injection 5 to 10 mins 2h 8h 12h 16h 24h

Figure 14.2.1.1 Individual pGSN Plasma Concentrations (ng/mL) (Linear scale) by Day Protocol: BTI-201 PK Populations

Day 1

### Programming Note:

The x-axis will represent the actual study time in hours (0 - 24 hours).

The y-axis will represent the pGSN Plasma Concentrations (ng/mL). The y-axis will be on the linear scale.

All subjects will be represented on a single page. Each dose level will be presented as a distinct line type. A separate figure will be created for each Day. SD and MAD subjects will be presented on the same page by Day.

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Figure 14.2.1.2 Individual pGSN Plasma Concentrations (ng/mL) (Semi-logarithmic) by Day Protocol: BTI-201 PK Populations

Day 1

### Programming Note:

The x-axis will represent the actual study time in hours (0-24 hours).

The y-axis will represent the pGSN Plasma Concentrations (ng/mL). The y-axis will be on the log scale.

All subjects will be represented on a single page. Each dose level will be presented as a distinct line type. A separate figure will be created for each Day. SD and MAD subjects will be presented on the same page by Day.

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Figure 14.2.2.1 Individual Estimated Plasma rhu-pGSN Plasma Concentrations (ng/mL) based on Changes from Pre-Injection (Linear scale) by Day

Protocol: BTI-201 PK Populations

#### Day 1

### Programming Note:

The x-axis will represent the actual study time in hours (0-24 hours).

The y-axis will represent the Estimated Plasma rhu-pGSN Concentrations (ng/mL). The y-axis will be on the linear scale.

All subjects will be represented on a single page. Each dose level will be presented as a distinct line type. A separate figure will be created for each Day. SD and MAD subjects will be presented on the same page by Day.

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY

Figure 14.2.2.2 Individual Estimated Plasma rhu-pGSN Plasma Concentrations (ng/mL) based on the Double Delta Analysis (Linear scale) by Day

Protocol: BTI-201 PK Populations

Day 1

### Programming Note:

The x-axis will represent the nominal study time in hours (0-24 hours).

The y-axis will represent the Estimated Plasma rhu-pGSN Concentrations (ng/mL). The y-axis will be on the linear scale.

All subjects will be represented on a single page. Each dose level will be presented as a distinct line type. A separate figure will be created for each Day. SD and MAD subjects will be presented on the same page by Day.

Clinical cut-off date: DDMMMYYYY

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Figure 14.2.3.1 Mean (+/-SD) pGSN Plasma Concentrations (ng/mL) (Linear scale) by Day Protocol: BTI-201 PK Populations

#### Day 1

### Programming Note:

The x-axis will represent the nominal study time in hours (0-24 hours).

The y-axis will represent the mean pGSN Plasma Concentrations (ng/mL) per Dose level. Whiskers will be included to reflect the SDs. The y-axis will be on the linear scale. All treatments will be represented on a single page. Each dose level will be presented as a distinct line type.

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY

Figure 14.2.3.2 Mean (+/-SD) pGSN Plasma Concentrations (ng/mL) based on Changes from Pre-Injection (Linear scale) by Day (Semi-logarithmic) by Day

Protocol: BTI-201 PK Populations

#### Day 1

Programming Note:

The x-axis will represent the nominal study time in hours (0-24 hours).

The y-axis will represent the mean rhu-pGSN Plasma Concentrations (ng/mL) per Dose level. Whiskers will be included to reflect the SDs. The y-axis will be on the log scale. All treatments will be represented on a single page. Each dose level will be presented as a distinct line type.

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Figure 14.2.4.1 Mean (+/-SD) Estimated Plasma rhu-pGSN Plasma Concentrations (ng/mL) based on Changes from Pre-Injection (Linear scale) by Day

Protocol: BTI-201 PK Populations

#### Day 1

### Programming Note:

The x-axis will represent the nominal study time in hours (0-24 hours).

The y-axis will represent the mean Estimated Plasma rhu-pGSN Plasma Concentrations (ng/mL) per Dose level. Whiskers will be included to reflect the SDs. The y-axis will be on the linear scale. All treatments will be represented on a single page. Each dose level will be presented as a distinct line type.

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Figure 14.2.4.2 Mean (+/-SD) Estimated Plasma rhu-pGSN Plasma Concentrations (ng/mL) based on the Double Delta Analysis (Linear scale) by Day

Protocol: BTI-201 PK Populations

#### Day 1

### Programming Note:

The x-axis will represent the nominal study time in hours (0-24 hours).

The y-axis will represent the mean Estimated Plasma rhu-pGSN Plasma Concentrations (ng/mL) per Dose level. Whiskers will be included to reflect the SDs. The y-axis will be on the linear scale. All treatments will be represented on a single page. Each dose level will be presented as a distinct line type.

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Figure 14.3.1.1 SD: Kaplan-Meier Plot of Overall Survival Time Protocol: BTI-201 Safety Population Note: Overall Survival is defined as the difference (in days) between the time of first study drug administration to the date of death + 1 (Include the day of the study drug administration.) Subjects who did not die will be censored at the study exit visit.

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: rhu-pGSN and combined Placebo treatments will be presented on one graph.


Figure 14.3.1.2 MAD: Kaplan-Meier Plot of Overall Survival Time Protocol: BTI-201 Safety Population

Note: Overall Survival is defined as the difference (in days) between the time of first study drug administration to the date of death + 1 (Include the day of the study drug administration.) Subjects who did not die will be censored at the study exit visit.

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: rhu-pGSN and combined Placebo treatments will be presented on one graph.

Figure 14.3.2.1 SD: Kaplan-Meier Plot of Length of Stay in Hospital (hours) Protocol: BTI-201 Safety Population

Note: Length of stay in hospital is defined as the date and time of discharge/date of study exit (23:59 PM ) - date and time of hospitalization admission due to CAP in hours

Clinical cut-off date: DDMMMYYYY Program: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: rhu-pGSN and combined Placebo treatments will be presented on one graph.

Figure 14.3.2.2 MAD: Kaplan-Meier Plot of Length of Stay in Hospital (hours) Protocol: BTI-201 Safety Population

Note: Length of stay in hospital is defined as the date and time of discharge/date of study exit (23:59 PM ) - date and time of hospitalization admission due to CAP in hours

Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM Clinical cut-off date: DDMMMYYYY

Programming Note: rhu-pGSN and combined Placebo treatments will be presented on one graph.

Figure 14.3.3.1 SD: Kaplan-Meier Plot of Duration of ICU Stay Protocol:  ${\tt BTI-201}$  Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: rhu-pGSN and combined Placebo treatments will be presented on one graph. Only include subjects that stayed in the ICU.

Figure 14.3.3.2 MAD: Kaplan-Meier Plot of Duration of ICU Stay Protocol: BTI-201 Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: rhu-pGSN and combined Placebo treatments will be presented on one graph. Only include subjects that stayed in the ICU.

Figure 14.3.4.1 SD: Kaplan-Meier Plot of Duration of Intubation Protocol:  ${\tt BTI-201}$  Safety Population

Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: rhu-pGSN and combined Placebo treatments will be presented on one graph. Only include subjects that were intubated.


Figure 14.3.4.2 MAD: Kaplan-Meier Plot of Duration of Intubation Protocol: BTI-201 Safety Population Clinical cut-off date: DDMMMYYYY
Program: filepath\_name, Output: filepath\_name (version x.x) Created: DDMMMYYYY HH:MM

Programming Note: rhu-pGSN and combined Placebo treatments will be presented on one graph. Only include subjects that were intubated.